### CLINICAL STUDY PROTOCOL

**Study Title:** A Two-Part Study of ZX008 in Children and Adults with

> Lennox-Gastaut Syndrome (LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures in Children and Adults with Assess Long-Term Safety of ZX008 in Children and Adults with LGS
>
> ZX008-1601
>
> Fenfluramine Hydrochloride Oral Solution; ZX008

**Study Number:** 

Fenfluramine Hydrochloride Oral Solution; ZX008 132604 **Study Product:** 

**IND Number:** 

2017-002628-26 **EudraCT Number:** 

Zogenix International Limited **Sponsor:** 

A wholly owned subsidiary of UCB Biosciences, Inc.

4000 Paramount Pkwy,

Morrisville, NC 27560,

Sponsor's Medical

**Contact:** 

Program Physician UCB Biosciences Inc

Date and Version of

25 July 2022 (PA 4.0 Japan)

**Study Protocol:** 

29 July 2020 (PA 3.2 Japan)

29 October 2018 (PA 1.6.1 Japan)

Based on 10 January 2018 (Amendment 1.0 ROW)

This protocol includes information and data that contain trade secrets and privileged or confidential information, which is the property of the sponsor. This information must not be made public without written permission from the sponsor. These restrictions on disclosure will apply equally to all future information supplied to you. This material may be disclosed to and used by your personnel and associates as may be necessary to conduct the clinical study.

And the application and any extensions of value of the lead to support any nativity as the real to support any nativity and any support any nativity as the real to support any nativity and any support any nativity as the real to support any nativity and any support any nativity and any support any nativity and any support and any support and any support any support and support any support and support any support and support any support and suppor


# **TABLE OF CONTENTS**

| CLINICAL STUDY PROTOCOL | 1 |
|---|---|
| LIST OF PERSONNEL AND ORGANIZATIONS RESPONSIBLE FOR CONDUCT OF STUDY | 2 |
| STUDY TABLE OF CONTENTS SIGNATURE OF SPONSOR | 3 |
| SIGNATURE OF SPONSOR | 11 |
| SIGNATURE OF COORDINATING INVESTIGATOR | ¢ 12 |
| SIGNATURE(S) OF THE PRINCIPAL INVESTIGATOR | <sub>13</sub> |
| LIST OF ABBREVIATIONS | 14 |
| STUDY SYNOPSIS | 16 |
| 1. INTRODUCTION | 34 |
| T L BACKGROUND INFORMATION ON INDICATION STUDIED | - 34 |
| 1.1.1 Existing Treatment for LGS | 34 |
| 1.1.1 Existing Treatment for LGS | 35 |
| 1.3 CLINICAL DATA | 35 |
| 1.4 PHARMACOKINETICS, PRECLINICAL DATA, AND CLINICAL PHARMACOLOGY | 38 |
| 1.4.1 Pharmacokinetics | 38 |
| 1.4.2 Preclinical Data | 39 |
| 1.4.3 Clinical Pharmacology | |
| 1.5 BACKGROUND INFORMATION ON REFERENCE PRODUCT | 40 |
| 1.6 RATIONALE FOR CURRENT STUDY | 40 |
| 1.7 RISK-BENEFIT ASSESSMENT | 42 |
| 2. STUDY OBJECTIVES AND ENDPOINTS | 43 |
| 2.1 PART 1 | 43 |
| 21.1 PRIMARY OBJECTIVE | |
| 2.1.2 KEY SECONDARY OBJECTIVES | 43 |
| 2.1 PART 1 | 43 |
| 2.1.4 SAFETY OBJECTIVE | 44 |
| 2.1.5 PHARMACOKINETIC OBJECTIVE | 44 |
| 2.1.6 EXPLORATORY OBJECTIVES | 45 |
| 2.2 PART 2 | 45 |

| | 2.2.1 PRIMARY OBJECTIVE | 45 |
|---|---|---|
| | 2.2.2 SECONDARY OBJECTIVES | 45 |
| | 2.2.3 EXPLORATORY OBJECTIVES | 46 |
| | 2.3 STUDY ENDPOINTS | 46 |
| | 2.3.1 Efficacy Endpoints | |
| | 2.3.2 Safety Endpoints | 47 |
| | 2.3.2 Safety Endpoints 2.3.3 Exploratory Endpoints INVESTIGATIONAL PLAN 3.1 OVERALL STUDY DESIGN AND PLAN 3.2 NUMBER OF SUBJECTS 3.3 STUDY DURATION 3.4 NUMBER OF STUDY CENTERS 3.5 RATIONALE FOR STUDY DESIGN AND CHOICE OF TREAT | 47 |
| 3. | INVESTIGATIONAL PLAN | 48 |
| | 3.1 OVERALL STUDY DESIGN AND PLAN | 48 |
| | 3.2 NUMBER OF SUBJECTS | 49 |
| | 3.3 STUDY DURATION | 49 |
| | 3.4 NUMBER OF STUDY CENTERS | 50 |
| | 3.5 RATIONALE FOR STUDY DESIGN AND CHOICE OF TREAT GROUPS | ΓΜΕΝΤ<br>51 |
| | 3.6 RATIONALE FOR STUDY DESIGN AND CHOICE OF TREAT GROUPS | <b>IMENT</b> |
| | 3.7 PREMATURE TERMINATION OF STUDY | 52 |
| | 3.8 STUDY MONITORING PROCEDURES | 52 |
| | 3.8.1 Independent Data Safety Monitoring Committee | 52 |
| | 3.8.2 International Cardiac Advisory Board (ICAB) | 53 |
| 4. | SELECTION OF STUDY POPULATION | 54 |
| | 4.1 PART 0 | 54 |
| | 4.1.1 INCLUSION CRITERIA | 54 |
| | 4.1.2 EXCLUSION CRITERIA | 55 |
| | 4.2 RANDOMIZATION INCLUSION CRITERIA | |
| 90cn | 4.3 PART 2 | 57 |
| | 4.4 SUBJECTS OF REPRODUCTIVE POTENTIAL | 58 |
| | 4.4.1 Sperm and Egg Donation | 59 |
| 90 | 4.4.2 Pregnancy | 59 |
| | 4.5 REMOVAL OF SUBJECTS FROM THERAPY OR ASSESSME | NT 59 |
| | 4.6 TERMINATION OF THE CLINICAL STUDY | 61 |
| | 4.7 REPLACEMENT OF SUBJECTS | 61 |
| 5 | INVESTIGATIONAL MEDICINAL PRODUCT INFORMATION | 62 |

| | 5.1 IDENTITY OF INVESTIGATIONAL MEDICINAL PRODUCT | 62 |
|---|---|---|
| | 5.1.1 Labeling and Packaging | 62 |
| | 5.2 DESCRIPTION OF REFERENCE TREATMENT, COMPARATOR, AND/OR PLACEBO | 63 |
| | 5.2.1 Labeling and Packaging | 63 |
| | 5.3 SHIPMENT AND STORAGE | . 63 |
| | 5.4 IMP ACCOUNTABILITY | 63 |
| | 5.5 TREATMENT ADMINISTRATION | . 64 |
| | 5.5.1 Part 1: Randomization 5.5.1.1 Blinding 5.5.2 Part 1: Titration Period 5.5.3 Part 1: Maintenance Period | 64 |
| | 5.5.1.1 Blinding | 64 |
| | 5.5.2 Part 1: Titration Period | 65 |
| | 5.5.3 Part 1: Maintenance Period | 66 |
| | 5.5.4 Part 1: Taper Period (for subjects not entering Part 2) | 66 |
| | 5.5.5 Part 1: Transition Period | 67 |
| | 5.5.6 Part 2: OLE Treatment Period | 68 |
| | 5.5.7 Taper Period | 69 |
| | 5.6 PRIOR AND CONCOMPTANT MEDICATION | 70 |
| | 5.6.1 Vagal Nerve Stimulation | 71 |
| | 5.6.2 Ketogenic Diet | 71 |
| | 5.6.3 Rescue Medication for Seizures | |
| | 5.6.4 Prohibited Concomitant Medications | 71 |
| | 5.7 TREATMENT COMPLIANCE | |
| 6. VISIT | SCHE <b>D</b> ULE | 73 |
| 6.1 Part 1 | | 73 |
| Α. | 6.1.1 BASELINE PERIOD (STUDY DAY -28 TO STUDY DAY -1) | 73 |
| ochwey | 6.1.11. Screening, Clinic Visit 1 (Study Day -28) | 73 |
| collin of | 6-1.1.2. Phone Visit 2 (Study Day -15) | 75 |
| 100 SK | 6.1.1.3. Clinic Visit 3 (Study Day -1): Randomization | 75 |
| <b>&gt;</b> | 6.1.2 TITRATION AND MAINTENANCE PERIODS | 77 |
| | 6.1.2.1 Titration Period Study Day 1 | 77 |
| | 6.1.2.2 Phone Visits 4 and 5 (Titration Period Study Days 4 and 8) | 77 |
| | 6.1.2.3 Clinic Visit 6 (Titration Period Study Day 15) | 77 |


| | 6.1.2.4 Phone Visit 7 (Maintenance Period Study Day 29) | 77 |
|---|---|---|
| | 6.1.2.5 Clinic Visit 8 (Maintenance Period Study Day 43) | 78 |
| | 6.1.2.6 Phone Visit 9 (Maintenance Period Study Day 57) | 78 |
| | 6.1.2.7 Clinic Visit 10 (Maintenance Period Study Day 71) | 79 |
| | 6.1.2.8 Phone Visit 11 (Maintenance Period Study Day 85) | 79 |
| | 6.1.2.9 Clinic Visit 12 (Maintenance Period Study Day 99): End of Study/Early Termination | 79 |
| | 6.1.3 POST-DOSE VISIT (CLINIC VISIT 13; STUDY DAY 113) | 81 |
| | 6.1.4 CARDIAC FOLLOW-UP VISIT (CLINIC VISIT 14; 3 and 6 morafter last dose) | $\smile$ |
| 6.2 | Part 2 | 82 |
| 6.2.1 | Clinic Visit 15 (OLE Study Day 1) | 83 |
| 6.2.2 | Clinic/Phone Visit 16 (OLE Study Day 15) | 84 |
| 6.2.3 | Clinic Visit 15 (OLE Study Day 1) Clinic/Phone Visit 16 (OLE Study Day 15) Clinic Visits 17-21 (OLE Months, 1, 2, 3, 6, and 9) Clinic Visit 22 (OLE Month 12) | 85 |
| 6.2.4 | Clinic Visit 22 (OLE Month 12) | 86 |
| 6.2.5 | Clinic Visits 23-41 (OLE Months 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 5 57, 60, 63, 66, 69) | 1, 54, |
| 6.2.6 | Clinic Visit 42: End of Study/Early Termination | 88 |
| 6.2.7 | POST-DOSE VISIT (CLINIC Visit 43; 14 DAYS AFTER LAST DOSE OF IM | P) 90 |
| 6.2.8 | CARDIAC FOLLOW-UP VISIT (CLINIC VISIT 44, 45; 3 AND 6 MONTHS A LAST DOSE OF IMP) | 90 |
| 6.3 | STUDY CONDUCT DURING COVID-19 | |
| 6.4 | ESTIMATED BLOOD VOLUME COLLECTION | |
| 7. | EFFICACY, SAFETY, AND PHARMACOKINETIC ASSESSMENTS | |
| | 7.1) EFFICACY/EFFECTIVENESS ASSESSMENTS | |
| | 7.1.1 Seizure Assessments | |
| | 7.1-2 Clinical Global Impression - Improvement | |
| | 7.1.1 Seizure Assessments 7.1.2 Clinical Global Impression - Improvement. 7.1.3 Vineland Adaptive Behavior Scale (VABS). 7.1.4 QOLCE. 7.1.5 Parent/Caregiver Affective Symptoms | |
| 100 | 7.1.4 QOLCE | |
| <u> </u> | , the Talena categories simples in | |
| | 7.2 SAFETY ASSESSMENTS | |
| | 7.2.1 Demographics, Medical/Neurological/Epilepsy History, and Pre-S Medication | - |
| | 7.2.2 Adverse Events | 97 |


| 7.2.3 Physical Examinations | 97 |
|---|---|
| 7.2.4 Neurological Examinations | 97 |
| 7.2.5 Vital Signs (Including Height and Weight) | 98 |
| 7.2.6 Laboratory Measurements | 98 |
| 7.2.7 Plasma Sample for Concomitant Antiepileptic Drug(s) | 99 |
| 7.2.8 Electrocardiograms | |
| 7.2.9 Doppler Echocardiography | 99 |
| 7.2.10 Behavior Rating Inventory of Executive Function (BRIEF | F)99 |
| 7.2.11 Tanner Staging | |
| 7.2.12 Columbia-Suicide Severity Rating Scale | |
| 7.3 PHARMACOKINETIC ASSESSMENTS | 100 |
| 7.4 EPILEPSY GENOTYPE PANEL | 100 |
| 7.2.11 Tanner Staging | 101 |
| A DAMED OF TAXABLE AND A STATE OF TAXABLE AND | 1.00 |
| 8.1 DEFINITIONS | 102 |
| 8.1.1 Adverse Events | 102 |
| 8.1.2 Serious Adverse Events | 103 |
| 8.1.3 Adverse Events of Special Interest | |
| 8.2 SEVERITY OF ADVERSE EVENTS | 104 |
| 8.3 CAUSALITY OF ADVERSE EVENTS | 105 |
| 8.4 OBSERVATION PERIOD FOR ADVERSE EVENT REPO | RTING 105 |
| 8.5 ADVERSE EVENT REPORTING | 106 |
| 8.5.1 Adverse Events | |
| 8.6 SERIOUS ADVERSE EVENTS REPORTING | 106 |
| 8.6.1 Requirements for Immediate Reporting of Serious Adverse | Events 107 |
| 8.7 REPORTING OF SERIOUS ADVERSE EVENTS BY INVI | |
| TO IEC/IRB | |
| 8.6.1 Requirements for Immediate Reporting of Serious Adverse 8.7 REPORTING OF SERIOUS ADVERSE EVENTS BY INVITABLE TO IEC/IRB | |
| 8.9 FOLLOW-UP OF ADVERSE EVENTS | 108 |
| 8.9.1 Follow-up of Echocardiogram Findings | 108 |
| 8.10 PREGNANCY | 110 |
| 9. DATA HANDLING PROCEDURES | 110 |


| | 9.1 RECORDING OF DATA | 110 |
|---|---|---|
| | 9.2 DATA QUALITY ASSURANCE | 111 |
| | 9.3 RECORD RETENTION | 111 |
| 10. | STATISTICS | 112 |
| | 10.1 STATISTICAL ANALYSIS: PART 1 | 112 |
| | 10.1.1 DETERMINATION OF SAMPLE SIZE | 112 |
| | 10.1.2 ANALYSIS POPULATIONS | 112 |
| | 10.1.2.1 Safety (SAF) Population | 112 |
| | 10.1.2.2 Modified Intent-to-Treat (mITT) Population | 113 |
| | 10.1.2.3 Per Protocol (PP) Population | 113 |
| | 10.1.3 SUBJECT COHORTS | 113 |
| | 10.1.3.1 Cohort A | 113 |
| | 10.1.3.2 Cohort B | 113 |
| | 10.1.1 DETERMINATION OF SAMPLE SIZE 10.1.2 ANALYSIS POPULATIONS 10.1.2.1 Safety (SAF) Population 10.1.2.2 Modified Intent-to-Treat (mITT) Population 10.1.2.3 Per Protocol (PP) Population 10.1.3 SUBJECT COHORTS 10.1.3.1 Cohort A 10.1.3.2 Cohort B 10.1.4 TREATMENT GROUPS | 113 |
| | 10.1.5 TICHTIMETOT LEIGODO | 113 |
| | 10.1.6 STATISTICAL ANALYSES AND METHODS | 114 |
| | 10.1.6.1 Efficacy Analyses | 114 |
| | 10.1.6.2 Safety Analyses | 115 |
| | 10.1.6.3 Pharmacokinetic Analyses | |
| | 10.2 STATISTICAL ANALYSIS: PART 2 | 116 |
| | 10.2.1 ANALYSIS POPULATIONS | 116 |
| | 10.2.1.1 OLE Population | 116 |
| | 10.212 OLE mITT Population | 116 |
| | 10.2.2 TREATMENT GROUPS | |
| | 10.2.3 TREATMENT PERIODS | 116 |
| 40cu | 1024 STATISTICAL ANALYSES AND METHODS | 117 |
| رن | 10.2.4.1 Safety Analyses | 117 |
| 700 | 10.2.4.2 Effectiveness Analyses | 117 |
| | 10.2.5 ANALYSES PROVIDED TO AN INDEPENDENT DATA A | |
| | SAFETY MONITORING COMMITTEE | |
| 11. | ETHICAL & REGULATORY CONSIDERATIONS | |
| | 11.1 ETHICAL CONSIDERATIONS | 117 |

| 11.2 INFORMED CONSENT | 118 |
|---|---|
| 11.3 REGULATORY CONSIDERATIONS AND INDEPENDENT ET COMMITTEE/INSTITUTIONAL REVIEW BOARD | |
| 11.4 PROTOCOL COMPLIANCE | 120 |
| 12. ADMINISTRATIVE ASPECTS | 120 |
| 12.1 CLINICAL TRIAL AGREEMENT | 120 |
| 12.2 FINANCIAL DISCLOSURE BY INVESTIGATOR | _ \ / |
| 12.3 CLINICAL STUDY REGISTRATION AND RESULTS DISCLO | SURE |
| 12.4 STUDY FILES AND MATERIALS | 121 |
| 12.5 INITIATION OF THE STUDY | 121 |
| 12.6 SUBJECT REIMBURSEMENT | 122 |
| 12.7 LIABILITY AND INSURANCE | 122 |
| 12.8 SUBJECT IDENTIFICATION AND CONFIDENTIALITY | 122 |
| 12.9 MONITORING OF THE STUDY | |
| 12.10 PROTOCOL AMENDMENTS | 123 |
| 12.11 AUDITS AND INSPECTIONS | 124 |
| 12.12 CLINICAL STUDY REPORT | 124 |
| 12.13 USE OF DATA AND PUBLICATIONS | 124 |
| 13. REFERENCE LIST | 126 |
| 14. APPENDICES | 129 |
| APPENDIX 1 – LIST OF PROHIBITED CONCOMITANT MEDICATIONS | 129 |
| APPENDIX 2 – COLUMBIA – SUICIDE SEVERITY RATING SCALE | 131 |
| APPENDIX 3 – BEHAVIOR RATING INVENTORY OF EXECUTIVE FUNCTION | 136 |
| APPENDIX 4 – VINELAND ADAPTIVE BEHAVIOR SCALE | 146 |
| APPENDIX 5 – TANNER STAGING | 164 |
| APPENDIX 6 QOLCE QUALITY OF LIFE | 167 |
| APPENDIX 7 HOSPITAL ANXIETY AND DEPRESSION SCALE | 179 |
| APPENDIX 8 – ZARIT CAREGIVER BURDEN INVENTORY | 182 |
| APPENDIX 9 – MAXIMUM ALLOWABLE BLOOD DRAW VOLUMES | 184 |
| APPENDIX 10 – STUDY CONDUCT DURING COVID-19 | 185 |
| APPENDIX 11 - SUMMARY OF PROTOCOL AMENDMENT 4.0 | 188 |


| LIST | <b>OF</b> | TA | BL | ES |
|------|-----------|----|----|----|
|------|-----------|----|----|----|

| Table 1. | Schedule of Assessments: Part 1 | 29 |
|---|---|---|
| Table 2. | Schedule of Assessments: Part 2 Cohort B only | 31 |
| Table 3 | Post Hoc Estimates of Fenfluramine and Norfenfluramine Steady-State | |
| Pharmac | okinetic Parameters in Subjects with Dravet Syndrome in Study 1 (Geometric Mean | l |
| [CV%]). | | |
| Table 4: | Investigational Medicinal Product – ZX008 | 62 |
| Table 5: | Titration Algorithm for Part 1. | |
| Table 6: | Taper Algorithm for Part 1 | 67 |
| Table 7: | Transition Algorithm for Part 1 | 67 |
| Table 8. | Transition Algorithm for Part 1 Taper Algorithm for Part 2 Time Windows for Assessments in Part 1 Schedule of Post-Treatment Cardiac Follow-up for Part 1 | 69 |
| Table 9: | Time Windows for Assessments in Part 1 | 73 |
| Table 10 | Schedule of Post-Treatment Cardiac Follow-up for Part 1 | 82 |
| Table 11 | : Schedule of Post-Treatment Cardiac Follow-up for Part 1 | 83 |
| Table 12 | Schedule of Post-Treatment Cardiac Follow-up for Part 2 | 91 |
| Table 13 | : Maximum Estimated Blood Volume Collection for Part 1* | 92 |
| Table 14 | . Maximum Estimated Blood Volume Collection for Part 2* | 92 |
| Table 15 | Maximum Estimated Blood Volume Collection for Part 2* Priorities for Blood Sample Collections Adverse Events of Special Interest Severity Definition of Adverse Events | 93 |
| Table 16 | : Adverse Events of Special Interest | . 104 |
| Table 17 | : Severity Definition of Adverse Events | . 105 |
| Table 18 | : Clinical Measures Enacted Upon Increasing Severity of ECHO Findings | . 108 |
| | 90,00 | |
| Figure 1: | ; Study Schema | 50 |
| This docu | Priorities for Blood Sample Collections | |


# **SIGNATURE OF SPONSOR**

| Study Number: | ZX008-1601<br>PA 4.0(Japan)<br>25 July 2022 |
|---|---|
| Sponsor's Responsible Officer: Signature | A Two-Part Study of ZX008 in Children and Adults with Lennox-Gastaut Syndrome (LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures in Children and Adults with LGS, Followed by Part 2: An Open-label extension to Assess Long-Term Safety of ZX008 in Children and Adults with LGS Zogenix International Limited A wholly owned subsidiary of UCB Biosciences, Inc. 4000 Paramount Pkwy, Morrisville, NC 27560, USA |
| allot be and and | 28-juil2022 |
| Signature | Date (Day/Month/Year) |
| On behalf of the control of the cont | |
| UCB Biosciences Inc. | |


### SIGNATURE OF COORDINATING INVESTIGATOR

ZX008-1601 **Study Number:** PA 4.0 (Japan)

25 July 2022

A Two-Part Study of ZX008 in Children and **Study Title:** 

Adults with Lennox-Gastaut Syndrome

(LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures Aduh
... Open-lai
... m Safety of Z
... s with LGS

Children's Hospital Colora
Ansolutz Medical Campus
Aurora, CO 80045 in Children and Adults with LGS, Followed by Part 2: An Open-label extension to Assess Long-Term Safety of ZX008 in Children and

Children's Hospital Colorado


# SIGNATURE(S) OF THE PRINCIPAL INVESTIGATOR

**Study Number**: ZX008-1601
PA 4.0 (Japan)
25July 2022

Study Title: A Two-Part Study of ZX008 in Children and

Adults with Lennox-Gastaut Syndrome (LGS);
Part 1: A Randomized, Double-blind, Placebocontrolled Trial of Two Fixed Doses of ZX008
(Fenfluramine Hydrochloride) Oral Solution as
Adjunctive Therapy for Seizures in Children and
Adults with LGS, Followed by Part 2: An Openlabel Extension to Assess Long-Term Safety of
ZX008 in Children and Adults with LGS

I have read this study protocol, including all appendices. By signing this study protocol, I agree to conduct the clinical study, following approval by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), in accordance with the study protocol, the current International Conference on Harmonization (ICH) Guideline for Good Clinical Practice (GCP), and applicable regulatory requirements. I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

Name and affiliation to be filled out by the investigator

| Principal Investigator | 7 01 |
|------------------------|------|
| (Name & Affiliation): | O |
| ing glice | |
| C/2, 20/2 | |
| 90, 01 | |
| .5 | |
| (U) | |

Signature Date (Day/Month/Year)


# LIST OF ABBREVIATIONS

| ABBREVIATION | DEFINITION |
|---|---|
| AE | Adverse Event |
| AEGI | Antiepileptic drug |
| AESI | Adverse Event of Special Interest |
| ANCOVA | Analysis of covariance |
| AS | Atonic seizure |
| AUC | Area under the concentration-time curve |
| AUC0-t | Area under the concentration-time curve from time zero to time=t |
| BID | bis in die; two times per day |
| BMI | Body Mass Index |
| BRIEF | Behavior Rating Inventory of Executive Function |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| Cavg•ss | Average plasma concentration |
| CBD | Cannabidiol |
| CFR | Code of Federal Regulations |
| CGI | Clinical Global Impression |
| C <sub>max</sub> | Maximum observed concentration determined directly from the |
| | concentration-time profile |
| CRF | Case report form |
| CS | Clonic seizures |
| Сур | Cytochrome p450 |
| dL | Deciliter |
| DS | Dravet syndrome |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram C |
| eCRF | electronic Case Report Form |
| EEG | electroencephalogram |
| EOS | End Of Study |
| EPAR | European Public Assessment Report |
| ET | Early Termination |
| FS | Focal seizure |
| FSH | Follicle Stimulating Hormone |
| GCP | Good Clinical Practice |
| GH | Growth Hormone |
| GMP | Good Manufacturing Practices |
| GTC | Generalized tonic-clonic seizure |
| HADS | Hospital Anxiety and Depression Scale |
| HIV CO | Human Immunodeficiency Virus |
| HR | Heart Rate |
| IB | Investigator's Brochure |
| ICF O | Informed Consent Form |
| ICH | International Council on Harmonization |
| IDSMC | Independent Data and Safety Monitoring Committee |
| IEC | Independent Ethics Committee |
| IGF-1 | Insulin-like Growth Factor-1 |
| ILAE | International League Against Epilepsy |
| IMP | Investigational Medicinal Product |
| IND | Investigational New Drug |
| ICAB | International Cardiology Advisory Board |
| | · |


| ABBREVIATION | DEFINITION |
|------------------|---------------------------------------------------------|
| IRB | Institutional Review Board |
| IU | International Unit |
| IWR | Interactive Web Response (System) |
| KD | Ketogenic diet |
| kg | Kilogram |
| Leiter-3 | Leiter International Performance Scale-Revised |
| LGS | Lennox-Gastaut syndrome |
| LH | Luteinizing Hormone |
| M | Maintenance period |
| MCDS | Mean change in number of seizures that results in drops |
| MCSF | Mean Convulsive Seizure Frequency |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mg/kg/day | Milligram per kilogram per day |
| Min | Minutes |
| mITT | Modified Intent-to-Treat |
| mL | Milliliter |
| MS | Myoclonic seizure |
| OLE | Open-label extension |
| PopPK model | Population Pharmacokinetic model |
| PK | Pharmacokinetics |
| PP | Per Protocol |
| QoL | Quality of Life |
| QOLCE | Quality of Life in Childhood Epilepsy |
| QTcF | corrected QT interval using Fredericia method |
| SAE | Serious Adverse Event |
| SAF | safety population |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SE | Status epilepticus |
| SMEI | Severe Myoclonic Epilepsy Of Infancy |
| STP | Stiripentol |
| SUDEP | Sudden Unexpected Death in Epilepsy |
| T+M | Titration plus Maintenance Periods |
| t <sub>1/2</sub> | Terminal half-life |
| TA | Tonic/atonic seizure |
| THC | Tetrahydrocannabinol |
| T <sub>max</sub> | Time to maximum concentration |
| TS | Tonic seizure |
| TSH O | Thyroid Stimulating Hormone |
| ULN | Upper Limit of Normal |
| USA | United States of America |
| USP | United States Pharmacopeia |
| VABS | Vineland Adaptive Behavior Scale |
| VNS | Vagal Nerve Stimulator/Stimulation |
| ZX008 | Fenfluramine Hydrochloride Oral Solution |


### STUDY SYNOPSIS

**Study Title:** A Two-Part Study of ZX008 in Children and Adults with Lennox-Gastaut Syndrome (LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures in Children and Adults with LGS, Followed by Part 2: An Open-label Extension to Assess Long-Term Safety of ZX008 in Children and Adults with LGS

Study Number: ZX008-1601

| Study Product: Fenfluramine Hydrochloric | de Oral Solution, ZX008 |
|---|---|
| Type of Study: | Indication Studied: |
| Part 1: Efficacy and safety study | Adjunctive therapy for seizures in Lennox- |
| Part 2: Long-term safety study | Gastaut syndrome (LGS) |
| <b>Phase of Development:</b> Phase III | Countries: North America, Europe, Japan, and |
| | Australia |

**Sponsor:** Zogenix International <u>Limited</u>

**Coordinating Investigator:** 

### **Estimated Duration of Individual Subject Participation:**

The duration of participation in the study for an individual subject in the double-blind study (Part 1) is expected to be up to 20 weeks. The duration of participation in the open-label extension (Part 2) is up to 72 months or until ZX008 is approved in a subject's country of residence and listed on a patient's health plan formulary, whichever occurs first. The total participation time is up to approximately 77 months. Regardless of whether subjects end participation early, do not continue with the open-label extension, or roll over to the open-label extension, all subjects who do not transition to commercial drug will have a follow-up visit 3 to 6 months after the last dose of study medication for final safety monitoring.

### **Objectives:**

The primary objective of Part 1 is the primary objective of the entire study.

#### Part 1

The primary objective of Part 1 is:

• To evaluate the effect of ZX008 0.8 mg/kg/day versus placebo as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with Lennox-Gastaut syndrome (LGS) based on the change in frequency of seizures that result in drops between baseline and the combined Titration and Maintenance Periods (T+M)

The key secondary objectives of Part 1 are:

- To evaluate the effect of ZX008 0.2 mg/kg/day versus placebo as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with LGS based on the change in frequency of seizures that result in drops between baseline and T+M
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the proportion of subjects who achieve a  $\geq$ 50% reduction from baseline in the frequency of seizures that result in drops
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the Clinical Global Impression Improvement rating, as assessed by the Principal Investigator

See Statistical Methods (Section 10.1.5.1) for hierarchical testing procedure.


Additional secondary efficacy objectives of Part 1 are:

- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
  - Change in the frequency of all countable motor seizures between baseline and T+M (countable seizures include: generalized tonic-clonic seizures [GTC], tonic seizures [TS], clonic seizures [CS], atonic seizures [AS], tonic/atonic seizures [TA], clearly recognizable focal seizures [FS], and myoclonic seizures [MS] that result in a drop)
  - Change in the frequency of all countable seizures (ie, motor and non-motor) between baseline and T+M
  - Change in frequency of seizures that result in drops between baseline and the Maintenance Period (M)
  - Change in the frequency of countable motor seizures that do not result in drops between baseline and M
  - The proportion of subjects who achieve a worsening or no change (i.e ≤ 0% reduction), >0%, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizure freedom" (ie, 0 or 1 seizures) between baseline and T+M, and baseline and M, in all countable motor seizures (GTC, TS, AS, TA, FS, MS with a drop); in countable motor seizures that do not result in drops; and in all seizures that result in drops
  - Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
  - Longest interval between seizures that result in drops
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
- Clinical Global Impression Improvement rating, as assessed by the parent/caregiver The safety objectives of Part 1 are:
  - To evaluate the safety and tolerability of ZX008 0.2 and 0.8 mg/kg/day versus placebo with regard to adverse events (AEs), laboratory parameters, physical examination, neurological examination, vital signs (blood pressure, heart rate, temperature, and respiratory rate), electrocardiograms (ECG), echocardiograms (ECHO), body weight, and BMI
  - To evaluate the change from baseline in cognition using age-appropriate Behavior Rating Inventory of Executive Function (BRIEF)

The pharmacokinetic (PK) objective of Part 1 is:

• To evaluate the PK of ZX008 0.2 and 0.8 mg/kg/day at steady state in subjects <18 years and ≥18 years with LGS using a non-compartmental analysis; and obtain exposure data that will be used in population pharmacokinetic (PopPK) analysis, the results of which will be reported separately..

The exploratory objectives of Part 1 are:

- To compare the ZX008 0.2 and 0.8 mg/kg/day doses on primary, secondary and safety endpoints
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
  - The frequency of rescue medication usage
  - The incidence of medical services used to treat seizures
  - The incidence of status epilepticus
  - The change from baseline in behavior using the Vineland Adaptive Behavior Scale (VABS) (Cohort A)
  - The change from baseline in QoL using the Quality of Life in Childhood Epilepsy (QOLCE)
     Assessment
  - The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory
  - The change from baseline in affective symptoms of the parent/caregiver using the Hospital Anxiety and Depression Scale (HADS)


#### Part 2

The primary objective of Part 2 is:

 To assess the long-term safety and tolerability of ZX008 in children and adults with LGS with regard to adverse events (AEs), laboratory parameters, physical examination, neurological examination, suicidality, cognition (BRIEF), vital signs (blood pressure, heart rate, temperature, and respiratory rate), electrocardiograms (ECG), echocardiograms (ECHO), body weight, and BMI.

The secondary objectives of Part 2 are:

- To assess the effect of ZX008 relative to the baseline on the following effectiveness measures:
  - The change in the frequency of seizures that result in drops
  - The change in the frequency of all countable motor seizures (GTC, TS, CS, AS, TA, FS, MS with a drop)
  - The change in the frequency of all countable seizures
  - The proportion of subjects who achieve a worsening or no change (ie, ≤0% reduction),>0%, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizure freedom" (ie 0 or 1 seizures) in frequency of all countable seizures that result in drops, countable motor seizures that do not result in drops, all countable motor seizures, all countable seizures that do not result in drops
  - Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
  - Longest interval between seizures that result in drops
- To evaluate the effect of ZX008 on the following endpoints:
  - Clinical Global Impression Improvement rating, as assessed by the Principal Investigator
  - Clinical Global Impression Improvement rating, as assessed by the parent/caregiver

The exploratory objectives of Part 2 are:

- To determine the incidence of the following on subjects receiving ZX008:
  - The incidence of medical services used to treat seizures
  - The incidence of status epilepticus
  - The use of rescue medication
- To assess the effect of ZX008 on the following measures:
  - The change from baseline in QoL using the QOLCE
  - The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory
  - The change from baseline in affective symptoms of the parent/caregiver using the Hospital Anxiety and Depression Scale (HADS)

#### Methodology:

This is an international multicenter study being conducted in two parts. Up to approximately 80 study sites in North America, Europe, Japan, and Australia are initially planned to participate. Part 1 is a double-blind, parallel-group, placebo-controlled, study to assess the efficacy and safety of two doses of ZX008 when used as adjunctive therapy for seizures in children and adult subjects with LGS. The study will include 2 cohorts: Cohort A will include randomized subjects from North America, Europe,


and Australia; Cohort B will include randomized subjects from Japan only. The primary study endpoint is assessed from Part 1 Cohort A data. The primary analysis will be conducted when the last subject in Cohort A has completed Part 1. Cohort B will be analyzed independently with an interim analysis occurring after the last subject in Cohort B completes 12 months in Part 2 and a final analysis when the last subject in Cohort B completes Part 2. Part 2 will be an open-label, flexible-dose extension for subjects completing Part 1 of the study.

Part 1 will consist of a 4-week baseline, 2-week titration, 12-week maintenance, and 2-week taper or transition period. The 4-week Baseline Period will consist of the establishment of initial eligibility during a screening visit to include an assessment of cardiac parameters (ECG and ECHO), followed by an observation period where subjects will be assessed for baseline seizure frequency based on recordings of daily seizure activity entered into a diary. Upon completion of the Baseline Period, subjects who qualify for the study will be randomized (1:1:1) in a double-blind manner to receive 1 of 2 doses of ZX008 (0.2 mg/kg/day, 0.8 mg/kg/day; maximum dose: 30 mg/day [or 0.5 mg/kg/day] maximum 20 mg/day, for subjects taking concomitant stiripentol (STP)]) or placebo. Randomization will be stratified by weight (<37.5 kilograms [kg],  $\ge 37.5$  kg) to ensure balance across treatment arms, and at least 25% of subjects will be in each weight group. All subjects will be titrated to their blinded randomized dose over a 2-week Titration Period. Following titration, subjects will continue treatment at their randomly assigned dose over a 12-week Maintenance Period. Total treatment time from the beginning of the Titration Period through the end of the Maintenance Period is 14 weeks. Subjects will have ECG and ECHO assessments at weeks 6 and 14 during the Maintenance Period. At the end of the Maintenance Period (or early discontinuation), all subjects will undergo a blinded 2-week taper or transition period (Post-Dosing Follow-Up) depending on whether they exit the study or are enrolled in Part 2, the long-term open-label extension, respectively. A follow-up ECG and ECHO will be performed 3-6 months after study drug discontinuation for early termination, or for those subjects who complete the study but do not enter the open-label extension part. If there are any findings at the 3month post-dose follow-up, a second follow-up will be repeated at 6 months and then every 3 months until resolved or stabilized.

Part 2 is an open-label, long-term safety study of ZX008 for subjects who have successfully completed 14 weeks of treatment (titration + maintenance) in Part 1 and are candidates for continuous treatment for an extended period of time; subjects who have not completed the entire 14 weeks of treatment in Part 1 may be eligible to participate in Part 2 on a case-by-case basis and only following sponsor approval. Part 2 will consist of a 12-month Open-Label Extension (OLE) Treatment Period and a 2-week Post-Dosing Period. Thus, subjects who complete 12 months of OLE in Part 2 will have been treated with ZX008 for at least 70 weeks (including their participation in both Part 1 and Part 2). If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary. Up to -5 annual extensions can be applied, for a total treatment time of up to 72 months in the OLE. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk.

During Part 2 all subjects will be treated initially with 0.2 mg/kg/day for 1 month to assess effectiveness of this dose in all study subjects and determine the minimally effective dose. After 1 month at a dose of 0.2 mg/kg/day, the investigator may adjust the dose for each subject based on effectiveness and tolerability. Dose changes should be made in maximum increments of 0.2 mg/kg/day, to a maximum of 0.8 mg/kg/day (or 0.5 mg/kg/day for subjects taking concomitant STP) but not to exceed total dose of 30 mg/day (or 20 mg/day for sujects taking concomitant STP). During


the 12-month OLE subjects will have ECG and ECHO assessments at months 1, 3, 6, and 9, and at the end of study visit. In the event the OLE is extended, subjects will continue to have ECG (if clinically indicated) and ECHO assessments every 6 months until the end of their participation in the study.

A follow-up ECG and ECHO will be performed at 3 and 6 months after study drug discontinuation for early termination and for those subjects who complete Part 2. If there are any findings at a post-dose follow-up, another follow-up will scheduled every 3 months until resolved or stabilized. Subjects who transition to commercially available ZX008 will not return for these follow-ups, but must have an ECHO within 3 to 6 months of the transition date and will have follow-up ECHOs within required timeframs while on commercial drug supply.

In both Part 1 and the first 12 months of Part 2, parents/caregivers will use a diary every day to record the number of seizures, type of seizures, time and duration of seizures, whether the seizure resulted in a drop, dosing of study drug, and use of rescue medication. Seizures that result in a drop are defined as seizures involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the subject's head hitting a surface or that could have led to a fall or injury, depending on the patient's position at the time of the seizure.

A schedule of assessments for Part 1 is provided in Table 1 and for Part 2 in Table 2.

**External Individuals and Committees:** The ZX008 clinical program will employ an Independent Data and Safety Monitoring Committee (IDSMC) that will be responsible for safety oversight. A separate International Cardiology Advisory Board (ICAB) advises the Sponsor on matters of cardiac safety of the ZX008 clinical trials. ECGs and Doppler ECHOs will be centrally read and interpreted under blinded conditions using pre-specified criteria, and if necessary, with review by the ICAB.

#### **Number of Subjects:**

Approximately 340 subjects will be screened and approximately 250 subjects will be randomized into Part 1 Cohort A, and at least 30 and up to 50 subjects will be randomized into Part 1 Cohort B. The number of screened subjects may exceed 340 depending on the screen fail rate. Only subjects that participated in Part 1 are eligible for participation in Part 2. Each clinical site will not randomize more than a maximum of 15 subjects into Part 1 without prior consent from the sponsor.

### **Selection Criteria for Part 1**

**Inclusion Criteria:** All subjects must meet all of the following inclusion criteria to be enrolled into the study:

- 1. Subject is male or non-pregnant, non-lactating female, age 2 to 35 years, inclusive as of the day of the Screening Visit. Female subjects of childbearing potential must not be pregnant or breast-feeding. Female subjects of childbearing potential must have a negative urine or serum pregnancy test at screening. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control (see Section 4.4), which includes abstinence, while being treated on this study and for 90 days after the last dose of study drug.
- 2. Subject must have a diagnosis of Lennox-Gastaut syndrome, where seizures that result in drops are not completely controlled by current antiepileptic treatments. (Subjects without a formal diagnosis may still be enrolled after review and consultation between the Investigator and Sponsor, and in some cases, the Epilepsy Study Consortium. Final decisions on enrollment are at the discretion of the sponsor if all other criteria are met.)
- 3. Subjects must meet all of the following 4 criteria for Lennox-Gastaut syndrome, as defined in this protocol:
  - a. Onset of seizures at 11 years of age or younger.


- b. Multiple seizure types (must include TS or TA), including countable motor seizures that result in drops. Countable motor seizure types eligible for inclusion are: GTC, TS, CS, AS, FS with observable motor symptoms, and MS with a drop.
- c. Abnormal cognitive development.
- d. Evidence of EEG in the medical history that shows abnormal background activity accompanied by slow spike and wave pattern <2.5 Hz. (Acceptable evidence includes a copy of the EEG trace, EEG report, or physician note that appropriately describes the EEG findings.)
- 4. Subject must have had at least 8 drop seizures in the last 4 weeks prior to Screening (minimum of 4 drop seizures in the first two weeks and 4 in the last two weeks before Screening), by parent/guardian report to investigator or investigator medical notes
- Receiving at least 1 concomitant AED and up to 4 concomitant AEDs, inclusive. KD and VNS are permitted but do not count towards the total number of AEDs. Rescue medications for seizures are not counted towards the total number of AEDs.
- 6. All medications or interventions for epilepsy (including KD and VNS) must be stable for at least 4 weeks prior to screening and are expected to remain stable throughout the study.
- 7. Subject has been informed of the nature of the study and informed consent has been obtained from the legally responsible parent/guardian.
- 8. Subject has provided assent in accordance with Institutional Review Board (IRB)/Ethics Committee requirements, if capable.
- 9. Subject's parent/caregiver is willing and able to be compliant with diary completion, visit schedule and study drug accountability.

**Exclusion Criteria:** Subjects who meet any of the following exclusion criteria will not be enrolled into the study:

- 1. Subject has a known hypersensitivity to fenfluramine or any of the excipients in the study medication.
- 2. Subject's etiology of seizures is a degenerative neurological disease.
- 3. Subject has a history of hemiclonic seizures in the first year of life.
- 4. Subject only has drop seizures in clusters, where individual seizures cannot be counted reliably.
- 5. Subject has pulmonary arterial hypertension.
- 6. Subject has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke, or clinically significant structural cardiac abnormality, including but not limited to mitral valve prolapse, atrial or ventricular septal defects, patent ductus arteriosis (note: Patent Foramen Ovale or a bicuspid valve are not considered exclusionary).
- 7. Subject has current or recent history of Anorexia Nervosa, bulimia, or depression within the prior year that required medical treatment or psychological treatment for a duration greater than 1 month.
- 8. Subject has a current or past history of glaucoma.
- 9. Subject has had an anoxic episode requiring resuscitation within 6 months of the Screening Visit.
- 10. Subject has moderate or severe hepatic impairment. Asymptomatic subjects with mild hepatic impairment (elevated liver enzymes < 3x ULN and/or elevated bilirubin <2x ULN) may be entered into the study after review and approval by the Medical Monitor in conjunction with the sponsor, in consideration of comorbidities and concomitant medications.
- 11. Subject has severe renal impairment (estimated glomerlular filtration rate <30mL/min/1.73m<sup>2</sup>)
- 12. Subject is receiving concomitant therapy with any of the following: centrally-acting anorectic agents; monoamine-oxidase inhibitors; any centrally-acting compound with clinically


appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; other centrally-acting noradrenergic agonists, including atomoxetine; or cyproheptadine (see Appendix 1 for a list of prohibited medications). (Note: Short-term medication requirements for prohibted medications will be handled on a per case basis by the Medical Monitor.)

- 13. Subject has positive result on urine or serum tetrahydrocannabinol (THC) Panel or whole blood cannabidiol (CBD) at the Screening Visit.
- 14. Subject is taking felbamate for less than 1 year prior to screening and/or does not have stable liver function and hematology laboratory tests, and/or the dose has not been stable for at least 60 days prior to the Screening Visit.
- 15. Subject is known to be human immunodeficiency virus (HIV) positive.
- 16. Subject is known to have active viral hepatitis (B or C)
- 17. Subject is currently receiving an investigational product.
- 18. Subject has participated in another clinical trial within the past 30 days (calculated from that study's last scheduled visit). Participation in non-treatment trials will be reviewed by the medical monitor.
- 19. Subject is at imminent risk of self-harm or harm to others, in the investigator's opinion, based on clinical interview and responses provided on the Columbia-Suicide Severity Rating Scale (C-SSRS). Subjects must be excluded if they report suicidal behavior in the past 6 months as measured by the C-SSRS at Screening or Baseline, which includes suicidal ideation with intent and plan (Item #5). If a subject reports suicidal ideation on Item 4 without specific plan, and the investigator feels that the subject is appropriate for the study considering the potential risks, the investigator must document appropriateness for inclusion, and discuss with the parent/caregiver to be alert to mood or behavioral changes, especially around times of dose adjustment.
- 20. Subject is unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
- 21. Subject is institutionalized in a general nursing home (ie, in a facility that does not provide skilled epilepsy care).
- 22. Subject does not have a reliable caregiver who can provide seizure diary information throughout the study.
- 23. Subject has a clinically significant condition, including chronic obstructive pulmonary disease, interstitial lung disease, or portal hypertension, or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Screening Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

**Randomization Inclusion Criteria:** Subjects must meet all of the inclusion criteria and none of the exclusion criteria above and meet the following criteria in order to be randomized:

- 1. Subject has been approved for study inclusion by the Epilepsy Study Consortium.
- 2. Subject does not have an exclusionary cardiovascular or cardiopulmonary abnormality based on ECHO, ECG or physical examination and is approved for entry by the central cardiac reader. Exclusionary abnormalities include, but are not limited to:
  - a. Trace or greater mitral or aortic valve regurgitation in subjects ≤18 years of age
  - b. Mild or greater mitral or a ortic valve regurgitation in subjects >18 years of age
  - c. Possible signs of pulmonary hypertension with abnormal or greater than upper range of normal values
  - d. Evidence of left ventricular dysfunction (systolic or diastolic)
- 3. Subject demonstrates a stable baseline with  $\geq 2$  seizures per week resulting in drops during the 4-week Baseline Period.


4. Subject's parent/caregiver has been compliant with diary completion during the Baseline Period, in the opinion of the Investigator and Sponsor.

#### **Selection Criteria for Part 2**

To be included in Part 2:

- 1. Subjects must continue to meet the Selection Criteria for Part 1 (except for criteria related to seizure frequency). If a subject entering Part 2 does not meet Randomization Criteria 2 regarding cardiovascular abnormalities, Section 8.9.1 Follow-up of Cardiovascular Findings will be applied to determine eligibility to continue into Part 2.
- 2. All subjects must have satisfactorily completed Part 1 of the study in the opinion of the investigator and the sponsor.
- 3. Review of inclusion and exclusion criteria and written informed parental or guardian consent and assent of minors (if the subject is capable of providing assent) for Part 2 must be obtained before a subject can start any of the Part 2 Visit 15 procedures.
- 4. Subjects must, in the medical opinion of the Investigator, be candidates for continued treatment for an extended period of time with ZX008. Candidates for continuous treatment should not meet Discontinuation criteria listed in Section 4.5 and should not meet the following criteria:
  - a. Clinically meaningful worsening of seizures, judged by Investigator or subject/caregiver such that treatment outside of the protocol and other than ZX008 is assumed to be in the subject's best interest. A clinically meaningful worsening is an increase in frequency, severity or duration of existing seizures, or (in some cases) emergence of a new seizure type. Frequent or increased use of rescue medication may be considered indicative of worsening.
  - b. Clinically significant clinical laboratory findings (e.g. elevated ALT levels, decrease in platelet count, etc. that are CTCAE Grade 3 or higher) in subjects with no prior relevant history, that were not present during Baseline, are confirmed by a repeat test within a week, and not attributable to other concomitant medications.
  - c. Weight loss >15% during the T+M period that has not stabilized and is considered, in the opinion of the Investigator, detrimental to continuing treatment with ZX008.
- 5. Those subjects who do not complete the 12-week Maintenance Period of Part 1 may, on a case-by-case basis, be eligible for entrance after consideration of the circumstances of the early termination and the potential benefit-risk of continued participation in a ZX008 trial. The decision whether to permit participation in Part 2 for subjects who do not complete Part 1 resides solely with the sponsor, who will require a formal request for early Part 2 continuation to be made by the site investigator as well as an evaluation of risk/benefit. The sponsor may also consult with the ICAB and/or the IDSMC, and take into consideration evidence of the following for approval:
  - a. The subject is experiencing a worsening in condition that is not likely to be related to Part 1 treatment, in the opinion of the Investigator
  - b. The subject has progressed at least half-way through Part 1 (i.e. Visit 8)
    - The subject has been compliant with assessments and requirements of Part 1
  - d. The subject does not exhibit other contraindications to initiating open-label treatment

#### Study Product, Dose, and Mode of Administration:

ZX008 is supplied as an oral solution in concentrations of 1.25, 2.5, and 5 mg/mL. Subjects will be randomized to receive 1 of 2 doses of ZX008 (0.2 mg/kg/day, 0.8 mg/kg/day; maximum dose: 30 mg/day) or placebo. Study medication will be administered twice a day (BID) in equally divided doses. (Note that subjects taking concomitant STP will be randomized to 0.5 mg/kg/day, maximum


dose 20 mg/day, or equivalent volume of placebo. Subjects randomized to 0.5 mg/kg/day will be included in analyses with the subjects randomized to 0.8 mg/kg/day not taking STP.)

#### Reference Product, Dose, and Mode of Administration:

Matching ZX008 placebo is supplied as an oral solution.

#### **Duration of Treatment:**

In Part 1 all subjects will receive ZX008 or matching placebo for up to approximately 16 weeks (Titration Period=2 weeks; Maintenance Period=12 weeks; Taper/Transition Period=2 weeks). At the end of the 12-week Maintenance Period, eligible subjects may enroll into Part 2, the open-label extension, after completing a 2-week transition period with blinded study medication. Subjects who enroll in Part 2 will have the option to receive ZX008 for up to 72 months (plus a 2-week taper at the end of the open-label extension), or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever comes first. Subjects who do not enroll in the open-label extension will undergo a taper off of study medication (doses will be administered in a blinded fashion similar to the titration, ie, doses will be decreased in 4-day increments). Follow-up cardiovascular safety assessments, including ECG and ECHO, will be performed following the last dose of study medication for all subjects that do not transition to commercial drug, regardless of whether they complete the entire study or terminate early, unless the subject was known to be taking placebo (ie, blind was broken). These follow-ups will occur 3 months following the last dose of study medication for any subject taking the medication for 2-13 weeks, and 3 and 6 months following the last dose for any subject taking the medication for >13 weeks. If there are any findings at a post-dose follow-up, another follow-up will scheduled every 3 months until resolved or stabilized. Subjects who transition to commercially available ZX008 will not return for a follow-up after EOS/ET or a cardiac follow up after last dose but must have had an ECHO within 3 to 6 months before the transition date and will have follow-up ECHOs within required timeframe while on commercial drug supply.

#### **Criteria for Evaluation:**

### Efficacy:

The efficacy endpoints for Part 1 of the study are

### Primary Endpoint:

Percent change from baseline in the frequency of seizures that result in drops in the combined Titration and Maintenance Periods (T+M) in the ZX008 0.8 mg/kg/day group compared to the placebo group.

Key Secondary Endpoints:

- Change from baseline in the frequency of seizures that result in drops in T+M in the ZX008
   0.2 mg/kg/day group compared to the placebo group.
- Proportion of subjects who achieve a ≥50% reduction from baseline in the frequency of seizures that result in drops comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo
- Proportion of subjects who achieve clinically-meaningful improvement (much or very much improved) in the Clinical Global Impression Improvement as assessed by Principal Investigator comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo.

Additional Secondary Endpoints:

- Change from baseline in the frequency of all countable motor seizures in T+M in the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo
  - Countable motor seizures include: generalized tonic-clonic seizures [GTC], tonic seizures [TS], clonic seizures [CS], atonic seizures [AS], tonic/atonic seizures [TA], clearly recognizable focal seizures [FS], and myoclonic seizures [MS] that result in a drop


- Change from baseline in the frequency of countable seizures that result in drops
- Change from baseline in the frequency of seizures that result in drops between baseline and the Maintenance Period (M)
- Change from baseline in frequency of countable seizures that do not result in drops
- Proportion of subjects who achieve a worsening from baseline (ie <= 0% reduction), or >0%, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizure freedom" (ie 0 or 1 seizures) between baseline and T+M, and baseline and M, in all countable motor seizures; in countable motor seizures that do not result in drops; in all countable seizures that do not result in drops; and in all seizures that result in drops
- Number of seizure-free days in the baseline, M and T+M period defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
- The longest interval (days) between seizures that result in drops comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo
- Clinical Global Impression Improvement as assessed by the parent/caregiver

The efficacy endpoints for Part 2 of the study are:

- The change from baseline in the frequency of seizures that result in drops.
- The change from baseline in the frequency of all countable motor seizures (GTC, TS, CS, AS, TA, FS, MS with a drop)
- The change from baseline in the frequency of all countable seizures
- The proportion of subjects who achieve a worsening from baseline (ie <= 0% reduction), or >0%, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizure freedom" (ie 0 or 1 seizures) from baseline in frequency of all countable seizures that result in drops, countable motor seizures that do not result in drops, all countable motor seizures, all countable seizures, and all countable seizures that do not result in drops
- Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
- Clinical Global Impression Improvement rating, as assessed by the Investigator.
- Clinical Global Impression Improvement rating, as assessed by the parent/caregiver.

#### Safety:

The safety endpoints for Part1 and Part 2 of the study are:

- AEs
- Laboratory safety (hematology, chemistry, urinalysis)
- Vital signs (blood pressure, heart rate, temperature, and respiratory rate)
- Physical examination
- Neurological examination
- BRIEF to measure changes in cognition of the subject
- Columbia Suicidality Severity Rating Scale (C-SSRS)
- 12-lead ECGs
- Doppler ECHOs
- Body weight and BMI

#### Exploratory:

The exploratory endpoints for Part 1 and Part 2 of the study are:

• Incidence of status epilepticus


- Incidence of rescue medication usage
- Number of days rescue medication used
- Incidence in use of medical services to treat seizures
- The change from baseline in behavior using the Vineland Adaptive Behavior Scale (VABS) (Part 1 Cohort A only)
- The change from baseline in quality of life using the QOLCE
- The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory
- The change from baseline in affective symptoms of parent/caregiver using the HADS scale.

#### Pharmacokinetics:

Steady-state plasma fenfluramine and norfenfluramine PK parameters (maximum and minimum plasma concentration (C<sub>min ss</sub>, C<sub>max ss</sub>) and area under the concentration time curve from time zero to time=t and time=24 hours (AUC0-t, AUC0-24) after administration of ZX008 derived using a population pharmacokinetic model.

### **Sample Size Determination:**

The sample size for Part 1 Cohort A was estimated under the assumption that adding ZX008 at 0.8 mg/kg/day to current therapy will lead to a mean decrease in the frequency of drop seizures that is 30 percentage points lower than adding placebo to current therapy. The variability expected in the trial was estimated from the confidence intervals reported in a Phase 3 trial of clobazam for patients with Lennox-Gastaut syndrome (Ng, 2011) leading to an assumption that the SD is 50%. Under these assumptions, and using a Wilcoxon rank-sum test to approximate the primary analysis, a sample size of 63 subjects per treatment group affords 90% power to detect a difference between groups that is significant at the  $\alpha$ =0.05 level. Assuming a 20% drop-out rate prior to the start of the maintenance period yields a requirement for an additional 16 subjects per group for a total of 79 subjects per treatment group. Similar calculations for the 0.2 mg/kg/day ZX008 group lead to a total required sample size of 237. The number of subjects randomized into Part 1 Cohort A is estimated to be approximately 250 due to the long baseline period. The sample size of 10 to 15 subjects per treatment group in Cohort B is expected to provide a descriptive assessment of whether the treatment effect in Japanese subjects is similar to that observed in Cohort A subjects from the rest of the world.

#### **Statistical Methods:**

#### Part 1

The primary analyses of the study will be performed on data from Part 1 Cohort A after the last subject enrolled in Cohort A has completed the last study visit of Part 1. Data from Part 1, Cohort B will be analyzed independently after the last subject in Cohort B completes Part 1. An interim analysis of Part 2 will be performed after all Cohort B subjects complete 12 months in Part 2. A secondary analysis will be conducted after the last Cohort B subject has enrolled and completed the last study visit of Part 2. Analysis results for Part 1 from Cohort A and Cohort B may be compared through descriptive statistics, and if reasonable, some analyses may be performed using data from Cohort A and Cohort B combined. Subjects randomized to 0.5 mg/kg/day (ie, those taking concomitant STP) will be grouped with subjects randomized to 0.8 mg/kg/day for all efficacy analyses.

Primary Efficacy Analysis: The primary efficacy endpoint for Part 1 is the percent change in frequency of seizures that result in drops (DSF: drop seizure frequency) per 28 days between the T+M and Baseline periods in Cohort A. The DCF will be calculated from all available data collected during the Baseline and treatment periods without imputation. The percent change in DSF will be calculated as the change in DSF between T+M and Baseline / DSF during Baseline× 100. Both the mean and median percent change in DCF frequency will be presented. The primary endpoint will be assessed using an non-parametric rank analysis of covariance (ANCOVA) with treatment and weight groups (<37.5 kg,  $\ge 37.5 \text{ kg}$ ) as factors, and with Baseline MCDS as a covariate rank baseline DSF as a


covariate, and rank percent change in DSF from baseline as the response variable. The primary analysis will compare the ZX008 0.8 mg/kg/day group to the placebo group at the alpha=0.05 level of significance. The difference between the ZX008 0.8 mg/kg/day and placebo groups in percent change in DSF, and its 95% confidence interval, will be estimated using the Hodges-Lehmann method. As a sensitivity analysis, the primary endpoint will also be analyzed using a parametric ANCOVA that incorporates treatment group and weight group as factors, log baseline DSF as a covariate; and log DSF during T+M as the response variable. Another sensitivity analysis will use a Wilcoxon rank-sum test to compare the ZX008 0.8 mg/kg/day group to the placebo group. Part 1 Cohort B will be analyzed using analogous methods.

A key secondary analysis will compare the ZX008 0.2 mg/kg/day group to the placebo group on percent change in DSF using the same method as the primary analysis. Other key secondary analyses will compare the ZX008 0.8 and 0.2 mg/kg/day groups to the placebo group on the proportion of subjects who achieve a ≥50% reduction from baseline in DSF. The analyses will utilize independent logistic regression models that incorporate the same factors and covariate as the primary analysis. Two other key secondary analyses will compare both ZX008 dose groups (independently) to placebo on the proportion of subjects assessed by the Principal Investigator as minimally, much, or very much improved on the Clinical Global Impression – Improvement (CGI-I). The comparisons will employ separate Cochran-Mantel-Haenszel tests (CMH) stratified by weight strata. A serial gatekeeper strategy will be used to maintain the Type 1 error rate at α=0.05 across the family of analyses that support the primary and key secondary objectives.

#### Safety

All safety data will be appropriately analyzed by treatment group. The number and percentage of subjects with AEs will be displayed by body system and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). Summaries in terms of severity and relationship to study drug will also be provided. Adverse Events of Special Interest (AESI) and Serious AEs (SAEs) will be summarized separately in a similar manner. Laboratory tests, vital signs, physical examinations, neurological examinations, ECG, Doppler echocardiogram, C-SSRS, Tanner Staging results, etc, will be summarized appropriately, by treatment. All safety summaries will be based on the Safety Population.

#### Pharmacokinetics

Model derived plasma PK parameters (C<sub>max\_ss</sub>, C<sub>min\_ss</sub>, AUC<sub>0-t</sub>, AUC<sub>0-24</sub>) will be summarized descriptively by treatment group, when sufficient data are available. A PopPK model of fenfluramine, previously developed using data from healthy adults and pediatric patients with Dravet syndrome, will be updated to include the fenfluramine and norfenfluramine concentrationtime data collected during the Maintenance Period of Part 1. This model will be informed by all relevant data available at the time of data collection (both adults and pediatrics). The results from the PopPK modeling will be reported separately and conducted according to a separate SAP.

#### Part 2

The primary objective of Part 2 is to assess the long-term safety and tolerability of ZX008 in children and adults with LGS with regard to AEs, laboratory parameters, physical examination, neurological examination, vital signs, ECG, ECHO, body weight, and BMI.

The number and percentage of subjects who experience treatment emergent AEs will be displayed by body system and preferred term using MedDRA. Summaries in terms of severity and relationship to study drug will also be provided. SAEs will be summarized separately in a similar manner. Laboratory tests, vital signs, physical examinations, neurological examinations, ECG, ECHO, cognition and body weight will be summarized using appropriate methods.

Effectiveness will be assessed by the change from baseline (prior to randomization into Part 1) in DSF. The DSF per 28 days will be calculated as the number of seizures that result in drops divided by the number of days in the period and multiplied by 28. The change in DSF during the first 12 months of


a prior to Par A prio


Table 1. Schedule of Assessments: Part 1

| Visit Number | Study Assessments – PART 1 | Baseline Period <sup>a</sup> Titration + Maintenance Period | | | | | | | | | Cardiac | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table Tabl | | | | | | | | | | | | | | | |
| Choncy C | Visit Number | Screening | | | T | 1 | eriod | | | | | 70 | | Dosingl | up <sup>c</sup> |
| Informed Consent (subject and parent/caregiver) | | 1 | _ | 3 | | | 6 | | 8 | | A | | + 12 | 13 | 14 |
| Inclusion/Exclusion Criteria X | Study Day | -28 | -15 | -1 | 1 | 4, 8 | 15 | 29 | 43 | 57 | 71 | 85 | | 113 | 197 |
| Inclusion/Exclusion Criteria | Informed Consent (subject and | X | | | | | | | | X | 0 | | | | |
| Demographics | parent/caregiver) | | | | | | | | | (0) | 10 | _ | (Part 2) | | |
| Medical/Neurological History X | | X | | X | | | | | | 1 | | | | | |
| Epilepsy history | Demographics | | | | | | | | 0 | | S | | | | |
| Review retrospective seizure X | Medical/Neurological History | | | | | | | | | | | | | | |
| Depth Dept | Epilepsy history | | | | | | | | | J.(O | | | | | |
| Prior Medication, including AEDs | | X | | | | | 7 | 5. | 3 | 0), | | | | | |
| Physical Examination, complete X | | X | | X | | | Y | (V) | | | | | | | |
| Physical Examination, abbreviated | | X | | | | _( | ) | X. | 10 | | | | X | | Ontional |
| Abbreviated Neurological Examination, X | | | | | | | Xm | | Xm | | Xm | | | | |
| Neurological Examination, X | | | | | | | | | | | | | | | |
| complete Neurological Examination, abbreviated X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X <td></td> <td>X</td> <td></td> <td></td> <td>•</td> <td></td> <td>S</td> <td></td> <td></td> <td></td> <td></td> <td></td> <td>X</td> <td></td> <td></td> | | X | | | • | | S | | | | | | X | | |
| Neurological Examination, abbreviated | | | | | | | 11 | 2 | | | | | | | |
| Abbreviated | | | | X | 0 | 9 | Xm | | Xm | | Xm | | | | |
| Weight | | | | ` | | | | | | | | | | | |
| Weight | Vital signs | | | X | 7 、 | | X | | X | | X | | X | | |
| 12-lead ECG | Weight | | | X | | | X | | X | | X | | | | |
| Doppler ECHO | Height | | | | -0 | | | | | | | | | | |
| Urine or Serum Pregnancy Test $X^c$ | 12-lead ECG | X | | X | 5 | 0.1 | | | | | | | | | |
| Clinical laboratory evaluation (hematology/ chemistry/urinalysis°, etc) Plasma sample for ZX008 PK Plasma sample for background AEDs Urine or serum THC Panel XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Doppler ECHO | X | | | <b>)</b> | 10 | | | Xd | | | | Xd | | Xc |
| Clinical laboratory evaluation (hematology/ chemistry/urinalysis°, etc) Plasma sample for ZX008 PK Plasma sample for background AEDs Urine or serum THC Panel XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Urine or Serum Pregnancy Test | Xe | | Xe | ~ | 4 | | | Xe | | | | | | |
| Plasma sample for ZX008 PK Plasma sample for background AEDs Urine or serum THC Panel X X X X X X X X X X X X X X X X X X | | X | | X | | , | | | X | | | | X | | |
| Plasma sample for background AEDs Urine or serum THC Panel X X X X X X X X X X X X X | | | × | | ,0, | | | | | | | | | | |
| AEDs Urine or serum THC Panel X X X X X X X X X X X X X X X X X X | | | $\sim$ | $^{\circ}$ $^{\circ}$ | - | | | | | | | | | | |
| Urine or serum THC Panel X X X X X X X X X X X X X X X X X X X | | | | $X^{g}$ | | | Xg | | X | | Xg | | Xg | | |
| Whole blood CBD X X X X X X X X X X X X X X X X X X X | | | 1 | (Q. | | | | | | | | | | | |
| Tanner Staging (for subjects >7 to 18 years old) Subject Diary D R C/R/D R C | | X | | | | | | | | | | | | | |
| 18 years old) Subject Diary D R C/R/D | | Х | $\cdot$ .O | | | | | | X | | | | | | |
| Subject Diary D R C/R/D R C/R | | 0, | 111 | X | | | | | | | | | X | | |
| Epilepsy genotype panel (optional) | | (2) | <b>O</b> | a/= /= | | | G/F '= | | | | 0.5.5 | L | a = -1 | | |
| (optional) | | D | R | C/R/D | | R | C/R/D | R | | R | C/R/D | R | C/R/D <sup>h</sup> | C/R | |
| | | 0// | | | | | | | X | | | | | | |
| | | ΔY, | | D | | Ri | C/R/D | R | C/R/D | R | C/R/D | R | C/R/Dh | C/R | |

Confidential

| Study Assessments – PART 1 | Basel | ine Perio | eriod <sup>a</sup> Titration + Maintenance Period | | | | | | | | Cardiac | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | Screening | | Random-<br>ization | Ti | tration Pe | eriod | | Main | tenance P | Period | 20 | EOS/<br>ET <sup>b</sup> | Post-<br>Dosing <sup>1</sup> | Follow-<br>up <sup>c</sup> |
| | 1 | 2<br>(Phone) | 3 | | 4, 5<br>(Phone) | 6 | 7<br>(Phone) | 8 | 9<br>(Phone) | 10 | 11<br>(Phone) | 12 | 13 | 14 |
| Study Day | -28 | -15 | -1 | 1 | 4, 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | 197 |
| C-SSRS | X | | X | | | X | | X | | X | .01 | X | | |
| Clinical Global Impression - | | | | | | X | | X | | X | | X | | |
| Improvement (assessed by | | | | | | | | | | , ~ | ) | | | |
| parent/caregiver) | | | | | | | | | 76 | 1/1/ | | | | |
| Clinical Global Impression - | | | | | | X | | X | | $c_{X}$ | | X | | |
| Improvement (assessed by | | | | | | | | ~( | ) ( | | | | | |
| investigator) | | | | | | | | 0, | . 0 | • | | | | |
| HADS (Effect of | | | X | | | 1 | | 1 | | | | X | | |
| parent/caregiver) | | | | | | 7 | \$ | $\sim$ $\sim$ | <b>7</b> | | | | | |
| BRIEF | | | X | | | | | | | | | X | | |
| QOLCE | | | X | | | | X | 10 | | | | X | | |
| Zarit Burden | | | X | | | | | X | | | | X | | |
| Randomize subject | | | Xn | | ) | | · ( | | | | | | | |
| First Day of Study Drug<br>Administration | | | $X^{j}$ | X <sup>j</sup> | 5 | 10h | 5 | , | | | | | | |
| Daily Diary Completion | | 1 | | | 1 6 | $\mathcal{O}$ | X | | | | | | 1 | |
| Concomitant Medication | | | • | W. | | ,(C | ) | | X | | | | | |
| Adverse events | | • | | ) | XO | 25, | X | | | | | | | |
| Adverse events of special interest | | | ~ | 2 | | -//- | X | | | | | | | $X^k$ |

AED=antiepileptic drug; BMI=body mass index; C=Collect; CBD=cannabidiol; D=Dispense; ECG=electrocardiogram; EOS=end of study; ET=early termination; HADS=Hospital Anxiety and Depression Scale; BRIEF=Behavior Rating Inventory of Executive Function: OoL=quality of life: R=Review

- The Baseline Period is comprised of the initial screening for the study and the assessment of baseline seizure activity recorded daily in the diary. The procedures to be completed at the Screening visit may be completed in a single day or split so that they are
- Subjects who are discontinued early and those who complete the study and choose not to enroll in the separate open-label extension will be tapered off study medication over an up to 2-week period.
- The safety follow-up visit will be conducted for subjects who either terminate early from Part 1, or who complete Part 1 but do not enter Part 2. Standard follow-up visits should occur 3 and 6 months after the last dose. If there are any findings at the last post-dose follow-up, a follow-up visit will be repeated every 3 months until resolved or stabilized.
- The Visit 8 ECHO must be performed any time between Study Day 40 and Study Day 54. The Visit 12 ECHO must be performed any time between Study Day 90 and Study Day 113; if a subject discontinues early from the study, the ECHO should be scheduled as soon as practical. If the Study Day 43 ECHO was completed 

  30 days prior to early termination, the Visit 12 ECHO will not be performed provided the parent/guardian agrees to bring the subject to the clinic for the cardiac follow-up visit.
- Females of child-bearing potential
- Plasma sample for pharmacokinetic assessment will be conducted prior to the dose at Visit 8 and 1, 2, and 4-6 hours after dose administration.
- Plasma sample for assessment of background AED(s) will be conducted prior to the dose of AED(s) at Visits 3, 8 and 12 (Visits 6 and 10 only if clinically indicated). Plasma sample may be collected after the morning dose of AED(s) are taken, if preferable, as long as the time of last dose is accurately recorded.
- Study drug/diary dispensed for the Transition Period for subjects entering the open-label extension and for the Taper Period for subjects exiting the study.
- Site personnel will review study medication dosing procedure (titration) with parent/caregiver.
- Study drug administration begins in the clinic on Study Day 1. Study Day 1 is considered the first day of dosing, even though subjects received an in-clinic dose on Study Day -1. The first dose taken in the clinic will be recorded in the eCRF, but not the subject diary; the next dose on the morning of Study Day 1 will be the first entry in the subject's diary. Only adverse events related to cardiac safety will be collected at this visit.
- Visit 13 may be conducted as a phone call, provided diaries and study medication are returned by this time.
- An abbreviated physical and/or neurological examination to be conducted as appropriate based on last exam and reported AEs.
- Randomization should not occur prior to receiving approval from the Epilepsy Study Consortium and ERT ECHO results.
- Urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability.

Table 2. Schedule of Assessments: Part 2 Cohort B only

After Visit 26/ Month 24 (or a later visit if V26/ Month 24 visit has already been performed at the time of Protocol Amendment 4.0 approval), in clinic study visits will occur every 6 months until ZX008 is approved by the subject country of residence and listed on the patient health plan formulary. A phone visit will be performed between in clinic visits (with a 3-month interval). During the phone visits, only a review of concomitant medications, adverse events and adverse events of special interest will be performed.

| Last Visit Number/Study Month pre approval of Amendment 4.0 | Next In Clinic Visits to be Scheduled (until ZX008 approval by health authority) -Every 6 months- | | | | |
|---|---|---|---|---|---|
| Visit 26 / Month 24 | Visit 28/M30 | Visit 30/M36 | Visit 32/M42 | Visit 34/M48 | Visit 36/M54 |
| Visit 27 / Month 27 | Visit 29/M33 | Visit 31/M39 | Visit 33/M45 | Visit 35/M51 | |
| Visit 28 / Month 30 | Visit 30/M36 | Visit 32/M42 | Visit 34/M48 | Visit 36/M54 | |
| Visit 29 / Month 33 | Visit 31/M39 | Visit 33/M45 | Visit 35/M51 | | |
| Visit 30 / Month 36 | Visit 32/M42 | Visit 34/M48 | Visit 36/M54 | | |
| | VISIT 30 / IVIOITITI 30 VISIT 32/1448 VISIT 30/14134 | | | | |

| Study Assessments – PART 2 | | Post-<br>Dosing | Cardiac Follow-up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | Visit 15 <sup>a</sup> | Visit 1 | 6 <sup>b</sup> | Visits 17-21 | Visit 22 | Visits 23-4 | 41 (Months | Visit 42 <sup>c</sup> | Visit 43 | Visit 44 and 45 |
| | | | | (Months 1, 2, | (Month 12) | 15, 18, 21, | , 24, 27, 30, | (EOS/ET) | | |
| | | | | <b>C3</b> , 6 and 9**) | | 33, 36, 39, | , 42, 45, 48, | | | |
| | | | | , 0' | | 51, 54, 57, | , 60, 63, 66, | | | |
| | | | -0. | | | | 9) | | | |
| OLE Study Day | 1 <sup>a</sup> | 15 | 70 | 30, 60, 90, | 360 | | , 630, 720, | 2160 | 2174 <sup>k,q</sup> | (3 and 6 months post |
| | | × | Y | <b>180</b> , and 270 | | | 990, 1080, | | | last dose) <sup>d,k</sup> |
| | | -0 | | | | | 60, 1350, | | | |
| | | | | 1 | | | 30, 1620, | | | |
| | | | <i>O</i> ; | | | | 300, 1890,<br>, 2070 | | | |
| | C | Clinic | Phone | | | Clinic | Phone | | | |
| Informed Consent | X | 2/0 | | | X** | X** | | | | |
| Entry Criteria | X | | | | | | | | | |
| Demographics | $X^a$ . ( | ,0 | | | | | | | | |
| Medical/Neurological History | Xa | | | | | | | | | |
| Epilepsy History | Xa | | | | | | | | | |
| Physical Examination, complete | $X^{\mathrm{a}}$ | | | | X | | | X | | X |
| Physical Examination, abbreviated | .0. | Xm | | Xm | | Xm | | | Xm | X |

Confidential

| Study Assessments – PART 2 | OLE Treatment Period** | | | | | | | | Post-<br>Dosing | Cardiac Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | Visit 15 <sup>a</sup> | Visit | : 16 <sup>b</sup> | Visits 17-21<br>(Months 1, 2,<br>3, 6 and 9**) | Visit 22<br>(Month 12) | | | Visit 42°<br>(EOS/ET) | Visit 43 | Visit 44 and 45 |
| Neurological Examination, complete | Xe | | | | X | | | X | | |
| Neurological Examination, abbreviated | | Xm | | X <sup>m</sup> | | X <sup>m</sup> | | , , , | X <sup>m</sup> | |
| Vital signs | X | X | | X | X | X | | X | | |
| Weight | Xa | X | | X | X | X | C | X | X | |
| Height | Xa | | | | X | 2,2 | , V- | X | | |
| 12-lead ECG | Xa | | | X | X | $X^q$ | .0 | Xq | | X |
| Doppler ECHO | Xa | | | $X^{f,g}$ | \X | Xg | XII | X | | X |
| Urine or Serum Pregnancy Testh | Xa | | | Xn | X | X | <i>D</i> - | X | | |
| Clinical laboratory evaluation (hematology/chemistry/urinalysis <sup>p</sup> , etc) | Xi | Xi | | X <sup>n</sup> | X | Xq | | Xq | | |
| Urine or serum THC Panel | Xa | | | Xn | X | 10 | | Xs | | |
| Whole blood CBD | Xa | | | Xn | X X | | | Xs | | |
| Plasma sample for background AEDs | | Xm | | Xn | X | Xq | | Xq | | |
| Tanner Staging (for subjects >7 to 18 years old) | Xa | | | X | X | | | Xs | | |
| C-SSRS | Xa | | | X | X | X | | X | | |
| CGI-I (assessed by parent/caregiver) | Xa | | | X | X | X | | X | | |
| CGI-I (assessed by investigator) | Xa | | | X | X | X | | X | | |
| Overall change in seizure frequency (assessed by investigator) | | | 8 | 00 00 | | Xr | | X <sup>r</sup> | | |
| HADS (Effect of parent/caregiver) | Xa | | | C X° | X | | | Xs | | |
| BRIEF | Xa | | | X° | X | | | Xs | | |
| OOLCE | Xa | | 0 | X° | X | | | Xs | | |
| Zarit Burden | Xa | | 5 | | X | | | Xs | | |
| Subject Diary | C/R/D | C/R/D | R | C/R/D | Xr | Xr | | C/R <sup>r</sup> | C/R | |
| Study Medication | C/R/D | C/R | R | C/R/D | C/R/D | C/R/D | | C/R/D | C/R | |
| Daily Diary Completion | | X | | J | | • | • | • | | |
| Concomitant Medication | Xa | | 7 | | X | | | | | |
| Adverse Events | Xa | OC | <u> </u> | | X | | | | | |
| Adverse events of special interest | X <sup>a</sup> O | | | | X | | | | | X <sup>l</sup> |

AED=antiepileptic drug; BMI=body mass index; C=Collect; CBD=cannabidiol; D=Dispense; ECG=electrocardiogram; EOS=end of study; ET=early termination; HADS=Hospital Anxiety and Depression Scale; BRIEF=Behavior Rating Inventory of Executive Function; QoL=quality of life; R=Review;

Use data collected at Visit 12 of Part 1.

At the discretion of the investigator, Visit 16 may be conducted as a phone visit.

Safety Follow-up visits will be conducted for subjects who terminate early from Part 2 and for those who complete Part 2. Standard follow-up visits should occur 3 and 6 months after the last dose. If there are any findings at a post-dose follow-up, a follow-up visit will be scheduled every 3 months until resolved or stabilized.

Use Part 1 Visit 12 information unless complete neurological examination is warranted based on significant changes in subject status.

| Study Assessments – PART 2 | | OLE Treatment Period** Post- Dosing | | | | | |
|---|---|---|---|---|---|---|---|
| Visit Number | Visit 15 <sup>a</sup> | Visit 16 <sup>b</sup> | Visits 17-21<br>(Months 1, 2,<br>3, 6 and 9**) | Visit 22<br>(Month 12) | Visits 23-41 (Months<br>15, 18, 21, 24, 27, 30,<br>33, 36, 39, 42, 45, 48,<br>51, 54, 57, 60, 63, 66,<br>69) | Visit 42°<br>(EOS/ET) Visit 43 | Visit 44 and 45 |

- f: ECHOs will be performed at Months 1, 3, 6, and 9.
- g: The Months 3, 6, 9, 12, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 & 72 ECHO may be performed any time within 3 weeks prior to the study visit. If a subject discontinues early from the study, the ECHO should be scheduled as soon as practical.
- h: Females of child-bearing potential
- i: For Visit 15, use data collected at Part 1 Visit 12 unless clinical laboratory evaluation is warranted based on significant changes in subject status. For Visit 16, clinical laboratory evaluation is optional based on subject status.
- i: Visit 20 only
- k: For subjects who are transitioning to commercial drug, do not initiate drug taper or conduct post-dosing and cardiac follow-up visits.
- Only adverse events related to cardiac safety will be collected at this visit.
- m: An abbreviated physical and/or neurological examination to be conducted as appropriate based on last exam and reported AEs.
- n: Visits 19, 20, and 21 (Months 3, 6, and 9) only.
- o: Visit 20 (Month 6) only
- Urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability.
- q As clinically indicated for subjects extending Part 2 participation past 12 months. Abnormal clinically significant findings must be reported as adverse events.
- r: Electronic diary is to be used the first 12 months of Part 2, and should be reviewed and collected on Visit 22 (for subjects continuing in Part 2 of the study) or Visit 42 (for subjects who do not continue in Part 2 of the study past 12 months). After 12 months in Part 2, seizure diaries are not required. Rather, based on discussions with the parent/caregiver, clinical evaluation, and review of any documentation provided by the caregivers, investigators will assess the percent improvement in seizure burden on a 5-point scale: <25%, ≥25%, ≥50%, ≥75%, 100% [ie, seizure-fee] improvement.
- s: Only applicable for subjects ending Part 2 participation within the first 12 months. Not applicable for subjects who completed Visit 22 and extended participation in Part 2.
  - \*\* If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study. Up to 5 annual extensions can be applied, for a total treatment time of 72 months in the OLE. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk. The decision to extend and informed consent should be completed before the start of the first visit of each annual extension (i.e. Month 12, 24, 36, 48 and 60). After approval from Investigator and Sponsor for extension and starting after Visit26/Month24 (or a later visit if Visit26/Month24 visit has already occurred at the time of Protocol Amendment 4.0 approval), subject will return to the clinic every 6 months and have a phone visit 3 months after the in clinic visit for each 1-year extension, until up to Month 72. The End of Study will be Visit 42. Further extensions can then be applied as required if marketing approval is not yet received

### 1. INTRODUCTION

#### 1.1 BACKGROUND INFORMATION ON INDICATION STUDIED

ZX008 (fenfluramine hydrochloride) is under clinical development for the adjunctive treatment of patients with Dravet syndrome and Lennox-Gastaut syndrome (LGS). Fenfluramine (Fintepla®) is authorized for sale in the United States for the treatment of seizures associated with Dravet syndrome in patients 2 years of age and older.

LGS is a rare epileptic encephalopathy. Onset of LGS usually occurs most commonly before age 11, with a peak between 3 and 5 years of age (Arzimanoglou 2009; Hancock and Cross, 2013). Patients with LGS account for 5–10% of children with seizures (Panayiotopoulos 2005). The diagnosis of LGS includes clinical signs combined with typical EEG features. The clinical presentation of LGS is heterogeneous, however LGS is always characterized by a triad of symptoms: multiple seizure types, slow spike-and-wave EEG, and abnormal cognitive development. The most common seizure types are generalized tonic-clonic seizures, tonic seizures, atonic seizures, and tonic/atonic seizures, all of which most often can result in "drop attacks." Other seizure types that occur in some LGS patients include atypical absences, non-convulsive seizures, focal seizures, and myoclonic seizures. Nearly all LGS patients have treatment-resistant, lifelong epilepsy. Prognosis for LGS is very poor: 5% of children die, 80–90% continue having seizures into adulthood, and nearly all have cognitive and behavioral problems (Panayiotopoulos 2005). Children and adults with LGS have an enormous impact on their families, and efforts to improve the quality of life for these patients are complex.

# 1.1.1 Existing Treatment for LGS.

Currently, two drugs are approved in Japan for the treatment of Lennox-Gastaut syndrome: lamotrigine (2008) and rufinamide (2013). Nine AEDs are approved for treating Lennox-Gastaut syndrome EU-wide and in selected EU Member States: felbamate, topiramate, lamotrigine, rufinamide, clonazepam, clobazam, valproate, nitrazepam, and cannabidiol (Epidyolex®). The same AEDs are approved in the US except valproate and nitrazepam. Other pharmacologic (valproate, benzodiazepines, zonisamide) and non-pharmacologic (KD, VNS, surgery) treatments also are prescribed based on clinical experience.

Because patients with LGS experience a range of different seizure types, the condition is notoriously difficult to treat (Arzimanoglou 2009, Cross 2017) and seizures in LGS are usually not fully controlled (Hancock, 2013). Initial treatment for LGS is usually monotherapy with one of the currently approved AEDs. If this is not successful, which is the most common case, a second agent is usually added; although some physicians move on to the second drug as monotherapy (Wheless 2007; Arzimanoglou 2009). The treatment of LGS frequently requires a combination of 2 or more of these compounds, but with continued suboptimal seizure control. The recommendation is to attempt to use drugs that have different mechanisms of action and the least amount of interaction with one other. After lack of response to 2 or more AEDs, non-pharmacological treatments such as KD, VNS, or surgery may be considered. A treatment that has been shown to be effective in common certain seizure types cannot be assumed to be effective in patients with LGS to treat that seizure type.

Given the suboptimal treatment of seizures in the majority of LGS patients, even with


polytherapy, and the developmental and cognitive consequences believed to be caused, at least in part, by frequent childhood seizure activity, there is a medical need for a new anticonvulsant treatment with a novel mechanism of action that can significantly reduce seizure activity in LGS.

### 1.2 BACKGROUND INFORMATION ON STUDY PRODUCT

Zogenix is developing a new formulation of fenfluramine hydrochloride, ZX008, for the adjunctive treatment of seizures associated with LGS. Fenfluramine is an amphetamine analogue that was first synthesized many years ago. It was approved in a large number of countries and widely prescribed as an appetite suppressant for the treatment of adult obesity. Brand names for fenfluramine formulations included Ponderax and Pondimin. Fenfluramine was also used extensively in an off-label combination with phentermine ("Fen-Phen"). Fenfluramine is a racemic compound and the single enantiomer D-fenfluramine (dexfenfluramine) was also approved and marketed for the treatment of obesity as Adifax, Redux, and others.

Fenfluramine was introduced in the USA in 1973. Products containing fenfluramine and D-fenfluramine were withdrawn from all markets between 1997 and 2000 after reports of heart valve disease and pulmonary hypertension (Connolly 1997; CDC 1997; Wong 1998). While the risk/benefit relationship for fenfluramine is thus considered unfavorable for the treatment of obesity in adults, establishing seizure control in LGS or any of the refractory catastrophic childhood epilepsies might lead to a more acceptable risk/benefit profile for fenfluramine.

As a result of this previous extensive use of fenfluramine, there is a large body of information in the public domain concerning its pharmacology, toxicology and use in the treatment of obesity. These data are summarized in the ZX008 Investigator Brochure (ZX008 IB). There is also a large body of information concerning its clinical safety profile.

# 1.3 CLINICAL DATA

Two double-blind, placebo-controlled, randomized Phase 3 studies (Study 1 and Study 1504 Cohort 2) of ZX008 in children and young adults with Dravet syndrome have been completed. Study 1 investigated two doses of ZX008 (0.2 and 0.8 mg/kg/day) or placebo and included 119 subjects with Dravet syndrome from North America, Europe and Australia. Study 1504 Cohort 2 included 87 subjects from North America and Europe, and compared addition of ZX008 (0.5 mg/kg/day) or placebo in subjects who were receiving standard of care anti-epileptic treatments where administration of STP was mandatory.

The primary efficacy measure in both studies was the change from baseline in the frequency of convulsive seizures (per 28 days) during the combined 14-week (Study 1) or 15-week (Study 1504 Cohort 2) Titration and Maintenance periods (T+M). The primary analysis in Study 1 compared ZX008 0.8 mg/kg/day to placebo and in Study 1504 Cohort 2 compared ZX008 0.5 mg/kg/day to placebo. A key secondary measure in Study 1 compared the 0.2 mg/kg/day group to the placebo group on the same measure. Other key secondary measures in both studies included a comparison of the  $\geq$  50% Responder Rate (ie, the number of subjects with a  $\geq$  50% reduction in the frequency of convulsive seizures), and the longest seizure free interval.


Both Study 1 and Study 1504 Cohort 2 met the primary endpoint with a highly statistically significant reduction in convulsive seizures in all active treatment groups.

In Study 1, subjects randomized to ZX008 0.8 mg/kg/day and 0.2 mg/kg/day had a median baseline convulsive seizure frequency of 20.7 and 17.5, respectively, compared to 27.3 for subjects randomized to placebo. Subjects randomized to ZX008 0.8 mg/kg/day (n= 40) achieved a 62.3% greater reduction in mean monthly convulsive seizure frequency (P<0.001) compared to those in the placebo group (n=40). In addition, subjects randomized to ZX008 0.2 mg/kg/day (n=39) had a 32.4% reduction compared to placebo (P = 0.021). Comparing the seizure reduction results for the 2 doses of ZX008 in Study 1 suggests a dose-response effect on seizures. The pattern of individual responses in the ZX008 0.2 mg/kg/day group supports the selection of 0.2 mg/kg/day as the minimally effective dose.

In Study 1504 Cohort 2, subjects randomized to ZX008 0.5 mg/kg/day had a median baseline convulsive seizure frequency 14.0 compared to 10.7 for subjects randomized to placebo. Subjects randomized to ZX008 0.5 mg/kg/day achieved a 54.0% reduction compared to placebo (P < 0.001).

Controlling for multiplicity with a hierarchical testing procedure, all key secondary endpoints were met in both studies, for ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups (Study 1) and ZX008 0.5 mg/kg/day (Study 1504 Cohort 2). In Study 1, the proportion of subjects achieving a  $\geq$  50% reduction from Baseline in CSF was 67.5% for the ZX008 0.8 mg/kg/day group, and 38.5% for the 0.2 mg/kg/day group, with both groups being statistically significantly different from placebo (12.5%; P < 0.001 and P = 0.009, respectively). In Study 1504 Cohort 2, 53.5% of subjects randomized to ZX008 0.5 mg/kg/day compared to 4.5% of subjects randomized to placebo achieved a  $\geq$  50% reduction from Baseline in CSF (P <0.001).

The proportion of subjects with a  $\geq$  50% reduction in monthly convulsive seizure frequency was also highly statistically significant for all ZX008 dose groups compared to placebo, with 38.5%, 53.5%, and 67.5% of subjects in the 0.2 mg/kg/day, 0.5 mg/kg/day, and 0.8 mg/kg/day cohorts achieving  $\geq$  50% reduction as compared to 8.3% in placebo. Additionally, in Study 1, subjects randomized to ZX008 0.2 and 0.8 mg/kg/day had a median 15- and 25-day convulsive seizure-free interval, respectively, compared to 9.5 days for placebo (P = 0.035 and P < 0.001). In Study 1504 Cohort 2, subjects randomized to ZX008 0.5 mg/kg/day had a median 22-day convulsive seizure-free interval compared to 13 days for placebo (P < 0.004).

ZX008 was generally well tolerated in both Study 1 and Study 1504 Cohort 2. Though more subjects randomized to ZX008 than to placebo reported TEAEs during the double-blind studies, the percent of subjects with serious TEAEs was similar. Additionally, the adverse events observed in the program were either already known to be associated with fenfluramine, are common to many other antiepileptic drugs being prescribed to these patients, and/or are common to the age group and population studied. Specifically, the most common adverse events seen were diarrhea, fatigue, pyrexia, upper respiratory tract infection, blood glucose decreased, weight decreased, decreased appetite, lethargy and tremor. No valvular heart disease, pulmonary arterial hypertension or abnormal valve structure was observed in any subject at any time during the entire program.


In an integrated analysis of safety of the double-blind studies, 117 (95.9%) subjects in any ZX008 treatment group and 68 (81.0%) subjects in the combined placebo group reported at least 1 TEAE. The most common (≥ 10%) TEAEs reported in subjects receiving any dose of ZX008 were: blood glucose decreased, constipation, decreased appetite, diarrhea, echocardiogram abnormal, fall, fatigue, lethargy, nasopharyngitis, pyrexia, seizure, somnolence, status epilepticus, tremor, upper respiratory tract infection, vomiting, and weight decreased. All of the echocardiogram abnormal TEAEs were trace mitral or trace aortic valve regurgitation, which are normal physiological findings seen in healthy children (Webb 2015). A total of 15 (12.3%) subjects in any ZX008 treatment group and 11 (13.1%) subjects in the combined placebo group reported at least 1 serious TEAE. The most frequently reported (≥ 5%) serious AEs (SAEs) were status epilepticus and seizure. A total of 76 (62.3%) subjects in any ZX008 treatment group and 22 (26.2%) subjects in the combined placebo group reported a TEAE determined by the Investigators to be related to the study drug, and 3 (2.5%) subjects in any ZX008 treatment group and 1 (1.2%) subject in the combined placebo group reported a serious TEAE determined to be related to the study drug. During the double-blind treatment periods, 7 (5.7%) subjects in any ZX008 treatment group and 1 (1.2%) subject in the combined placebo group reported a TEAE that lead to discontinuation from study participation. There were no deaths during the doubleblind treatment periods.

Subjects in Study 1 and Study 1504 if eligible could participate in Study 1503, an open-label long-term, safety extension study that is currently ongoing. All subjects in Study 1503 started ZX008 at 0.2 mg/kg/day and could flexibly titrate to a maximum dose of 0.8 mg/kg/day, maximum 30 mg/day (if not receiving a concomitant STP regimen) or 0.5 mg/kg/day, maximum 20 mg/day (if receiving concomitant STP regimen), based on effectiveness, safety and tolerability. Though primarily a safety study, subjects in Study 1503 maintained a daily seizure diary and continued to complete rating scales on overall effectiveness and quality of life measures.

In a safety update of Study 1503 (cut-off date 14-Oct-2019, n=330 enrolled), the median percent change in CSF compared to baseline (core study) for the overall open-label Treatment period (Day 1 to End of Study [EOS]) was -66.8% (P < 0.001). The reduction from baseline in monthly CSF observed at Month 1 of the open-label Treatment period was maintained through Month 24, the longest treatment duration included in the analysis. A total of 317/330 subjects reported at least 1 TEAE during the open-label Treatment period. The most common (≥ 10%) TEAEs reported during the open-label Study 1503 at the time of the cut-off date were blood glucose decreased, decreased appetite, diarrhea, ear infection, echocardiogram abnormal, influenza, nasopharyngitis, pyrexia, seizure, and upper respiratory tract infection. As in the double-blind studies, all of the echocardiogram abnormal TEAEs in Study 1503 were trace mitral or trace aortic valve regurgitation, which are not considered pathologic as stated in current guidelines on the use of ECHO for the assessment of valve function (Zoghbi 2017, Lancellotti 2010a, Lancellotti 2010b). At least 1 treatment-emergent SAE was reported by 80/330 (24.2%) subjects. The most frequently reported ( $\geq 5\%$ ) SAE was seizure, occurring in 24/330 (7.3%) of subjects. A total of 176/330 subjects (53.3%) experienced at least 1 TEAE that was considered to be related to study treatment and 8/330 subjects (2.4%) reported at least 1 SAE that was considered to be related to study treatment. A total of 11/330 (3.3%) subjects discontinued due to a TEAE.


Please reference the ZX008 IB for more detailed information on the safety and efficacy of ZX008.

# 1.4 PHARMACOKINETICS, PRECLINICAL DATA, AND CLINICAL PHARMACOLOGY

#### 1.4.1 Pharmacokinetics

The pharmacokinetics of fenfluramine, norfenfluramine and their respective isomers have been studied in mice, rats, dogs and humans. Fenfluramine and norfenfluramine were more slowly eliminated in humans than in other species. In vitro metabolism studies have shown considerable species differences in the metabolism of fenfluramine, with no single species having a profile similar to humans. No human-specific metabolites were detected and both rat and dog showed good coverage of the human fenfluramine metabolites. In humans, fenfluramine is metabolized primarily to norfenfluramine. Fenfluramine is partially metabolized by CYP1A2, CYP2B6, and CYP2D6, with additional metabolism by CYP2C9, CYP2C19, and CYP3A4. Norfenfluramine does not appear to be strong substrate of any CYP450 enzyme, but is metabolized by CYP1A2, CYP2B6, CYP2C19, and CYP2D6 in vitro. There is also some contribution of renal clearance to the elimination of dexfenfluramine (8%-16%) and nordexfenflurmaine (7%-8%) from the body. Because fenfluramine and its active metabolite norfenfluramine have multiple pathways of elimination, interference with a single pathway is unlikely to cause a significant change in fenfluramine's clearance though the probability of an interaction increases if multiple elimination mechanisms are affected simultaneously.

While in vitro studies showed that both fenfluramine and norfenfluramine cause weak inhibition of CYP2D6 and fenfluramine causes weak induction of CYP3A4 and CYP2B6, further analysis based on the FDA's mechanistic static model shows that fenfluramine and its major metabolite norfenfluramine are unlikely to alter the pharmacokinetics of substrates of CYP450 enzymes in the range of ZX008 doses that will be administered in this study.

In Study 1 and Study 1504 Cohort 2, pharmacokinetic parameters of fenfluramine and norfenfluramine for patients with Dravet syndrome were determined using a population pharmacokinetic (PopPK) model developed using PK data from both healthy volunteers and patients with Dravet syndrome. The Study 1 data are provided in Table 3.

Table 3 Post Hoc Estimates of Fenfluramine and Norfenfluramine Steady-State Pharmacokinetic Parameters in Subjects with Dravet Syndrome in Study 1 (Geometric Mean [CV%])

| Analyte: | Fenfluramine | | Norfenfluramine | |
|---|---|---|---|---|
| ZX008 Dose | 0.2 mg/kg/day | 0.8 mg/kg/day | 0.2 mg/kg/day | 0.8 mg/kg/day |
| C <sub>max</sub> (ng/mL) | 18.5 (29.1) | 68.0 (40.7) | 9.60 (52.8) | 37.8 (49.9) |
| $AUC_{0\text{-}24}(ng.hr/mL)$ | 375 (32.9) | 1390 (43.5) | 220 (55.5) | 872 (52.1) |
| T <sub>max</sub> (hr) Median (Min, Max) | 3.00 (3.00 to 3.50) | 3.00 (3.00 to 3.50) | 4.00 (3.50 to 5.00) | 4.50 (3.50 to 5.00) |

Source: ICPD Report 00445-3, Table 5.

Abbreviations: AUC<sub>0.24</sub> = area under the plasma concentration-time curve from time 0 to 24 hours; BID = twice daily;


 $C_{max}$  = peak plasma drug concentration; CV= coefficient of variation; Max = maximum; Min = minimum;  $T_{max}$  = time of peak plasma drug concentration.

Study 1504 Cohort 2 required STP as a concomitant medication. Although the dose of ZX008 in Study 1504 Cohort 2 was lower than the high dose in Study 1, fenfluramine AUC0-24 values were approximately 130% higher in Study 1504 Cohort 2, than the high dose in Study 1, and norfenfluramine AUC0-24 values were approximately 60% lower than in Study 1. However, the clinical results indicated that the efficacy and AE profile were similar between Study 1 and Study 1504, indicating that the dose adjustment studied for the concomitant use of the STP regimen met the intended clinical outcome.

#### 1.4.2 Preclinical Data

A 10-week GLP juvenile toxicology and toxicokinetic study in rats, which included fenfluramine doses of 3.5, 9 and 20 mg/kg/day by oral gavage for 10 weeks (post natal day (PND) 7 to 76). The data from the juvenile toxicology studies suggest that the effects of fenfluramine in juvenile animals (CNS-related clinical signs, effects on body weight and food consumption, and neurobehavioral deficits) are similar to effects previously reported in neonatal and adult rats (Morford, 2002; Williams, 2002). There was no evidence of CNS histopathology; importantly, there were also no histopathologic findings in aortic or mitral cardiac valves, and no adverse effects on any other tissues at necropsy.

The NOAEL for the juvenile rats was determined to be 9 mg/kg/day. A NOAEL of 9 mg/kg/day corresponds to PND 76 AUC0-t of 3480 hr\*ng/mL for males and 4680 hr\*ng/mL for females for fenfluramine, and 4470 hr\*ng/mL for males and 6210 hr\*ng/mL for females for norfenfluramine. The AUC(0-t) at the NOAEL provided a safety factor (both sexes combined) of approximately 3-fold or higher for fenfluramine and approximately 6-fold or higher for norfenfluramine.

# 1.4.3 Clinical Pharmacology

Please see the ZX008 IB for details on clinical pharmacology. Below are the clinical pharmacology conclusions.

- Coadministration of ZX008 with the STP regimen (STP with CLB and/or VPA) resulted in an increased fenfluramine and decreased norfenfluramine concentrations, and therefore a dose adjustment is used in the clinical trials.
- STP is the predominant perpetrator of the interaction; while VPA and CLB do not have a significant independent impact on the PK of fenfluramine or norfenfluramine, whether administered with or without STP.
- Coadministration of ZX008 with CBD at steady state resulted in increased fenfluramine concentrations but this increase was within the range of safe dosing used in Study 1504 Cohort 2; thus, no dose adjustment is recommended when fenfluramine is coadministered with CBD.
- In the population PK analysis, intrinsic patient factors (age, gender, race/ethnicity, and BMI) demonstrated no substantial impact on the clearance or exposure to fenfluramine or norfenfluramine when dosed on a mg/kg basis to a maximum of 30 mg/day.


- ZX008 had no effect on QTc intervals at either the therapeutic or supratherapeutic dose, and no relationship was observed between fenfluramine or norfenfluramine exposure and QTcF.

Surveype for CYP1A2, CYP2B6, CYP2C19, CYP2D6, or Surveype for CYP1A2, CYP2B6, CYP2C19, CYP2B6, or Surveype for CYP1A2, CYP2B6, CYP2B6, CYP2B6, or Surveype for CYP2B6, CYP2B6, CYP2B6, CYP2B6, or Surveype for CYP2B6, CYP2B6, CYP2B6, CYP2B6, or Surveype for CYP2B6, CYP2B6, CYP2B6, CYP2B6, CYP2B6, or Surveype for CYP2B6, CYP2B6, CYP2B6, or Surveype for CYP2B6, CYP2B6, CYP2B6, or Surveype for CYP2B6, CYP2B6, or Surveype for CYP2B6, or Surveype for CYP2B6, CYP2B6, or Surveype for

# BACKGROUND INFORMATION ON REFERENCE PRODUCT le. RATIONALE FOR CUIDDENT STATES.

Not applicable.

#### 1.6 RATIONALE FOR CURRENT STUDY

There have been several published reports of fenfluramine's successful treatment of refractory childhood epilepsy in the 1980s (Aicardi 1985; Aicardi 1988) and its successful treatment of 11 refractory pediatric epilepsy patients in Belgium (Boel 1996).

A number of small studies and case series have been published describing the use of fenfluramine in epilepsy. In 1996, a Belgian group reported on the use of fenfluramine in 11 children (ages 18 months to 15.5 years old) with refractory or self-induced epilepsy (Boel 1996). Patients were treated with fenfluramine at 0.5 - 1 mg/kg/day for 3 to 8.5 years (average duration 5 years 7 months). Seven children (64%) became seizure-free and the remaining 4 patients experienced ≥75% reduction in seizure frequency.

In 2002, Casaer and Boel published a brief update of their study with fenfluramine. The study population was expanded to 22 patients with intractable or self-induced seizures, including the previously reported 11 patients (Casaer 2002). The duration of treatment was between 1 and 12 years. In this study, of the 22 patients treated, 6 (27%) became seizure-free, 10 (45%) patients had a 90% reduction in seizure frequency and 6 (27%) patients were non-responders.

Fenfluramine was also shown to be effective in multiple seizures types in Dravet syndrome (DS), another very drug resistant pediatric epileptic encephalopathy syndrome (Ceulemans 2012; Schoonjans 2015; Ceulemans 2016; Schoonjans 2017). Zogenix is currently evaluating ZX008 in Dravet Syndrome in two Phase 3 double-blind, randomized, placebo-controlled studies and one open-label extension (clinicaltrials.gov identifiers: NCT02826863, NCT02682927, and NCT02823145).

Currently, a small cohort of refractory patients with Lennox-Gastaut syndrome in Belgium are being treated in an ongoing Phase 2 open-label, pilot, dose-finding trial of fenfluramine as an add-on therapy to conventional therapy (Lagae, 2017; Study S58545; clinicaltrials.gov identifier: NCT02655198).

The study includes a 20-week Core period, in which subjects are titrated to ≥50% response and then held at that dose until the end of the 20-week period, and an Extension period, in which subjects are titrated to maximum efficacy and tolerability. Subjects aged 3 to 18 years, fulfilling the diagnostic criteria for LGS as described by the ILAE in 1989, who have failed at least two


AEDs (including VNS), and have had at least 4 documented convulsive seizures (General Tonic Clonic, Tonic Seizures, Atonic Seizure, and Focal Seizure with a motor component) and on at least two AEDs at stable doses in the prior 4 weeks are eligible for this study. After the initial 4-week baseline period to record seizure type and frequency, treatment with fenfluramine, 0.2 mg/kg/day, is initiated. An efficacy response ("responder") is defined as a  $\geq$ 50% reduction in major motor seizure frequency (GTC+TS+AS+FS). At the 8-week visit (following 4 weeks of ZX008 treatment), subjects who were non-responders and have no intolerable side effects receive an increased dose of 0.4 mg/kg/day. At the 12-week visit, subjects who were non-responders and have no intolerable side effects receive an increased dose of 0.8 mg/kg/day. At any visit, subjects who achieve a  $\geq$ 50% reduction in major motor seizure frequency remain at their currently administered dose. As this is a pilot dose-finding study, it is important to note that per protocol, dose escalation stops when a subject's convulsive seizure frequency is reduced by  $\geq$ 50% of baseline. It is possible that a higher dose could result in even greater seizure reduction. The maximum allowed dose is 30 mg/day.

Results have been presented for the 13 LGS subjects who completed the Core study: (Lagae, 2017). Overall, subjects had received a median of 8 years of antiepileptic treatment and were failing a median of 5 AEDs prior to entry. Upon study entry, patients were taking a median of 4 concurrent anti-epileptic therapies. All subjects received ZX008 treatment for at least 20 weeks with the exception of 3 subjects who discontinued due to lack of efficacy; of which 2 also discontinued due to side effects. For subjects who completed the 20-week Core period, the median seizure frequency was reduced from a mean of 60 major motor seizures per month in the pre-ZX008 baseline period to a mean of 22 major motor seizures per month at the end of the Core ZX008 treatment period. At week 20, 8 of the 13 enrolled patients (62%) had at least a 50% reduction in major motor seizures with ZX008 treatment. Nine of the 13 patients completed the Core period and entered the Extension period. At the time of each of subjects' most recent visit, 6 of 9 patients (67%) had at least a 50% reduction in major motor seizures and 2 of 9 (22%) had a 75% or greater seizure reduction. In the Extension period, there was a 58% median reduction in seizure frequency as compared to baseline. The most common treatment emergent adverse events to date include decreased appetite (n=4) and decreased alertness/fatigue (n=3). Sleep problems, tiredness, and sleepiness were each reported in one subject.

No clinical signs of valvulopathy or pulmonary hypertension have been observed in any patients in the Belgian cohort (ZX008 IB).

In addition, numerous publications discuss the use of fenfluramine in over 500 children with neurobehavioral conditions for the treatment of mostly autism and ADHD, without any reports of any cardiovascular adverse events (summarized in ZX008 IB).

Prior to being withdrawn from the market, fenfluramine was marketed at doses of 20 mg and 40 mg three times daily for the management of obesity in adults. The doses tested thus far in DS range from 0.12 to 0.9 mg/kg/day in subjects over 1 year of age to adults in the Belgian cohort, and 0.2 and 0.8 mg/kg/day in the Zogenix Phase 3 trials. Doses tested in pediatric studies evaluating autism and ADHD ranged from 0.65 mg/kg/day to 3.6 mg/kg/day, but a commonly used dose was 1.5 mg/kg/day. Occasionally, fixed doses of 30 to 80 mg were used. The PK exposure associated with the doses in the LGS study of 0.2 mg/kg/day and 0.8 mg/kg/day, administered orally (in equally divided doses BID) is expected to be lower than that obtained at the doses used in the past for the treatment of obesity in adults and of neurobehavioral conditions


in children and adolescents (ZX008 IB). The doses used in this study are based on the data from the DS and LGS patients being successfully treated in Belgium discussed above.

In summary, fenfluramine has been shown to be effective in reducing the frequency of seizures in patients with Dravet syndrome and LGS, and its activity persists over a long duration of time (Ceulemans 2012, Ceulemans 2016, Schoonjans 2017, Lagae 2018). Though the mechanism remains to be fully elucidated, data from in vitro receptor binding, functional assays, and zebrafish models suggest that fenfluramine reduces seizures by acting as an agonist at the 5-HT1D and the 5-HT2C receptors and by acting on the sigma-1 receptor. Fenfluramine may also exert anti-seizure activity through the 5-HT1A and the 5-HT2A receptors (ZX008 IB 2018).

The lack of consistent efficacy and individual tolerability and safety concerns with current treatments available for LGS have resulted in the continued significant unmet need for a new treatment with a novel mechanism of action for children and adults with LGS.

The rationale for conducting the Part 2 open-label extension period is primarily to evaluate the long-term safety of ZX008 in subjects with LGS. This protocol also provides the opportunity for continued treatment for subjects responding to treatment from Part 1 and an opportunity for initial treatment with ZX008 for subjects randomized to placebo in Part 1. The study will also allow access to ZX008 for the treatment of LGS for eligible Japanese subjects until commercial product is available, as it is not approved in Japan. The period from the approval of this drug to its launch is positioned as a post-marketing study.

# 1.7 RISK-BENEFIT ASSESSMENT

As described above, fenfluramine has been used successfully for up to 30 years in Belgium in refractory pediatric epilepsy patients, including those with LGS and DS (<u>Boel 1996</u>, <u>Ceulemans 2012</u>, <u>Schoonjans 2015</u>, <u>Schoonjans 2017</u>). The doses tested thus far in DS range from 0.12 to 0.9 mg/kg/day in subjects over 1 year of age to adults. No patients have developed valvulopathy or pulmonary hypertension.

The clinical benefit of ZX008 in the Lennox-Gastaut syndrome has been evaluated in an open label study (Lagae 2017, 2018) as mentioned in Section 1.6. In addition, 2 positive, adequate and well-controlled, multi-national, randomized, double-blind, placebo-controlled trials of ZX008 in subjects with Dravet syndrome, Study 1 and Study 1504 Cohort 2, demonstrated a statistically significant and clinically meaningful reduction in monthly convulsive seizure frequency and was generally well tolerated. There was no clinical or echocardiographic evidence of cardiac valvulopathy or pulmonary hypertension in any study and no patient discontinued participation or required a change in monitoring in the study due to cardiac factors. The PK exposure associated with the doses of ZX008 in the Dravet syndrome studies of 0.2 mg/kg/day to 0.8 mg/kg/day administered orally [in equally divided doses twice per day (BID)] is lower than that obtained at the doses used in the past for the treatment of obesity in adults and of neurobehavioral conditions in children and adolescents (ZX008 IB). The doses used in this study are based on the data from the patients being successfully treated in Belgium discussed above, Study 1, and Study 1504 Cohort 2 data.

The pharmacologic and toxicological profile for the active pharmaceutical ingredient,


fenfluramine, following oral administration is well established (see ZX008 IB).

The safety monitoring practices employed by this protocol are adequate to protect the subjects' safety and should detect expected and unexpected treatment-emergent adverse events, and are the same as those currently being utilized for the global Phase 3 DS program.

The approximate volume of blood (194.0 mL) planned for collection from each subject over the course of the entire study (Screening to End of Study Part 2, but not including repeat or additional tests ordered by the investigator) presents no undue risk to the subjects.

The ZX008 0.2 mg/kg/day and 0.8 mg/kg/day doses are believed to be likely therapeutic doses, which could provide sufficient anti-epileptic effect for a sustained period of time during the study.

The available information suggests that the present clinical study has an acceptable risk-benefit ratio.

# 2. STUDY OBJECTIVES AND ENDPOINTS

#### 2.1 PART 1

#### 2.1.1 PRIMARY OBJECTIVE

The primary objective of Part 1 is the primary objective of the entire study.

The primary objective of Part 1 is:

• To evaluate the effect of ZX008 0.8 mg/kg/day versus placebo as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with Lennox-Gastaut syndrome (LGS) based on the change in frequency of seizures that result in drops between baseline and the combined Titration and Maintenance Periods (T+M).

# 2.1.2 KEY SECONDARY OBJECTIVES

The key secondary objectives of Part 1 are:

- To evaluate the effect of ZX008 0.2 mg/kg/day versus placebo as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with LGS based on the change in frequency of seizures that result in drops between baseline and T+M.
  - To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the proportion of subjects who achieve a ≥50% reduction from baseline in the frequency of seizures that result in drops.
  - To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the Clinical Global Impression Improvement rating, as assessed by the principal investigator.

See Statistical Methods (Section 10.1.5.1) for hierarchical testing procedure.

#### 2.1.3 ADDITIONAL SECONDARY OBJECTIVES

Additional secondary objectives of the study are:


- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
  - Change in the frequency of all countable motor seizures between baseline and T+M (countable seizures include: generalized tonic-clonic seizures [GTC], tonic seizures [TS], clonic seizures [CS], atonic seizures [AS], tonic/atonic seizures [TA], clearly recognizable focal seizures [FS], and myoclonic seizures [MS] that result in a drop).
  - Change in the frequency of all countable seizures (ie, motor and non-motor) between baseline and T+M
  - Change in frequency of seizures that result in drops between baseline and the Maintenance Period (M)
  - Change in the frequency of countable motor seizures that do not result in drops between baseline and M
  - The proportion of subjects who have a worsening or no change (i.e. ≤0% reduction), >0%, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizures freedom" (ie 0 or 1 seizures) between baseline and T+M, and baseline and M, in all countable motor seizures (GTC, TS, AS, TA, FS, MS with a drop); in countable motor seizures that do not result in drops; in all countable seizures; in all countable seizures that do not result in drops, and in all seizures that result in drops

\_

- Longest interval between seizures that result in drops
- Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the Clinical Global Impression Improvement rating, as assessed by the parent/caregiver.

## 2.1.4 SAFETY OBJECTIVE

The safety objectives of Part 1 are:

- To evaluate the safety and tolerability of ZX008 0.2 and 0.8 mg/kg/day versus placebo with regard to adverse events (AEs), laboratory parameters, physical examination, neurological examination, vital signs (blood pressure, heart rate, temperature, and respiratory rate), electrocardiograms (ECG), echocardiograms (ECHO), body weight, and BMI
- To evaluate the change from baseline in cognition using age-appropriate versions of the BRIEF

#### 2.1.5 PHARMACOKINETIC OBJECTIVE

The pharmacokinetic (PK) objective of the study is:

• To evaluate the PK of ZX008 0.2 and 0.8 mg/kg/day at steady state in subjects < 18 years and ≥18 years with LGS using a non-compartmental analysis; and obtain exposure data that will be used in population pharmacokinetic (PopPK) analysis, the results of which will be reported separately.


#### 2.1.6 EXPLORATORY OBJECTIVES

The exploratory objectives of the study are:

- To compare the ZX008 0.2 and 0.8 mg/kg/day doses on primary, secondary, and safety endpoints.
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
  - The frequency of rescue medication usage
  - The incidence of medical services to treat seizures
  - The incidence of status epilepticus
  - The change from baseline in behavior using the Vineland Adaptive Behavior Scale (VABS)(Cohort A)
  - The change from baseline in QoL using the QOLCE
  - The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory
  - The change from baseline in affective symptoms of the parent/caregiver using the Hospital Anxiety and Depression Scale (HADS)

#### 2.2 PART 2

#### 2.2.1 PRIMARY OBJECTIVE

The primary objective of Part 2 is to assess the long-term safety and tolerability of ZX008 in children and adults with LGS with regard to adverse events (AEs), laboratory parameters, physical examination, neurological examination, cognition (BRIEF), vital signs (blood pressure, heart rate, temperature, and respiratory rate), ECG, ECHO, body weight, and BMI.

# 2.2.2 SECONDARY OBJECTIVES

The secondary objectives of Part 2 are:

- To assess the effect of ZX008 relative to the baseline on the following effectiveness measures:
  - The change in the frequency of seizures that result in drops
  - The change in the frequency of all countable motor seizures (GTC, TS, CS, AS, TA, FS, MS with a drop)
  - The change in the frequency of all countable seizures
  - The proportion of subjects who have a worsening or no change (i.e. ≤ 0% reduction), >0 %, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizure freedom (ie, 0 or 1 seizures) in frequency of all countable seizures that result in drops, countable motor seizures that do not result in drops, all countable motor seizures, all countable seizures, and all countable seizures that do not result in drops
  - Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
  - Longest interval between seizures that result in drops


- To evaluate the effect of ZX008 on the following endpoints:
  - Clinical Global Impression Improvement rating, as assessed by the principal investigator
  - Clinical Global Impression Improvement rating, as assessed by the parent/caregiver

#### 2.2.3 EXPLORATORY OBJECTIVES

The exploratory objectives of Part 2 are:

- To estimate the incidence of the following on subjects receiving ZX008:
  - The incidence medical services use to treat seizures
  - The incidence of status epilepticus
  - The use of rescue medication
- To assess the effect of ZX008 on the following measures:
- Tusing to - The change from baseline in affective symptoms of the parent/caregiver using the HADS
  - The change from baseline in QoL using the QOLCE
  - The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory

#### 2.3 STUDY ENDPOINTS

#### 2.3.1 **Efficacy Endpoints**

The efficacy endpoints for Part 1 of the study are:

Primary Endpoint:

• Percent change from baseline in the frequency of seizures that result in drops in the combined Titration and Maintenance Periods (T+M) in the ZX008 0.8 mg/kg/day group compared to the placebo group.

Key Secondary Endpoints:

- Change from baseline in the frequency of seizures that result in drops in T+M in the ZX008 0.2 mg/kg/day group compared to the placebo group
- Proportion of subjects who achieve a  $\geq$ 50% reduction from baseline in the frequency of seizures that result in drops comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo
- Proportion of subjects who achieve improvement (minimally, much, or very much improved) in the Clinical Global Impression – Improvement as assessed by Principal Investigator comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo.
- Number, frequency, and duration of countable seizures that result in drops
- Number, frequency, and duration of countable seizures that do not result in drops
- Number, frequency, and duration of all countable seizures by type
- Proportion of subjects who achieve a  $\geq 25\%$ ,  $\geq 50\%$ ,  $\geq 75\%$ , or 100% reduction from baseline in seizure frequency
- Number of seizure-free days
- Clinical Global Impression Improvement as assessed by parent/caregiver


The efficacy endpoints for Part 2 of the study are:

- The change from baseline in the frequency of seizures that result in drops.
- The change from baseline in the frequency of all countable motor seizures (GTC, TS, CS, AS, TA, FS, MS with a drop)
- The change from baseline in the frequency of all countable seizures
- The proportion of subjects who achieve a worsening from baseline (i.e. <= 0% reduction), or >0%, ≥ 25%, ≥ 50%, ≥ 75%, and 100% reduction from baseline in frequency of all countable seizures that result in drops, countable motor seizures that do not result in drops, all countable motor seizures, all countable seizures that do not result in drops
- Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops
- Number of instances of rescue medication use and number of doses of rescue medication
- Longest interval between seizures that result in drops
- Clinical Global Impression Improvement rating, as assessed by the Principal Investigator.
- Clinical Global Impression Improvement rating, as assessed by the parent/caregiver.

## 2.3.2 Safety Endpoints

The safety endpoints for Part1 and Part 2 of the study are

- AEs
- Laboratory safety (hematology, chemistry, urinalysis)
- Vital signs (blood pressure, heart rate, temperature, and respiratory rate)
- Body weight and BMI
- Physical examination
- Neurological examination
- BRIEF to measure changes in cognition of the subject
- Columbia Suicidality Severity Rating Scale (C-SSRS)
- 12-lead ECGs
- Doppler ECHOs

#### 2.3.3 Exploratory Endpoints

The exploratory endpoints for Part 1 and Part 2 of the study are:

- The incidence of medical services used to treat seizures
- The incidence of status epilepticus
- Incidence of rescue medication usage
- Number of days rescue medication used
- The change from baseline in behavior using the Vineland Adaptive Behavior Scale (VABS) (Part 1 Cohort A only)
- The change from baseline in quality of life using the QOLCE
- The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory


The change from baseline in affective symptoms of parent/caregiver using the HADS scale

#### 3. INVESTIGATIONAL PLAN

This is an international multicenter study being conducted in two parts. Up to approximately 80 study sites in North America, Europe, Japan, and Australia are initially planned to participate. Part 1 is a double-blind, parallel-group placeholicated and safety of two 3. children and adult subjects with LGS. Part 1 will include 2 cohorts: Cohort A will include randomized subjects from North America, Europe, and Australia; Cohort B will include randomized subjects from Japan only. The primary study endpoint is assessed from Part 1 Cohort A data. The primary analysis will be conducted when the last subject in Cohort A has completed Part 1. Part 2 will be an open-label, flexible-dose extension for subjects completing Part 1 of the study.

Part 1 will consist of a 4-week baseline, 2-week titration, 12-week maintenance, and 2-week taper or transition period. The 4-week Baseline Period will consist of the establishment of initial eligibility during a screening visit to include an assessment of cardiac parameters (ECG and ECHO), followed by an observation period where subjects will be assessed for baseline seizure frequency based on recordings of daily seizure activity entered into a diary. Upon completion of the Baseline Period, subjects who qualify for the study will be randomized (1:1:1) in a double-blind manner to receive 1 of 2 doses of ZX008 (0.2 mg/kg/day, 0.8 mg/kg/day; maximum dose: 30 mg/day) or placebo. Randomization will be stratified by weight (<37.5 kilograms [kg],  $\ge 37.5$  kg) to ensure balance across treatment arms, and at least 25% of subjects will be in each weight group. All subjects will be titrated to their blinded randomized dose over a 2-week Titration Period. Following titration, subjects will continue treatment at their randomly assigned dose over a 12-week Maintenance Period. Total treatment time from the beginning of the Titration Period through the end of the Maintenance Period is 14 weeks. Subjects will have ECG and ECHO assessments at weeks 6 and 14 during the Maintenance Period. At the end of the Maintenance Period (or early discontinuation), all subjects will undergo a 2-week taper or transition period (Post-Dosing Follow-Up) depending on whether they exit the study or are enrolled in Part 2, the long-term open-label extension, respectively. A follow-up ECG and ECHO will be performed after study drug discontinuation for early termination, or for those subjects who complete the study but do not enter the openlabel extension (Part 2), as outlined in Table 9.

Part 2 is an open-label, long-term safety study of ZX008 for subjects who have successfully completed 14 weeks of treatment (titration + maintenance) in Part 1, are candidates for continuous treatment for an extended period of time, have met the Selection Criteria for Part 1 (except for criteria related to seizure frequency), and signed informed consent/assent forms prior to the start of Part 2. Subjects who have not completed the entire 14 weeks of treatment in Part 1 may be eligible to participate in Part 2 on a case-by-case basis and only following sponsor approval. Other requirements for participation in Part 2 are described in Section 4.3. Part 2 will consist of a 12-month Open-Label Extension (OLE) Treatment Period and a 2-week Post-Dosing Period. Thus, subjects who complete 12 months of OLE in Part 2 will have been


treated with ZX008 for at least 70 weeks (including their participation in both Part 1 and Part 2). If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary. Up to 5 annual extensions can be applied, for a total treatment time of 72 months in the OLE. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk.

During Part 2 all subjects will be treated initially with 0.2 mg/kg/day for 1 month to assess effectiveness of this dose in all study subjects and determine the minimally effective dose. After 1 month at a dose of 0.2 mg/kg/day, the investigator may adjust the dose for each subject based on effectiveness and tolerability. Dose changes should be made in maximum increments of 0.2 mg/kg/day, to a maximum of 0.8 mg/kg/day but not to exceed total dose of 30 mg/day. During the 12-month OLE subjects will have ECG and ECHO assessments at months 1, 3, 6, and 9, and at the end of study visit. In the event the OLE is extended, subjects will continue to have ECG (if clinically indicated) and ECHO assessments every 6 months until the end of their participation in the study. See Section 5.5 for instructions on dosing and dose adjustments.

A follow-up ECG and ECHO will be performed after study drug discontinuation for early termination and for those subjects who complete Part 2, as outlined in Table 11. Subjects who transition to commercially available ZX008 will not return for these follow-ups, but must have an ECHO within 3 to 6 months of the transition date and will have follow-up ECHOs within required timeframes while on commercial drug supply.

In both Part 1 and the first 12 months of Part 2, parents/caregivers will use a diary every day to record the number of seizures, type of seizures, time and duration of seizures, whether the seizure resulted in a drop, dosing of study drug, and use of rescue medication.

A schedule of assessments for Part 1 is provided in Table 1 and for Part 2 in Table 2.

# 3.2 NUMBER OF SUBJECTS

Approximately 340 subjects will be screened to obtain 250 subjects randomized into Part 1 Cohort A (75 subjects per treatment arm), and at least 30 (and up to 50) subjects will be randomized into Part 1 Cohort B. The number of screened subjects may exceed 340 depending on the screen fail rate. Each clinical site will not randomize more than a maximum of 15 subjects without prior consent from the sponsor.

#### 3.3 STUDY DURATION

The duration of participation in the study for an individual subject is expected to be up to 20 weeks in Part 1 to include:

- Baseline Period 4 weeks
- T+M Period 14 weeks
- Taper/Transition Period 2 weeks after


Subjects who do not enroll in the open-label extension (Part 2) will undergo a taper off of study medication; eligible subjects who enroll in the open-label extension will undergo a 2-week transition period

Subjects who enroll in Part 2 will have the option to receive ZX008 for up to 72months (plus a 2-week taper at the end of the open-label extension), or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever occurs first

Follow-up cardiovascular safety assessments, including ECG and ECHO, will be performed following the last dose of study medication for all subjects that do not transition to commercial drug, regardless of whether they complete the entire study or terminate early. These follow-ups will occur 3 months following the last dose of study medication for any subject taking the medication for 2-13 weeks, and 3 and 6 months following the last dose for any subject taking the medication for >13 weeks. If there are any findings at a post-dose follow-up, another follow-up will be repeated every 3 months until resolved or stabilized. Subjects who transition to commercially available ZX008 will not return for a follow-up after EOS/ET or a cardiac follow up after last dose but must have had an ECHO within 3 to 6 months before the transition date and will have follow-up ECHOs within required timeframe while on commercial drug supply.

The study schema is shown in Figure 1.

Figure 1; Study Schema



#### 3.4 NUMBER OF STUDY CENTERS

The study expects to use up to approximately 80 research centers from North America, Europe, Japan, or Australia. Additional study centers within or outside of these geographic areas may be added if enrollment cannot be completed in a timely manner. Sites also may be closed if they fail to enroll.


# 3.5 RATIONALE FOR STUDY DESIGN AND CHOICE OF TREATMENT GROUPS

It is recognized that performing clinical studies in young children or in subjects with reduced cognitive capacity presents particular practical and ethical issues. However, given the seriousness of LGS, and the possible consequences of current inadequate treatments, the inclusion of children with LGS and adults with LGS who may have intellectual disability in this study is considered justified. Eligible subjects include males and females between 2 and 35 years of age inclusive. Because an accurate diagnosis of LGS is difficult in children younger than 2 years, and seizures that result in drops may not be accurately counted in this age group, children younger than 2 years are not included. Although seizures persist into adulthood, the primary seizure types and the treatment setting may differ, thus adults older than 35 years have not been included in this protocol.

Stratifying the randomization by weight is considered appropriate since the daily dosage of ZX008 increases with weight up to a maximum of 30 mg/day. The two strata in the study will be subjects who weigh less than 37.5 kg and subjects who weigh 37.5 kg or more. The study design has incorporated a titration period to enable subjects randomized to the high dose group adequate time to acclimate to this dose. Following the Titration Period, subjects will enter a 12-week Maintenance Period where they will continue on their randomized dose for the remainder of the study. The 12-week duration of the Maintenance Period is in keeping with the current standard study duration for evaluating the efficacy of chronic medications. Given the individual variability in seizure frequency and seizure type in this patient population, the primary endpoint, which seeks to compare an appropriate baseline of motor seizure that can result in a drop frequency to the motor seizure that can result in a drop frequency following treatment, is an appropriate primary endpoint for efficacy in this population.

Subjects will receive investigational medicinal product (IMP; ZX008 or placebo) in addition to their existing antiepileptic medications at their stable doses throughout the entire Part 1. Thus, subjects receiving placebo will not be denied active therapy; they will continue to receive their existing medications at the exact same dosages. As the principal study measurement (seizures that result in drops) might be considered subjective, a double-blind study design will prevent subjective bias. Upon completion of Part 1, eligible subjects will be able to receive ZX008 in Part 2, the open-label extension, for up to 5 additional years of treatment.

# 3.6 RATIONALE FOR STUDY DESIGN AND CHOICE OF TREATMENT GROUPS

Initial enrollment in Study 1601 was planned at up to 115 study sites in North America, Europe, Australia, and Japan. During the first 14 months of enrollment (ie, between November 2017 and January 2019), 50% of patients were randomized. During the next 5 months of enrollment (ie, between February 2019 and June 2019), enrollment proceeded faster than projected, with the remaining 50% of patients being randomized across a total of 70 active sites.

The speed of enrollment signifies the strong need for new medications for patients with LGS. Amending the Study 1601 protocol to split enrollment into 2 cohorts -- Cohort A (randomized


subjects from North America, Europe, and Australia) and Cohort B (randomized subjects from Japan only) -- and pre-specifying the primary analysis endpoint in the protocol and statistical analysis plan to include only subjects from Cohort A allows analyses to be conducted on a suitable number of subjects that are in accordance with the sample size estimations. Moreover, this approach allows evaluation of ZX008 in a Japanese population as part of a global clinical study while adhering to the requirements of the sample size estimation. The number of subjects in Japan will be increased from 15 to at least 30 (with the possibility to include up to 50) in order to provide a suitable sample for comparison, acknowledging that the speed of enrollment in Japan could mimic that of the other countries.

Japan has a large patient population with a high unmet medical need. Cultural differences between Japanese patients and Western patients are well documented in the literature. Moreover, due to operational challenges in clinical trial conduct, patients in Japan are typically not included in global studies, and when they are, it is often in very small numbers proportionally. Analyzing Cohorts A and B independently enables a properly powered primary analysis on Cohort A while providing the opportunity to increase enrollment in Japan in Cohort B, thus allowing for a more substantial comparison of safety and efficacy between Japanese patients and non-Japanese patients.

# 3.7 PREMATURE TERMINATION OF STUDY

The sponsor can terminate the study prematurely at any time for medical, ethical, or administrative reasons at individual or at all study sites. The investigator will be notified in writing, outlining the reasons for the termination. Instructions will be provided if assessments beyond those described in the study protocol need to be conducted.

The Independent Data Safety Monitoring Committee (IDSMC) may request that the study be terminated after review of the safety information at any time during the study.

If the study is terminated prematurely for any reason, the investigator should promptly inform the subjects participating at his or her study site and should ensure that appropriate follow-up care is available and that End-of-Study procedures are conducted, as described in Section 6.1.2.9 and Section 6.2.4.

All study materials including IMP (unless prior approval for onsite destruction is granted by sponsor) and completed, partially completed, and blank documentation, except documents needed for archiving requirements, will be returned to the sponsor. The study monitor will ensure that any outstanding data clarification issues and queries are resolved, and that all study records at the study site are complete.

In accordance with applicable regulatory requirements, the sponsor will promptly inform the competent regulatory authorities of the termination and its reason(s), and the investigator or sponsor will promptly inform the Independent Ethics Committee (IEC)/IRB.

#### 3.8 STUDY MONITORING PROCEDURES

#### 3.8.1 Independent Data Safety Monitoring Committee

The IDSMC is an independent advisory body that monitors participant safety, data quality and progress of the clinical trial. The IDSMC charter will outline the roles and responsibilities of the committee and guide its operations and frequency of meetings. The IDSMC will consist of


individuals external to the sponsor who have relevant clinical trial expertise and experience in safety assessment.

At regularly defined intervals, the IDSMC will convene to review and monitor study progress, AEs and SAEs, other measures of safety such as ECGs or ECHOs, and efficacy data as dictated by the charter.

#### The IDMSC will:

- Be responsible for providing recommendations to the sponsor surrounding study conduct
  matters that affect safety. The IDMSC will review the data for the development of heart
  valve disease and pulmonary hypertension as they occur on a case-by-case basis and at
  regular meetings.
- Review safety data at ad hoc time points and identify if significant safety concerns arise during the study.
- Review data that may affect subject continuation.
- Make recommendations regarding the continuation, suspension, or termination of the study.

#### 3.8.2 International Cardiac Advisory Board (ICAB)

The ICAB is an advisory body to the sponsor that assists in monitoring cardiac safety of the ZX008 clinical trials and provides advice to the IDMSC. The ICAB consists of individuals external to the sponsor who have relevant experience in cardiology, pediatric cardiology, and echocardiography. The ICAB will advise the sponsor and the IDSMC on the cardiac safety monitoring plan, including alert criteria and decision pathway for subject management relative to cardiac safety in the clinical studies of ZX008 when requested. ICAB members also provide secondary review or adjudication of ECHOs and ECGs, as well as risk assessment, as needed.


#### 4. SELECTION OF STUDY POPULATION

The study population will be selected on the basis of the inclusion and exclusion criteria described in the sections below. Before evaluating these criteria and deciding on the eligibility of subjects to participate in the study, it is important that the investigator is familiar with the safety profile of ZX008 by referring to the Investigator's Brochure, as supplied by the sponsor. Subjects receiving concomitant STP are not prohibited from study participation. For these subjects the maximum dose will be 0.5 mg/kg/day, with a maximum 20 mg/day, or equivalent placebo volume. For analyses purposes these subjects will be grouped with subjects randomized to 0.8 mg/kg/day. The dose of 0.5 mg/kg/day (maximum 20 mg/day) was selected for concomitant administration with STP based on the predicted effects of concomitant STP on ZX008 and the dose that best matches the exposure for the reference dose (ie, 0.8 mg/kg/day with a maximum of 30 mg/day, in the absence of STP). Both the mg/kg and maximum dose were modified to ensure the best match of exposure in young children (0.5 mg/kg/day) as well as to ensure that individual older patients did not have excursions in exposure (20 mg/day).

#### 4.1 PART 1

#### 4.1.1 INCLUSION CRITERIA

Subjects meeting all of the following inclusion criteria may be enrolled into the study:

- 1. Subject is male or non-pregnant, non-lactating female, age 2 to 35 years, inclusive as of the day of the Screening Visit. Female subjects of childbearing potential must not be pregnant or breast-feeding. Female subjects of childbearing potential must have a negative urine or serum pregnancy test at screening. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control (see Section 4.4), which includes abstinence, while being treated on this study and for 90 days after the last dose of study drug.
- 2. Subject must have a diagnosis of Lennox-Gastaut syndrome, where seizures that result in drops are not completely controlled by current antiepileptic treatments. (Subjects without a formal diagnosis may still be enrolled at sponsor discretion if all other criteria are met.)
- 3. Subjects must meet all of the following 4 criteria for Lennox-Gastaut syndrome, as defined in this protocol:
  - a. Onset of seizures at 11 years of age or younger.
  - b. Multiple seizure types (must include TS or TA), including countable motor seizures that result in drops. Countable motor seizure types eligible for inclusion are: GTC, TS, CS, AS, FS with observable motor symptoms, and MS that result in a drop.
  - c. Abnormal cognitive development.
  - d. Evidence of EEG in the medical history that shows abnormal background activity accompanied by slow spike and wave pattern <2.5 Hz. (Acceptable evidence includes a copy of the EEG trace, EEG report, or physician note that appropriately describes the EEG findings.)


- 4. Subject must have had at least 8 drop seizures in the last 4 weeks prior to Screening (minimum of 4 drop seizures in the first two weeks and 4 in the last two weeks before baseline), by parent/guardian report to investigator or investigator medical notes
- 5. Receiving at least 1 concomitant AED and up to 4 concomitant AEDs, inclusive. KD and VNS are permitted but do not count towards the total number of AEDs. Rescue medications for seizures are not counted towards the total number of AEDs.
- All medications or interventions for epilepsy (including KD and VNS) must be stable
  for at least 4 weeks prior to screening and are expected to remain stable throughout the
  study.
- 7. Subject has been informed of the nature of the study and informed consent has been obtained from the legally responsible parent/guardian.
- 8. Subject has provided assent in accordance with Institutional Review Board (IRB)/Ethics Committee requirements, if capable.
- 9. Subject's parent/caregiver is willing and able to be compliant with diary completion, visit schedule and study drug accountability.

#### 4.1.2 EXCLUSION CRITERIA

Subjects who meet any of the following exclusion criteria must not be enrolled into the study:

- 1. Subject has a known hypersensitivity to fenfluramine or any of the excipients in the study medication.
- 2. Subject's etiology of seizures is a degenerative neurological disease.
- 3. Subject has a history of hemiclonic seizures in the first year of life.
- 4. Subject only has drop seizure clusters, where individual seizures cannot be counted reliably.
- 5. Subject has pulmonary arterial hypertension.
- 6. Subject has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke, or clinically significant structural cardiac abnormality, including but not limited to mitral valve prolapse, atrial or ventricular septal defects, patent ductus arteriusis (note: Patent Foramen Ovale or a bicuspid valve are not considered exclusionary).
- 7. Subject has current or recent history of Anorexia Nervosa, bulimia, or depression within the prior year that required medical treatment or psychological treatment for a duration greater than 1 month.
- 8. Subject has a current or past history of glaucoma.
- Subject has had an anoxic episode requiring resuscitation within 6 months of the Screening Visit.
- 10. Subject has moderate or severe hepatic impairment. Asymptomatic subjects with mild hepatic impairment (elevated liver enzymes < 3x ULN and/or elevated bilirubin <2x ULN) may be entered into the study after review and approval by the Medical Monitor in conjunction with the sponsor, in consideration of comorbidities and concomitant medications.
- 11. Subject has severe renal impairment (estimated glomerular filtration rate <30mL/min/1.73m<sup>2</sup>)
- 12. Subject is receiving concomitant therapy with: centrally-acting anorectic agents; monoamine-oxidase inhibitors; any centrally-acting compound with clinically


appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; other centrally-acting noradrenergic agonists, including atomoxetine; or cyproheptadine (see Appendix 1 for a list of prohibited medications). (Note: Short-term medication requirements for prohibted medications will be handled on a per case basis by the Medical Monitor.)

- 13. Subject has positive result (as defined in the laboratory manual) on urine or serum tetrahydrocannabinol (THC) Panel or whole blood cannabidiol (CBD) at the Screening Visit.
- 14. Subject is taking felbamate for less than 1 year prior to screening and/or does not have stable liver function and hematology laboratory tests, and/or the dose has not been stable for at least 60 days prior to the Screening Visit.
- 15. Subject is known to be human immunodeficiency virus (HIV) positive.
- 16. Subject is known to have active viral hepatitis (B or C)..
- 17. Subject is currently receiving an investigational product.
- 18. Subject has participated in another clinical trial within the past 30 days (calculated from that study's last scheduled visit). Participation in non-treatment trials will be reviewed by the Medical Monitor.
- 19. Subject is at imminent risk of self-harm or harm to others, in the investigator's opinion, based on clinical interview and responses provided on the Columbia-Suicide Severity Rating Scale (C-SSRS). Subjects must be excluded if they report suicidal behavior in the past 6 months as measured by the C-SSRS at Screening or Baseline, which includes suicidal ideation with intent and plan (Item #5). If a subject reports suicidal ideation on Item 4 without specific plan, and the investigator feels that the subject is appropriate for the study considering the potential risks, the investigator must document appropriateness for inclusion, and discuss with the parent/caregiver to be alert to mood or behavioral changes, especially around times of dose adjustment.
- 20. Subject is unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
- 21. Subject is institutionalized in a general nursing home (ie, in a facility that does not provide skilled epilepsy care).
- 22. Subject does not have a reliable caregiver who can provide seizure diary information throughout the study.
- 23. Subject has a clinically significant condition, including chronic obstructive pulmonary disease, interstitial lung disease, or portal hypertension, or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Screening Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

#### 4.2 RANDOMIZATION INCLUSION CRITERIA

Subjects must meet all of the inclusion criteria and none of the exclusion criteria above and meet the following criteria in order to be randomized:

- 1. Subject has been approved for study inclusion by the Epilepsy Study Consortium.
- 2. Subject does not have an exclusionary cardiovascular or cardiopulmonary abnormality based on ECHO, ECG or physical examination and is approved for entry by the central cardiac reader. Exclusionary abnormalities include, but are not limited to:


- a. Trace or greater mitral or a ortic valve regurgitation in subjects ≤18 years of age
- b. Mild or greater mitral or a rtic valve regurgitation in subjects >18 yrs of age
- c. Possible signs of pulmonary hypertension with abnormal or greater than upper range of normal values
- d. Evidence of left ventricular dysfunction (systolic or diastolic)
- 3. Subject demonstrates a stable baseline with  $\geq 2$  seizures per week resulting in drops during the 4-week Baseline Period.
- 4. Subject's parent/caregiver has been compliant with diary completion during the Baseline Period, in the opinion of the investigator and sponsor.

#### 4.3 PART 2

To be included in Part 2:

- 1. Subjects must continue to meet the Selection Criteria for Part 1 (except for criteria related to seizure frequency). If a subject entering Part 2 does not meet Randomization Criteria 2 regarding cardiovascular abnormalities, Section 8.9.1 Follow-up of Cardiovascular Findings will be applied to determine eligibility to continue into Part 2.
- 2. All subjects must have satisfactorily completed Part 1 of the study in the opinion of the investigator and the sponsor.
- 3. Review of inclusion and exclusion criteria and written informed parental or guardian consent and assent of minors (if the subject is capable of providing assent) for Part 2 must be obtained before a subject can start any of the Part 2 Visit 15 procedures.
- 4. Subjects must, in the medical opinion of the Investigator, be candidates for continued treatment for an extended period of time with ZX008. Candidates for continuous treatment should not meet Discontinuation criteria listed in Section 4.5 and should not meet the following criteria:
  - Clinically meaningful worsening of seizures, judged by Investigator or subject/caregiver such that treatment outside of the protocol and other than ZX008 is assumed to be in the subject's best interest. A clinically meaningful worsening is an increase in frequency, severity or duration of existing seizures, or (in some cases) emergence of a new seizure type. Frequent or increased use of rescue medication may be considered indicative of worsening.
  - Clinically significant clinical laboratory findings (e.g. elevated ALT levels, decrease in platelet count, etc. that are CTCAE Grade 3 or higher) in subjects with no prior relevant history, that were not present during Baseline, are confirmed by a repeat test within a week, and not attributable to other concomitant medications.
  - Weight loss >15% during the T+M period that has not stabilized and is considered, in the opinion of the Investigator, detrimental to continuing treatment with ZX008.
- 5. Those subjects who do not complete the 12-week Maintenance Period of Part 1 may, on a case-by-case basis, be eligible for entrance after consideration of the circumstances of the early termination and the potential benefit-risk of continued participation in a


ZX008 trial. The decision whether to permit participation in Part 2 for subjects who do not complete Part 1 resides solely with the sponsor, will require a formal request for early Part 2 continuation to be made by the Investigator as well as an evaluation of risk/benefit. The Sponsor who may consult with the site investigator, the ICAB and/or the IDSMC, and take into consideration evidence of the following for approval:

- a. The subject is experiencing a worsening in condition that is not likely to be related to Part 1 treatment, in the opinion of the Investigator
- b. The subject has progressed at least half-way through Part 1 (i.e. Visit 8)
- c. The subject has been compliant with assessments and requirements of Part 1
- d. The subject does not exhibit other contraindications to initiating open-label treatment

#### 4.4 SUBJECTS OF REPRODUCTIVE POTENTIAL

Male subjects who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception from the time of informed consent until 90 days after the last dose of study drug.

The following methods are acceptable:

- Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
  - o oral
  - o intravaginal
  - o transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation:
  - o oral
  - o iniectable
  - o implantable intrauterine device
  - o intrauterine hormone-releasing system
- Surgical sterilization (vasectomy or bilateral tubal occlusion)

Female subjects who are not of childbearing potential do not need to use any methods of contraception. A woman is considered of childbearing potential, unless they are at least 2 years post-menopausal or permanently sterile, or if she has not yet reached menarche. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Female subjects who are sexually active and are of childbearing potential must use, with their partner, an approved method of highly effective contraception from the time of informed consent until 90 days after the last dose of study drug.

The following methods are acceptable:

- Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation and a barrier method (ie, condom for male partner):
  - o oral
  - o intravaginal


- o transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation and a barrier method (ie, condom for male partner):
  - o oral
  - o injectable
  - o implantable intrauterine device
  - o intrauterine hormone-releasing system
- Surgical sterilization (vasectomy or bilateral tubal occlusion)

Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, they, with their partner, they must comply with the contraceptive requirements detailed above.

#### 4.4.1 Sperm and Egg Donation

Male subjects should not donate sperm and female subjects should refrain from egg donation for the duration of the study and for at least 90 days after the last day of study medication administration.

#### 4.4.2 Pregnancy

Subjects will be instructed that if they/their partner become pregnant during the study this should be reported to the investigator. The investigator should also be notified of pregnancy occurring during the study but confirmed after completion of the study. In the event that a subject/subject's partner is subsequently found to be pregnant after the volunteer is included in the study, then consent will be sought from the partner and, if granted, any pregnancy will be followed and the status of mother and/or child will be reported to the sponsor after delivery. Any subject reporting a pregnancy during the study will be withdrawn from the study drug by completing the taper schedule. All safety follow-up activities must be completed.

#### 4.5 REMOVAL OF SUBJECTS FROM THERAPY OR ASSESSMENT

While subjects are encouraged to complete all study evaluations, subjects may voluntarily withdraw from the study for any reason at any time. They may be considered withdrawn if they fail to return for visits, or become lost to follow-up for any other reason.

If premature withdrawal occurs for any reason, the investigator must make a genuine effort to determine the primary reason for a subject's premature withdrawal from the study and record this information on the electronic case report form (eCRF). All subjects who withdraw from the study with an ongoing AE must be followed until the event is resolved or deemed stable. If a subject withdraws prematurely after dosing, all data to be collected prior to discharge from the clinical site should be collected at the time of premature discontinuation or at the scheduled discharge.

For subjects who are lost to follow-up (ie, those subjects whose status is unclear because they failed to appear for study visits without stating an intention to withdraw), the investigator should show "due diligence" by documenting in the source documents the steps taken to


contact the subject (eg, dates of telephone calls, registered letters).

Subjects must be discontinued from the study for the following reasons, if deemed appropriate by the sponsor or investigator:

- 1. Development of signs or symptoms indicative of cardiac valvulopathy or regurgitation (mitral, aortic, tricuspid, pulmonary valves), or pulmonary hypertension for which IDSMC, in consultation with cardiac readers and the investigator believe the benefit of continued participation does not outweigh the risk.
- 2. Subject is found to have entered the clinical investigation in violation of the protocol.
- 3. Subject requires or starts using unacceptable or contraindicated concomitant medications, or currently utilized chronic daily seizure therapy is changed.
- 4. Subject's condition changes after entering the clinical investigation so that the subject no longer meets the inclusion criteria or develops any of the exclusion criteria.
- 5. Subject is noncompliant with procedures set forth in the protocol in an ongoing or repeated manner.
- 6. Subject experiences an AE that warrants withdrawal from the clinical investigation.
- 7. Clinically significant worsening of seizures, judged by investigator or subject/caregiver such that treatment outside of the protocol and other than ZX008 is assumed to be in the subject's best interest. Frequent or increased use of rescue medication may be considered indicative of worsening.
- 8. An "actual suicide attempt" as classified by the Columbia-Suicide Severity Rating Scale (C-SSRS).
- 9. It is the investigator's opinion that it is not in the subject's best interest to continue in the study.
- 10. Subject is found to be pregnant while on study. Subject will be withdrawn following the taper schedule; all safety follow-up activities must be completed.

Discontinuation decisions will be made at each participating site by the site investigator. Discontinuations due to development of cardiovascular or cardiopulmonary complications are to be made by the IDMSC.

If feasible, the process of discontinuation should be discussed with the Medical Monitor. The decisions regarding the discontinuation of the investigational therapy, whether the study medication should be stopped immediately or tapered should be discussed with the Medical Monitor, but final decisions about the process will remain at the discretion of the site principal investigator.

Subjects who are discontinued from the clinical investigation for any reason will not be replaced.

Subjects may withdraw their consent to participate in the study at any time without having to justify the reason for doing so. The decision to withdraw consent and discontinue participation in the study will not prejudice the subject's future medical treatment in any way.

Subjects <u>must</u> be discontinued from receiving ZX008 and/or participating in any further study procedures under the following circumstances:

The subject or the subject's legally authorized representative wishes to discontinue


participation in the study.

- The investigator advises that the subject's safety or well-being could be compromised by further participation in the study.
- The sponsor requests that a subject discontinues participation in the study (eg, due to suspicion of fraud, multiple enrollments in clinical studies, lack of compliance).

In the event that the study is terminated prematurely then the procedure for termination should be followed as described in Section 3.7. Concern for the interests of the subject will always prevail over the interests of the study.

The reason for, and date of discontinuation from participation in the study must be recorded in detail in the eCRF and in the subject's medical records (eg, AEs, lack of compliance, lost to follow-up, etc). If possible, the subject/subject's legally authorized representative should confirm his decision in writing.

The investigator will attempt to complete all procedures usually required at the end of the study at the time when the subject's participation in the study is discontinued or as close as possible to that time. Specific procedures required for each Part of the study are described in Section 6.1.2.9 and Section 6.2.4. As far as possible, a complete final examination must be performed on all subjects who do not complete the study according to the study protocol.

Data collected until the time a subject discontinues participation in the study will be handled in the same manner as data for subjects completing the study. Where possible, further information will be collected if any AEs are experienced by a subject after discontinuing participation in the study.

#### 4.6 TERMINATION OF THE CLINICAL STUDY

If the investigator, the sponsor, the Medical Monitor, or the IDSMC becomes aware of conditions or events that suggest a possible hazard to subjects if the clinical study continues, then the clinical study may be terminated. The decision to terminate the study lies solely with the sponsor. The clinical study may be terminated at the sponsor's discretion at any time also in the absence of such a finding.

Conditions that may warrant termination of the clinical study include, but are not limited to:

- The discovery of an unexpected, relevant, or unacceptable risk to the subjects enrolled in the clinical study.
- Failure to enroll subjects at the required rate.
- A decision of the sponsor to suspend or discontinue development of ZX008.

#### 4.7 REPLACEMENT OF SUBJECTS

Enough subjects will be enrolled in Part 1 of the trial to ensure that approximately 250 subjects are randomized into the T+M Period of Part 1 Cohort A, and at least 30 subjects are randomized into Part 1 Cohort B. Randomized subjects will not be replaced.


#### 5. INVESTIGATIONAL MEDICINAL PRODUCT INFORMATION

ZX008/matching placebo will be administered in the current study. A brief description of the ZX008 product is provided below (Table 4).

**Table 4:** Investigational Medicinal Product – ZX008

| | Study Product |
|---|---|
| Substance Code | ZX008 |
| Active Substance (INN) | Fenfluramine Hydrochloride |
| Trade Name | Not applicable |
| Formulation (including dosage form and strength) | Solution 1.25, 2.5, and 5 |
| mg/mL Route/Mode of Administration | Oral |
| Manufacturer | PCI Pharma Services on behalf of Zogenix |
| | International Limited |

#### 5.1 IDENTITY OF INVESTIGATIONAL MEDICINAL PRODUCT

ZX008 drug product is an oral aqueous solution of fenfluramine hydrochloride buffered to pH 5 and provided in concentrations of 1.25 mg/mL, 2.5 mg/mL, and 5 mg/mL. The excipients selected have been approved for use in the formulations of currently marketed drug products and are considered to be safe. The solution formulations will be suitably flavored, and will contain preservatives and a thickening agent. The product is sugar free and is intended to be compatible with a KD.

The formulation for Part 1 will be provided in bottles with tamper-evident, child-resistant caps. The clinical trials material will be supplied in 1 bottle size with nominal fill volume of 120 mL. Matching placebo also will be provided. Doses to be studied include ZX008 0.2 mg/kg/day and ZX008 0.8 mg/kg/day divided into two daily (BID) doses, up to a maximum of 30 mg/day (subjects taking concomitant STP will receive 0.5 mg/kg/day, up to a maximum of 20 mg/day, or equivalent volume of placebo). An intermediate dose of 0.4 mg/kg/day will be used for titration. The concentration of ZX008 oral solution received by subjects (1.25 mg/mL, 2.5 mg/mL, and/or 5 mg/mL) will be randomized across the 3 available concentrations in order to ensure blinding.

For Part 2 flexible dosing will be studied, up to 0.8 mg/kg/day divided into two daily doses, up to a maximum of 30 mg/day (subjects taking concomitant STP will receive up to 0.5 mg/kg/day, up to a maximum of 20 mg/day). ZX008 drug product will be provided in a concentration of 2.5 mg/mL in 1 bottle size with nominal fill volume of 120 mL.

#### 5.1.1 Labeling and Packaging

The ZX008 product will be packaged and labeled according to current International Conference on Harmonization (ICH), Good Manufacturing Practices (GMP), and Good Clinical Practices (GCP) guidelines, and national legal requirements.

Dosing directions for the product can be found in the Pharmacy Manual for the study subjects and for the investigator.


# 5.2 DESCRIPTION OF REFERENCE TREATMENT, COMPARATOR, AND/OR PLACEBO

Placebo solution is identical in aspect and composition to ZX008 and is composed of identical ingredients used in the ZX008 formulation, except that it does not contain the active ingredient, fenfluramine hydrochloride. Subjects randomized to placebo will receive concentration equivalent volumes of investigational product that does not include the active ingredient.

No comparators or reference treatments will be used.

#### 5.2.1 Labeling and Packaging

Placebo solution will be packaged in an identical manner to ZX008. The matching placebo product will be packaged and labeled according to current ICH, GMP, and GCP guidelines, and national legal requirements.

Dosing directions for the product can be found in the IMP handling instructions for the study subjects and for the investigator.

#### 5.3 SHIPMENT AND STORAGE

IMP will be supplied to the study sites by the sponsor or its delegate

All IMP will be transported, received, stored, and handled strictly in accordance with the container or product label, the instructions supplied to the research site and its designated pharmacy, the site's standard operating procedures, and applicable regulations. IMP must be stored separately from normal hospital or practice inventories, in a locked facility with access limited to the investigator and authorized personnel. The investigator must ensure that the IMP is dispensed only to subjects enrolled in this study according to this study protocol.

Appropriate storage temperature and transportation conditions will be maintained for the study drug from the point of manufacture up to delivery of the study drug. Study medication must be stored at 15-25°C (59-77°F) with excursions of 5-40°C (41-104°F) permitted; do not refrigerate or freeze.

Storage and handling instructions of the IMP maintained at the subject's home are described in the subject's IMP handling instructions.

All unused IMP will be saved by the site for final disposition according to the sponsor's directive.

## 5.4 IMP ACCOUNTABILITY

The investigator or delegate will confirm receipt of all shipments of the IMP in writing using the receipt form(s) provided by the sponsor or vendor.

Assignment of ZX008 or placebo to the subject will be handled through an interactive voice randomization (IVR)-or Interactive Web Response (IWR) platform. The investigator or delegate will be required to register the subject through IVR/IWR and all study medication will be assigned to the subject through the IVR/IWR. The IVR/IWR will also maintain a log of all received and dispensed medication.

All supplies must be accounted for throughout the study using the drug accountability form


provided by the sponsor before the start of the study. Drug accountability is the process of documenting all aspects of IMP receipt, storage, use, and disposition so that a full accounting of each unit can be made. This includes administration, and return and/or destruction of IMP. At the end of the study, the dated and signed (by the investigator or delegate, eg, pharmacist)

Records for the delivery of the IMP to the study site, the inventory at the study site, the use by each subject (use by subject will be documented in the subject diary), and the destruction are return of the IMP to the sponsor must be maintained by the records will include det records will include dates, quantities, batch numbers, and unique code numbers assigned to the IMP and to the subjects. The investigator must maintain records documenting that subjects. were provided with the doses of the IMP specified in this study protocol. Furthermore, the investigator must reconcile all IMPs received from the sponsor. The investigator must provide reasons for any discrepancies in drug accountability. Forms will be provided by the sponsor to ensure standardized and complete drug accountability.

#### 5.5 TREATMENT ADMINISTRATION

#### 5.5.1 Part 1: Randomization

Upon completion of the Baseline Period in Part 1, subjects who qualify for the study will be randomized (1:1:1) in a double-blind manner to receive 1 of 2 doses of ZX008 (0.2 mg/kg/day, 0.8 mg/kg/day; 30mg/day maximum [0.5 mg/kg/day; 20 mg/day maximum for subjects taking concomitant STP]) or placebo. The randomization will be stratified by weight ( $<37.5 \text{ kg}, \ge 37.5$ kg) to ensure balance across treatment arms, with a target of at least 25% in each weight group. Subjects will be assigned a randomization number by the IWR system upon confirmation that subject qualifies for enrollment in the Titration Period. Once a randomization number is assigned to a subject, the site will record the subject's initials and identification number on the corresponding study drug bottles. Each bottle will contain the appropriate concentration and volume of liquid to administer the assigned treatment (ZX008 0.2 mg/kg/day, ZX008 0.8 mg/kg/day [or 0.5 mg/kg/day for subjects taking concomitant STP], or placebo). ZX008 and placebo will be identical, thus rendering the study drug and placebo indistinguishable. For each IMP bottle and randomization number assigned, the following information will be recorded on the drug accountability form: subject initials, unique bottle number, date each bottle is assigned, and drug used and unused during the study.

#### 5.5.1.1 Blinding

The blinding scheme instituted for this study will ensure that the volume of study medication taken cannot be associated with the dose group, thus unblinding the study. This is achieved by random assignment of different concentrations of the ZX008 oral solution (1.25 mg/mL, 2.5 mg/mL, and/or 5 mg/mL) by the IWR system. The IWR system will instruct site personnel to the volume of oral solution to be administered based on that subject's weight. (Dose will be recalculated by the system based on weight once at the midpoint of the study.) During the Titration, Maintenance, and Taper/Transition Periods, the subjects and study personnel (investigators, clinical staff, personnel involved in data collection and analysis, the Medical Monitor, and the sponsor) will be blinded to the treatment allocation and to the concentration of


ZX008 oral solution. If an investigator feels the blind should be broken, he/she can do so when necessary for treatment decisions. However, the investigator should endeavor to discuss with the Medical Monitor or Sponsor's Medical Representative, if available. The blind should only be broken in the event the knowledge of whether the subject is on active study medication versus placebo is needed to determine course of medical treatment for the event. The subject will be discontinued from the clinical trial upon breaking of the blind and the decision whether the subject can enter Part 2 will rest with the Sponsor if the subject exited Part 1 prior to completion.

#### 5.5.2 Part 1: Titration Period

The investigator (or delegate) will dispense IMP only to subjects included in Part 1 of this study following the procedures set out in this study protocol. Subjects will be required to stay in the clinic for monitoring of adverse reactions until the investigator determines it is safe to leave. Those considered by the investigator to need further monitoring will be hospitalized until the investigator determines they can be safely discharged.

Study medication will be administered as equal doses BID in the morning and in the evening approximately 12 hours apart. Each dose should be separated by a minimum of 8 hours and a maximum of 12 hours. A missed dose of study medication may be taken later up to 8 hours before the next scheduled dose; otherwise, the missed dose should not be given.

If the parent/caregiver is unable to administer the full dose due to spillage (eg, dose was spilled during measuring, subject spit dose out during administration), he/she should attempt to give the full dose noting the extra amount used to fulfill the dose. If the subject vomits within the first 15 minutes of administration the dose may be readministered. **Care must be taken not to overdose.** If the amount spilled is not known, the parent/caregiver should not give additional medication to avoid potential overdose.

Administration of the IMP will be based on the randomized dose and subject's weight (kg) at Visit 3 (Part 1; Study Day -1). At Visit 8 (Part 1; Study Day 43), if the subject's weight (kg) has changed ±25% of the weight at Part 1; Study Day-1, the IMP dose will be recalculated. Subjects should be dosed using the oral dosing syringe provided.

In order to maintain the blind across all dose groups in Part 1 (Section 5.5.1.1) and allow step titration to the high dose, the dose for each subject will be titrated starting with a dose of ZX008 0.2 mg/kg/day (or placebo equivalent) BID. After 4 days at this dose level (Study Day 5), subjects randomized to the ZX008 0.8 mg/kg/day (or 0.5 mg/kg/day for subjects taking concomitant STP) group will increase their dose to 0.4 mg/kg/day (maximum 30 mg/day or 20 mg/day for subjects taking concomitant STP) while doses in the other two groups will remain constant. On Study Day 9, the dose for the 0.8 mg/kg/day group (or 0.5 mg/kg/day for subjects taking concomitant STP) will increase to the target dose or a maximum of 30 mg/day (or 20 mg/day for subjects taking concomitant STP). The titration is expected to take a total of 14 days (Table 5). A new bottle of IMP will be started by the subject at each level of the titration step. See Section 5.1 for more information about the volume of ZX008 or placebo to be administered. If a subject does not tolerate IMP during titration, slower titration may be considered after consultation with the Medical Monitor.


Table 5: Titration Algorithm for Part 1

| Randomized Group | Titration Step 1<br>Study Day 1-4 | Titration Step 2<br>Study Days 5-8 | Titration Step 3<br>Study Days 9-14 |
|---|---|---|---|
| ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day |
| ZX008 0.8 mg/kg/day<br>(0.5 mg/kg/day for subjects<br>taking concomitant STP) | ZX008 0.2 mg/kg/day | ZX008 0.4 mg/kg/day | ZX008 0.8 mg/kg/day<br>(0.5 mg/kg/day for subjects<br>taking concomitant STP) |
| Placebo | Placebo | Placebo | Placebo |
| Note: maximum daily dose of ZX008 is 30 mg (20mg for subjects taking concomitant STP) | | | |

#### 5.5.3 Part 1: Maintenance Period

After completion of the Titration Period, subjects will enter the Maintenance Period and continue to receive the randomized dose of ZX008 or placebo and be treated for an additional 12 weeks. Study medication will continue to be administered BID in the morning and in the evening, approximately 12 hours apart. Each dose should be separated by a minimum of 8 hours and a maximum of 12 hours. A missed dose of study medication may be taken later up to 8 hours before the next scheduled dose; otherwise, the missed dose should not be given.

# 5.5.4 Part 1: Taper Period (for subjects not entering Part 2)

Subjects who complete the Maintenance Period and will not be continuing into Part 2, the open-label extension, and subjects who discontinue from Part 1 early, will be tapered off of study medication. Study medication will be administered as equal doses BID in the morning and in the evening approximately 12 hours apart. Each dose should be separated by a minimum of 8 hours and a maximum of 12 hours. A missed dose of study medication may be taken later up to 8 hours before the next scheduled dose; otherwise, the missed dose should not be given. IMP should be administered using the oral dosing syringe provided.

If the parent/caregiver is unable to administer the full dose due to spillage (eg, dose was spilled during measuring, subject spit dose out during administration), he/she should attempt to give the full dose noting the extra amount used to fulfill the dose. If the subject vomits within the first 15 minutes of administration the dose may be readministered. **Care must be taken not to overdose.** If the amount spilled is not known, the parent/caregiver should not give additional medication to avoid potential overdose.

In order to maintain the blind across all dose groups, all subjects who do not continue into Part 2 will participate in a blinded dose-tapering procedure over the course of 8 days. On the first day of the tapering period subjects in the ZX008 0.8 mg/kg/day group (or 0.5 mg/kg/day for subjects taking concomitant STP) will decrease to a dose of ZX008 0.4 mg/kg/day BID (maximum 30 mg/day or 20 mg/day for subjects taking concomitant STP). After 4 days at this dose level (Study Day 5), subjects in this group will decrease their dose to 0.2 mg/kg/day. Subjects in the ZX008 0.2 mg/kg/day group will decrease their dose to placebo on the first day of tapering while doses in the placebo group will remain constant throughout the tapering procedure. On Study Day 9, all subjects will stop taking study medication. The taper is expected to take a total of 8 days (Table 6). A new bottle of IMP will be started by the subject at each level of the taper step.


**Table 6:** Taper Algorithm for Part 1

| Randomized Group | Taper Step 1 Day 1-4 after study completion or early termination | Taper Step 2 Days 5-8 after study completion or early termination |
|---|---|---|
| ZX008 0.2 mg/kg/day | Placebo | Placebo |
| ZX008 0.8 mg/kg/day<br>(0.5 mg/kg/day for subjects<br>taking concomitant STP) | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |
| Placebo | Placebo | Placebo |
| Note: maximum daily dose | of ZX008 is 30 mg. (20mg for subjects | s taking concomitant STP) |

#### 5.5.5 Part 1: Transition Period

Subjects who complete the Maintenance Period and will be continuing into the open-label extension (Part 2) will be transitioned from double-blind study medication to open-label ZX008 (Table 7).

All subjects entering the open-label extension (Part 2) will be transitioned from their blinded daily dose to the 0.2 mg/kg dose during the 2-week interval between Visits 12 and 15, without breaking the blind. The IWR system will assign two bottles of IMP to the subject, one for each step in the transition. A new bottle of IMP will be started by the subject at each level of the transition step. See Section 5.1 for more information about the volume of ZX008 or placebo to be administered.

**Table 7:** Transition Algorithm for Part 1

| Dose Group in Double- | Transition Step 1 | Transition Step 2 |
|---|---|---|
| Blind Study | Day 1-4 after Visit 12 | Days 5-14 after Visit 12 |
| ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day |
| ZX008 0.8 mg/kg/day | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |
| (0.5 mg/kg/day for subjects taking concomitant STP) | En o | |
| Placebo | ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day |
| Note: maximum daily dose of ZX008 is 30 mg (or 20 mg for subjects taking concomitant STP). | | |

Subjects who had been randomized to placebo increase their dose to 0.2 mg/kg/day beginning on Day 1 of the transition. The first dose should be taken in the clinic during Visit 12. Subjects will be required to stay in the clinic for monitoring of adverse reactions until the investigator determines it is safe to leave. Those considered by the investigator to need further monitoring will be hospitalized until the investigator determines they can be safely discharged. Subjects who had been randomized to 0.2 mg/kg/day will continue to receive that dose. Subjects who had been randomized to 0.8 mg/kg/day or were receiving the maximum dose of 30 mg/day (or subjects taking concomitant STP and randomized to 0.5 mg/kg/day; 20 mg/day maximum) decrease to a dose of ZX008 0.4 mg/kg/day, or a maximum of 30 mg/day (20 mg/day for subjects taking concomitant STP). After 4 days at this dose level (Day 5), these subjects will decrease their dose to 0.2 mg/kg/day. Subjects will report to the clinic on Day 14 for enrollment into the open-label extension.


Study medication will be administered as equal doses BID in the morning and in the evening approximately 12 hours apart. Each dose should be separated by a minimum of 8 hours and a maximum of 12 hours. A missed dose of study medication may be taken later up to 8 hours before the next scheduled dose; otherwise, the missed dose should not be given. Study medication should be administered using the oral dosing syringe provided.

If the parent/caregiver is unable to administer the full dose due to spillage (eg, dose was spilled during measuring, subject spit dose out during administration), he/she should attempt to give the full dose noting the extra amount used to fulfill the dose. If the subject vomits within the first 15 minutes of administration the dose may be readministered. Care must be taken not to overdose. If the amount spilled is not known, the parent/caregiver should not give additional medication to avoid potential overdose.

#### 5.5.6 Part 2: OLE Treatment Period

During the Part 2 OLE Treatment Period, all subjects will be treated initially with 0.2 mg/kg/day for 1 month to assess effectiveness of this dose in all study subjects. After 1 month at a dose of ZX008 0.2 mg/kg/day, the investigator may adjust the dose of each subject based on effectiveness and tolerability.

Administration of the initial IMP will be based on the 0.5 mg/kg/day (maximum 30 mg/day or 20 mg/day for subjects taking concomitant STP) dose and subject's weight recorded for Visit 15 (Part 2; Study Day 1). At Visits 19, 20, and 21 of Part 2 (Months 3, 6, and 9), if the subject's weight has changed  $\pm$  25% of the weight recorded for Visit 15, the IMP dose will be recalculated. Subjects will be dosed using the oral dosing syringe provided.

Dose increases should not occur earlier than every 14 days at each dose level. Dose increases may only occur after a review of the diary and reported AEs, and if, in the investigator's opinion, seizure frequency, severity, and/or duration indicates a change in medication regimen is warranted. Temporary dose decreases for tolerability can occur at the investigator's discretion, in dose amounts and frequency appropriate for the situation. Subsequent dose rechallenge should occur at the investigator's discretion in consultation with the Medical Monitor. ZX008 dose adjustments outside of these parameters should be discussed with the Medical Monitor and must be approved by the Sponsor prior to initiation.

If after approximately the midway point of the first 30 days on ZX008 0.2 mg/kg/day there is a clinically meaningful worsening in seizure type, frequency, and/or duration compared with the recent treatment in the core study, the investigator, in consultation with the Medical Monitor and approval of the sponsor, may increase the dose to 0.4 mg/kg/day (maximum 30 mg/day or 20 mg/day for subjects taking concomitant STP). A clinically meaningful worsening would be an increase in frequency, severity or duration of existing seizures, or (in some cases) emergence of a new seizure type. The description of clinical worsening must be documented in the source notes and case report form (CRF). Further increase to 0.8 mg/kg/day (maximum 30 mg/day or 0.5 mg/kg/day; maximum 20 mg/day for subjects taking concomitant STP) could also be undertaken for the same conditions after a minimum of 4 days on 0.4 mg/kg/day, if the condition has not stabilized on the 0.4 mg/kg/day dose. Dosing outside of the specified range (ie, up to 0.8 mg/kg/day [or 0.5 mg/kg/day for subjects taking concomitant STP]) may be considered after


consultation between the investigator and Medical Monitor and approval of the Sponsor; however, excursions over 30 mg/day (or 20 mg/day for subjects taking concomitant STP) are prohibited.

Study medication will be administered as equal doses BID in the morning and in the evening, approximately 12 hours apart. Each dose should be separated by a minimum of 8 hours and a maximum of 12 hours. A missed dose of study medication may be taken later up to 8 hours before the next scheduled dose; otherwise, the missed dose should not be given.

If the parent/caregiver is unable to administer the full dose due to spillage (eg, dose was spilled during measuring, subject spit dose out during administration), he/she should attempt to give the full dose noting the extra amount used to fulfill the dose. If the subject vomits within the first 15 minutes of administration the dose may be readministered. Care must be taken not to overdose. If the amount spilled is not known, the parent/caregiver should not give additional medication to avoid potential overdose.

#### 5.5.7 Taper Period

All subjects (those who complete the Part 2 OLE Treatment Period and those who discontinue from the study early) will be tapered off of study medication, unless they are transitioning to commercial drug.

The tapering scheme is a 2-step process as described in Table 8

Study medication will be administered as equal doses BID in the morning and in the evening, approximately 12 hours apart. Each dose should be separated by a minimum of 8 hours and a maximum of 12 hours. A missed dose of study medication may be taken later up to 8 hours before the next scheduled dose; otherwise, the missed dose should not be given. IMP will be administered using the oral dosing syringe provided.

Table 8. Taper Algorithm for Part 2

| Table 6: Taper Augustinia 1017 art 2 | | |
|---|---|---|
| | Taper Step 1 Days 1-4 after study | Taper Step 2 Days 5-8 after study completion |
| Current Dose | completion or early<br>termination | or early termination |
| 777000 0 2 /1 (1) | | NY . 11 11 |
| ZX008 0.2 mg/kg/day | Not applicable | Not applicable |
| ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day | Not applicable |
| ZX008 0.5 mg/kg/day | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |
| (for subjects taking | | |
| concomitant STP) | | |
| ZX008 0.6 mg/kg/day | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |
| ZX008 0.8 mg/kg/day | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |
| Note: maximum daily do | se of ZX008 is 30 mg (or 20 mg fo | or subjects taking concomitant STP). |


#### 5.6 PRIOR AND CONCOMITANT MEDICATION

All medications taken by a subject before receiving study medication (ie, during the Screening and Baseline Seizure Assessment Periods in Part 1) and stopped before the first administration of IMP are regarded as prior therapy and must be documented in the eCRF. Significant medications (eg, antibiotics) taken within 30 days prior to the Screening visit should also be captured. All prior and concomitant AEDs will be collected in the eCRF.

All medications taken by a subject after the first administration of IMP, including those that started before the first administration of IMP and are continuing, are regarded as concomitant medication and must be documented in the eCRF, including over-the-counter medication, herbal and vitamin/supplement preparations.

Subjects are required to take at least one concomitant AED during study participation. No new concomitant AEDs may be introduced while in this study without discussion with the Medical Monitor prior to initiation. Non-study medications and therapies (this does not include KD, VNS, and RNS) that are considered necessary for the subject's welfare and will not interfere with the response to the study medication may be given at the discretion of the investigator, informing the Medical Monitor as soon as possible.

It should be noted for any subject receiving hypoglycemic agents, the investigator should consider diabetic medication changes in the setting of weight loss and hypoglycemia.

#### Part 1

All subjects will continue to receive their existing AED(s) with the same doses throughout the Part 1 Double-blind Treatment Period. Every effort should be made to ensure that the regimen of existing medications remains stable during Part 1; any changes must be discussed with the sponsor prior to implementation. If a decrease in a concomitant AED is necessary to manage an AE, this must be discussed with the sponsor as soon as possible after implementation if not before implementation. Increases in dose or number of concomitant AEDs are not permitted during Part 1 of the study.

#### Part 2

During at least the first 6 months of the Part 2 OLE Treatment Period, subjects will continue to receive their existing AEDs at the same dose and frequency as prior to starting Part 2. However, once the subject has been stable on a ZX008 dose for at least 6 months with good seizure control, investigators will be allowed as per typical clinical practice to alter one or more other concomitant AED doses as deemed clinically appropriate. Subjects who achieve robust seizure control may be considered to decrease concomitant AEDs earlier than 6 months after review/discussion with the Medical Monitor and approval from the Sponsor. Concomitant AEDs may be withdrawn completely but all subjects must remain on a minimum of 1 concomitant AED plus ZX008. Addition of new concomitant AEDs must be discussed with and approved by the Medical Monitor prior to initiation. AED doses may be lowered for safety considerations at any time. All medication dose changes must be documented with a clinical explanation and


justification. Concomitant AED dose adjustments outside of these parameters should be discussed with the Medical Monitor prior to initiation.

#### **5.6.1** Vagal Nerve Stimulation

Subjects receiving treatment with a VNS may be included as long as the VNS has been in place for at least 6 months prior to entry into the study, the VNS battery is not due for replacement during the study, and stimulation parameters have been kept constant for 4 weeks prior to screening and must remain so throughout the study. VNS may not be the only anti-epileptic treatment (ie, it does not count as an AED but it does count as a treatment for LGS). The subject's use of VNS will be recorded in the eCRF.

During at least the first 6 months of the Part 2 OLE Treatment Period, VNS stimulation parameters will be kept constant. However, once the subject has been stable on a ZX008 dose for at least 6 months with good seizure control, investigators will be allowed as per typical clinical practice to alter VNS stimulation parameters as deemed clinically appropriate. All VNS stimulation parameter changes must be documented with a clinical explanation and justification. VNS stimulation parameter adjustments outside of these boundaries should be discussed with the Medical Monitor prior to initiation.

#### 5.6.2 Ketogenic Diet

Adherence to the KD, or a modified version of KD, is permitted during the study if the dietary habits were initiated more than 4 weeks prior to Screening and remain stable throughout the study. KD may not be the only anti-epileptic treatment (ie, it does not count as an AED but does count as a treatment for LGS). The subject's use of KD will be recorded in the eCRF.

During at least the first 6 months of the Part 2 OLE Treatment Period, the KD will be adhered to. However, once the subject has been stable on a ZX008 dose for at least 6 months with good seizure control, investigators will be allowed as per typical clinical practice to alter the KD as deemed clinically appropriate. All KD changes must be documented with a clinical explanation and justification. KD adjustments outside of these parameters should be discussed with the Medical Monitor prior to initiation.

#### 5.6.3 Rescue Medication for Seizures

The subject's usual or prescribed regimen and frequency of rescue therapy for seizures should be entered into the concomitant medication sections of the eCRF and identified as a rescue medication by selecting the appropriate box.

Use of rescue medication is permitted during the study and should be recorded on the eCRF (day, medication[s], dose[s]) and in the diary (day, timeframe associated with seizure episodes). Repeated administrations within the same episode should be recorded separately.

#### 5.6.4 Prohibited Concomitant Medications

Examples of concomitant medications in the classes prohibited are listed in Appendix 1 and summarized below. If medical necessity requires short-term use of one or more of these medications during the course of the study, please contact the Medical Monitor for approval.


- Felbamate is prohibited as a concomitant medication unless the subject has been on felbamate for at least 12 months prior to screening, has stable liver function and hematology laboratory tests, and the dose has been stable for at least 60 days prior to
- Drugs that interact with central serotonin: imipramine, monoamine oxidase inhibitors, selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, vortioxetine.

  Drugs that increase cardiovas
- Drugs intended to facilitate weight loss.
- Ergot alkaloids and their derivatives, including pergolide and cabergoline
- Phenylpropanolamine and other decongestants may be used for short-term use only.

#### 5.7 TREATMENT COMPLIANCE

dose, dosir.

eir used, partiall,

monitored by meas

pensation log and diary Each subject or parent/caregiver will record the dose, dosing frequency and IMP consumption in the subject's diary. Subjects will bring their used, partially used, and unused IMP to every study visit. Treatment compliance will be monitored by measuring the volume of IMP in these bottles and comparing to the dispensation log and diary records.

> 
## 6. VISIT SCHEDULE

## 6.1 Part 1

Study procedures for the Part 1 Double-blind Treatment Period will be conducted according to the Schedule of Assessments in Table 1. Time windows for all assessments in Part 1 are detailed in Table 9

**Table 9:** Time Windows for Assessments in Part 1

| Visit / Procedure | Time window (relative to scheduled visit / procedure) |
|---|---|
| Visit 1 (Clinic; Study Day -29 to -28 or -28 to -27): | Not applicable |
| Visit 2 (Phone; Study Day -15) | ± 3 days |
| Visit 3 (Clinic; Study Day -1; Randomization) | + 4 days <sup>a</sup> |
| Visits 4, 5 (Phone: Study Days 4, 8) | ± 3 days |
| Visit 6 (Clinic; Study Day 15) | ± 4 days |
| Visit 7 (Phone: Study Day 29) | ± 4 days |
| Visit 8 (Clinic; Study Day 43) | ± 4 days |
| Visit 9 (Phone: Study Day 57) | ± 4 days |
| Visit 10 (Clinic; Study Day 71) | ± 4 days |
| Visit 11 (Phone: Study Day 85) | ± 4 days |
| Visit 12 (Clinic: Study Day 99) | ± 4 days |
| Visit 13 (Clinic; Study Day 113; post dosing) | ± 4 days |
| Visit 14 (ECHO clinic; 3-6 months after last dose) | + 30 days |
| Blood collection for ZX008 PK | ± 15 minutes |

AED=antiepileptic drug (s); ECHO=echocardiogram; PK = pharmacokinetics

# 6.1.1 BASELINE PERIOD (STUDY DAY -28 TO STUDY DAY -1)

The Baseline Period of the study encompasses the screening activities that will occur on Study Day -28 as well as the observation period where subjects will be assessed for baseline seizure activity based on recordings of daily seizure activity entered into a diary.

# 6.1.1.1. Screening, Clinic Visit 1 (Study Day -28)

Screening is the predetermined series of procedures with which each investigator selects an appropriate and representative sample of subjects for enrollment into the study. Select screening data will be documented in the IWR and eCRF.

Written informed parental or guardian consent and assent of minors (if the subject is capable of providing assent) must be obtained before a subject can start any of the screening procedures. The procedure(s) for obtaining written informed consent and assent of minor (if the subject is capable of providing assent) are described in Section 11.2.

The Screening visit will occur on Study Day -28; however, the procedures may be split over 2 consecutive days (eg, Study Day -29 and Study Day -28 or Study Day -28 and Study Day -27). Splitting the visit procedures across 2 nonsequential days requires the approval of the medical monitor. The following procedures will be performed for all subjects before the start of seizure activity observation:


In cases where the screening period is extended beyond 28 days, the immediate 28 days before the Randomization visit will be used to calculate the baseline seizure frequency

- Obtain written informed consent for the study
- Obtain written informed consent from parent/caregiver to collect information about parent/caregiver symptoms and burden via the Zarit Caregiver Burden, and HADS rating
- Review inclusion and exclusion criteria
- Review retrospective seizure diary data
- Record demographic information
- Record medical, neurological, and epilepsy history
- Record current epilepsy status (number/type/duration seizures per month); submit form to Epilepsy Study Consortium
- Collect past 6 months (or available duration) of parent/caregiver seizure diary data if available (screen shots of cell phones are acceptable, as are photocopies of paper diaries or print outs) and place in source file
- Record prior medications
- Complete physical examination, including height and weight
- Complete neurological examination
- 12-lead electrocardiogram
- Doppler ECHO (this may be obtained any time between Study Day -28 and Study Day -15)
- Vital signs
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, and urinalysis)
- Urine or serum THC panel
- Whole blood CBD
- C-SSRS Baseline/Screening Assessment (Appendix 2)
- Instruct parent/caregiver on use of diary
- Dispense diary (after above procedures have been concluded; the 28-day period for determining baseline seizure frequency begins when screening assessments are completed and the seizure diary is dispensed)
- Record AEs
- Record AESIs

Only eligible subjects as specified by the inclusion and exclusion criteria who are independently confirmed to be eligible by the Epilepsy Study Consortium will be enrolled into the study.

After enrollment into the study, each subject will be issued a "Subject Card" containing information about the subject's participation in the study. The subject or parent/caregiver will be advised to retain this card on his person for the entire duration of the study so that the investigator or the sponsor can be contacted in case of emergency.


In certain circumstances the sponsor may allow subjects who did not meet all inclusion/exclusion criteria at the time of the Screening Visit to have the screening period extended, or to be rescreened for eligibility. In all cases the investigator should consult with the Medical Monitor. Decisions whether to permit rescreening resides solely with the sponsor.

The decision whether to permit extended screening or rescreening can be influenced by many factors individual to that subject case. Some general principles apply:

- 1. If baseline seizure screening is extended or the subject is discontinued and then rescreened the screening period for establishing the baseline seizure frequency will be the immediate 4 weeks before the randomization visit.
- 2. Subjects who are found to be on a prohibited medication at the screening visit may be weaned off of that medication provided:
  - a. Decisions to withdraw a disallowed concomitant medication must be made with the agreement of the prescribing physician
  - b. If the medication has antiepileptic properties, a wash out of at least 5 half-lives must be completed before collection of baseline seizure data.
  - c. If a decision has been made to wear off of a medication without antiepileptic properties and the washout period (at least 5 half-lives) is expected to be shorter than 3 weeks, then the subject may remain in screening and chart seizures using the seizure diary.
- 3. If screening is extended, laboratory and ECHO assessments must be at least 6 weeks current at the time of Randomization. Assessments older than 6 weeks will need to be repeated prior to Randomization. If laboratory assessments are repeated within 2 weeks of Randomization, samples do not need to be collected during Visit 3, provided valid results are obtained.

## **6.1.1.2.** Phone Visit 2 (Study Day -15)

Site personnel will contact the subject via telephone on Study Day -15 and record the following:

- AEs
- AESI

In addition, site personnel with review the diary entries with the parent/caregiver. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.

## 6.1.1.3. Clinic Visit 3 (Study Day -1): Randomization

This period is intended to ensure that subjects meet the study entry criteria and confirm they have experienced  $\geq 2$  seizures resulting in drops per week during the 4-week Baseline Period. Subjects must have at least 28 days of prospective diary data at Visit 3.

The following procedures will be performed on Study Day -1:

- Review inclusion and exclusion criteria
- Review current seizure activity (number/type/duration) from diary since previous


visit and calculate the number of seizures resulting in drops per week and over the 4-week observation period.

- Ensure approval for enrollment has granted by the Epilepsy Study Consortium and after ECHO review (ERT).
- Record prior medications since previous visit
- Complete physical examination, including weight
- Abbreviated neurological examination
- Vital signs
- 12-lead ECG
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, coagulation,, and urinalysis (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability))
- Collect plasma sample for AED pharmacokinetic evaluation (must document time of last dose)
- Urine or serum THC panel
- Whole blood CBD
- Obtain (optional) blood sample for epilepsy genotype panel (if not obtained at this visit, it should be obtained by Visit 12)
- Tanner Staging for subjects >7 to 18 years of age (Appendix 5)
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.
- C-SSRS Since Last Visit Assessment (Appendix 2)
- BRIEF (Appendix 3)
- QOLCE (Appendix 6)
- HADS (Appendix 7)
- Zarit Caregiver Burden Inventory (Appendix 8)
- Record AEs
- Record AESI
- When eligibility for the Titration Period is confirmed, obtain treatment assignment from the IWR
  - Dispense and administer study medication. Subjects will be required to stay in the clinic for monitoring of adverse reactions until the investigator determines it is safe to leave. Those considered by the investigator to need further monitoring will be hospitalized until the investigator determines they can be safely discharged. The first dose taken in the clinic will be recorded in the eCRF, but not the subject diary, and the next dose should be at least 8 hours later or the following morning. The dose on the following morning will count as Study Day 1 and be recorded in the subject diary.


#### 6.1.2 TITRATION AND MAINTENANCE PERIODS

### 6.1.2.1 **Titration Period Study Day 1**

Site personnel will contact the subject via telephone on Titration Period Study Days 4 and 8 and record the following:

• AEs
• AESI
• Concomitant medications

In addition, site personnel will review study medication dosing per with the parent/caregiver. Subjects will take their second dose of study medication on the morning of Study Day 1. Study

## Clinic Visit 6 (Titration Period Study Day 15) 6.1.2.3

Subjects will report to the clinic in the morning on Titration Period Study Day 15. The following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications
- Obtiain weight
- Obtain vital signs
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.
- C-SSRS Since Last Visit Assessment (Appendix 2)
- Clinical Global Impression Improvement (assessed by parent/caregiver)
- Clinical Global Impression Improvement (assessed by investigator)
- Record AEs
  - o Perform an abbreviated physical and/or neurological examination as appropriate based on last exam and reported AEs
  - Collect plasma sample for AED pharmacokinetic evaluation if clinically indicated (must document time of last dose)
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

## Phone Visit 7 (Maintenance Period Study Day 29)

Site personnel will contact the subject via telephone on Maintenance Period Study Day 29 and record the following:

- **AEs**
- AESI
- Concomitant medications


In addition, site personnel will review the diary entries with the parent/caregiver. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.

## 6.1.2.5 Clinic Visit 8 (Maintenance Period Study Day 43)

- Subjects will report to the clinic in the morning on Maintenance Period Study Day 43. Subjects should not take their morning dose(s) of study medication. The following procedures will be performed:
- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications
- Obtain weight (Note: if the subject's weight is ±25% of the weight at Study Day-1 the IMP dose will be recalculated)
- Obtain vital signs
- 12-lead electrocardiogram
- Doppler ECHO (this must be obtained any time between Study Day 40 and Study Day 54)
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin hormones, and urinalysis (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability))
- Urine or serum THC panel
- Whole blood CBD
- Collect plasma sample for ZX008 pharmacokinetic evaluation at the following timepoints: within 1 hour prior to the morning dose of study medication, and 1, 2 and 4-6 hours after the morning dose of study medication
- Collect plasma sample for AED pharmacokinetic evaluation (must document time of last dose)
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.
- C-SSRS Since Last Visit Assessment (Appendix 2)
- Zarit Caregiver Burden Inventory (Appendix 8)
- Clinical Global Impression Improvement (assessed by parent/caregiver)
- Clinical Global Impression Improvement (assessed by investigator)
- Perform an abbreviated physical and/or neurological examination as appropriate based on last exam and reported AEs
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

## 6.1.2.6 Phone Visit 9 (Maintenance Period Study Day 57)

Site personnel will contact the subject via telephone on Maintenance Period Study Day 57 and record the following:

- AEs
- AESI


Concomitant medications

In addition, site personnel with review the diary entries with the parent/caregiver. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.

## 6.1.2.7 Clinic Visit 10 (Maintenance Period Study Day 71)

Subjects will report to the clinic on Maintenance Period Study Day 71. The following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications
- Obtain weight
- Obtain vital signs
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.
- C-SSRS Since Last Visit Assessment (Appendix 2)
- Clinical Global Impression Improvement (assessed by parent/caregiver)
- Clinical Global Impression Improvement (assessed by investigator)
- Record AEs
- Perform an abbreviated physical and/or neurological examination as appropriate based on last exam and reported AEs
- Collect plasma sample for AED pharmacokinetic evaluation if clinically indicated
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

At Clinic Visit 10, compliant subjects who have tolerated IMP should be presented with the ICF for the open-label extension (Part 2). Informed consent for the open-label extension should be signed at Visit 12 or earlier in order to enter the open-label extension.

## 6.1.2.8 Phone Visit 11 (Maintenance Period Study Day 85)

Site personnel will contact the subject via telephone on Maintenance Period Study Day 85 and record the following:

- AEs
- AESI
- Concomitant Medications

In addition, site personnel with review the diary entries with the parent/caregiver. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.

# 6.1.2.9 Clinic Visit 12 (Maintenance Period Study Day 99): End of Study/Early Termination

The End-of-Study participation in Part 1 for an individual subject occurs after he/she has received IMP for 12 weeks in the Maintenance Period. At the Part 1 End-of-Study visit, the


subject may enroll into the Part 2 OLE Treatment Period if they have completed 12 weeks of treatment in the Maintenance Period. Other circumstances for participation in Part 2 are described in Section 4.3. Informed consent for the Part 2 OLE Treatment Period should be signed before data collection begins on Visit 12 (if not signed earlier) in order to participate in Part 2.

The End-of-Study visit may also occur if the subject withdraws participation from the study or the sponsor terminates the study. If the subject withdraws participation from the study, they may on a case-by-case basis, be eligible for entrance into the Part 2 OLE Treatment Period after consideration of the circumstances of the early termination and the potential benefit-risk of continued participation in a ZX008 trial. The decision whether to permit Part 2 participation resides solely with the sponsor, who may consult with the site investigator. If the sponsor terminates the study early, the subject may or may not be offered enrollment into Part 2, depending on the reason for termination.

Subjects will visit the clinic for the End-of-Study visit if one the following events occur:

- 1. The subject withdraws or is withdrawn from participation in the study.
- 2. The sponsor terminates the study.
- 3. The subject completes all study related visits and

procedures. The following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications
- Complete physical examination, including height and weight
- Complete neurological examination
- Obtain vital signs
- 12-lead electrocardiogram
- Doppler ECHO (must be performed any time between Study Day 90 and Study Day 113; if subject terminates early from the study, the ECHO should be scheduled as soon as practical). If the Study Day 43 ECHO was completed ≤30 days prior to early termination, the Visit 12 ECHO will not be performed provided the parent/guardian agrees to bring the subject to the clinic for the cardiac follow-up visit (see Table 9).
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability))
- Urine or serum THC panel
- Whole blood CBD
- Collect plasma sample for AED pharmacokinetic evaluation (must document time of last dose)
- Tanner Staging for subjects >7 to 18 years of age (Appendix 5)
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver
- C-SSRS Since Last Visit Assessment (Appendix 2)
- Clinical Global Impression Improvement (assessed by parent/caregiver)


- Clinical Global Impression Improvement (assessed by investigator)
- BRIEF (Appendix 3)
- QOLCE (Appendix 6)
- HADS (Appendix 7)
- Zarit Caregiver Burden Inventory (Appendix 8)
- Record AEs
- Record AESIs
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication for taper for subjects not continuing into Part 2.
- Dispense and administer study medication for transition for subjects continuing into Part 2. Subjects will be required to stay in the clinic for monitoring of adverse reactions until the investigator determines it is safe to leave. Those considered by the investigator to need further monitoring will be hospitalized until the investigator determines they can be safely discharged.

# 6.1.3 POST-DOSE VISIT (CLINIC VISIT 13; STUDY DAY 113)

For subjects entering the Part 2 OLE Treatment Period, the subject will visit the clinic on Day 113, which will also be Part 2 Day 1. The procedures described in Section 6.2 will be followed.

If the subject does not enter the Part 2 OLE Treatment Period (or discontinues from the study early), the subject will visit the clinic on Study Day 113 (or 14 days after the day of discontinuation). If necessary, Visit 13 may be conducted as a phone call, provided diaries and study medication are returned by this time. The following will be recorded/performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- AEs
- AESIs
- Concomitant medications
- Collect and review diary with parent/caregiver
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver

# 6.1.4 CARDIAC FOLLOW-UP VISIT (CLINIC VISIT 14; 3 and 6 months after last dose)

If the subject completes the study but does not enter the Part 2 OLE Treatment Period or discontinues from the study early, the subject will return to the clinic after study drug discontinuation for follow-up cardiac testing. The timing and frequency of exams are in Table 10. Subjects on blinded medication who are found to have been on placebo are not required to participate in follow-up testing once the blind is broken. As the ECHO and ECG will be administered in a separate clinic than the pediatric neurology clinic, an asymptomatic subject receiving a follow-up ECHO and ECG does not require a physical examination.

Subjects with positive findings on safety evaluations at post-dose follow-ups should have


repeat examinations every 3 months until the finding is resolved or stable and unlikely to change, with reports submitted as AEs to the ZX008 safety database.

Table 10: Schedule of Post-Treatment Cardiac Follow-up for Part 1

| | Duration of Blinded <sup>a</sup> or Fenfluramine Treatment | | | |
|---|---|---|---|---|
| D | Less than 2 weeks | 2 and | | Have had any cardiac sign or symptom regardless of the time on study drug <sup>b</sup> |
| Parameter | Cumulative | ≤13 weeks | >13 weeks | *** |
| ЕСНО | No | Yes, 3 months post- treatment | Yes,<br>3 and 6 months<br>post-treatment | Yes, 3 and 6 months post- treatment, and every 3 months until resolved, or stable and unlikely to change |
| ECG | No | Yes,<br>3 months post-<br>treatment | Yes,<br>3 and 6 months<br>post-treatment | Yes, 3 and 6 months post- treatment and every 3 months until resolved, or stable and unlikely to change |
| Physical examination | No | Yes,<br>3 months post-<br>treatment | Yes,<br>3 months post-<br>treatment only | Yes, 3 and 6 months post- treatment, and every 3 months until resolved, or stable and unlikely to change |

<sup>&</sup>lt;sup>a</sup> If blind is broken at the end of the study and a subject revealed to have taken only placebo, no further testing is required.

## 6.2 Part 2

Review of inclusion and exclusion criteria and written informed parental or guardian consent and assent of minors (if the subject is capable of providing assent) for Part 2 must be obtained before a subject can start any of the Part 2 Visit 15 procedures. This includes review and approval (or adjudication if required) of the ECG and/or ECHO findings by the central reader, and approval for continuation in the open-label extension (if applicable) by the IDSMC.

Only eligible subjects as specified by the inclusion and exclusion criteria who have successfully completed Part 1, or have permission from the Sponsor, will be enrolled into Part 2. Other circumstances for participation in Part 2 are described in Section 4.3.

Study procedures for the Part 2 OLE Treatment Period will be conducted according to the Schedule of Assessments in Table 2. Time windows for all assessments are detailed in Table 11.


Positive sign or symptom includes any development of valve thickening or regurgitation ("trace" or greater in mitral, aortic; mild or greater in pulmonary, tricuspid), or sign or symptom indicative of potential pulmonary hypertension as adjudicated by the ICAB.

**Table 11:** Time Windows for Assessments in Part 2

| Visit / Procedure | Time window (relative to scheduled visit / procedure) |
|---|---|
| Visit 15 (Clinic; OLE Study Day 1) | ± 4 days <sup>a</sup> |
| Visits 16 (Clinic/Phone; OLE Study Day 15) | ± 3 days |
| Visits 17-41 (Clinic: OLE Study Days 30, 60, 90, 180, 270, 360, 450, 540*, 630, 720*, 810, 900*, 990, 1080*, 1170,1260*, 1350, 1440*,1530, 1620*, 1710, 1800*, 1890, 1980*, 2070) | ± 4 days |
| Visit 42 (Clinic; OLE Study Day2160; EOS) | ± 4 days |
| Visit 43 (Clinic; OLE Study Day 2174; post dosing) | ± 4 days |
| Visit 44, 45 (ECHO clinic; 3 and 6 months after last dose) | + 30 days |

AED=antiepileptic drug (s); ECHO=echocardiogram

# 6.2.1 Clinic Visit 15 (OLE Study Day 1)

Part 2 Visit 15 will occur 14 days ( $\pm$  4 days) after Part 1 Visit 12. The 14-day transition period preceding Visit 15 may be extended up to 14 days in the case of a required safety adjudication of a Visit 12 ECHO alert.

The following procedures will be performed during Visit 15:

- Ensure entry criteria for Part 2 are met
- Vital signs
- Record prior and concomitant medications (use core study Visit 12 information)
- Instruct parent/caregiver on use of diary
- Record ongoing AEs as medical history
- Record ongoing AESI as medical history
- Collect, review, and dispense diary (after above procedures have been concluded)
- Dispense study medication

Data collected from Part 1 Visit 12 may be used for the following procedures unless otherwise indicated:

- Record medical, neurological, and epilepsy history
- Complete physical examination, including height and weight (use data collected at Part 1 Visit 12, unless there was a significant change in subject status warranting a new complete examination)
- Complete neurological examination (use data collected at Part 1 Visit 12, unless there was a significant change in subject status warranting a new complete examination)


<sup>&</sup>lt;sup>a</sup> In the case of a required safety review of a Visit 12 ECHO alert, the transition period between Visit 12 and Vist 15 may be extended up to 14 days to allow time for adjudication.

<sup>\*</sup>If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study. Up to 5 annual extensions can be applied, for a total treatment time of 72 months in the OLE. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk. The decision to extend and informed consent should be completed before the start of the first visit of the extension (e.g. Month 12, 24, 36, 48 or 60). After approval from Investigator and Sponsor for extension and starting after Visit 26/ Month24 (or at a later visit if Visit 26/ Month 24 visit has already occurred at the time of Protocol Amendment 4.0 approval), subject will return to the clinic every 6 months for the 1 year extension (i.e. Month 30, 36). The End of Study will be Visit 42, unless another extension is granted, in which case the subject will continue to return for clinic visits every 6 months and will have a phone visit 3 months after the in-clinic visit. Further extensions can then be applied as required if marketing approval is not yet received.

- 12-lead ECG
- Doppler ECHO
- marketing authorization ariations thereof. Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (use Part 1 Visit 12 information, unless investigator determines new laboratory evaluation is warranted due to change in subject status) (if collecting urine for urinalysis, urine may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
- Pregnancy test
- Urine or serum THC panel
- Whole blood CBD
- C-SSRS Since Last Visit Assessment (Appendix 2)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- BRIEF (Appendix 3)
- QOLCE (Appendix 6)
- HADS (Appendix 7)
- Zarit Caregiver Burden Inventory (Appendix 8)

## Clinic/Phone Visit 16 (OLE Study Day 15) 6.2.2

Part 2 Visit 16 may be performed in the clinic, or, at the discretion of the investigator, performed via phone.

If Visit 16 is performed in the clinic, subjects will report to the clinic in the morning of that day. The following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications since previous visit
- Obtain weight
- Vital signs
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (only if investigator determines new laboratory evaluation is warranted due to change in subject status since Visit 15) (if collecting urine for urinalysis, urine may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.
- Record AEs
  - Perform an abbreviated physical and/or neurological examination as appropriate based on last exam and reported AEs
  - Collect plasma sample for AED pharmacokinetic evaluation if clinically indicated (must document time of last dose)
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver


• Collect and review study medication

If the visit is performed as a phone visit, site personnel will contact the subject on Study Day 15 and record/review the following:

- Concomitant medications
- AEs
- AESI
- Study medication use
- Diary entries

# 6.2.3 Clinic Visits 17-21 (OLE Months, 1, 2, 3, 6, and 9)

Subjects will report to the clinic for Part 2 Clinic Visits 17 through 21. The following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications
- Obtain weight (Note: if the subject's weight is ±25% of the weight at Part 2 Day 15, the IMP dose will be recalculated)
- Obtain vital signs
- 12-lead ECG
- Doppler ECHO (at Months 1, 3, 6, and 9)
- Urine or serum pregnancy test for females of child-bearing potential (at Months 3, 6, and 9)
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis; at Months 3, 6 and 9 unless otherwise clinically indicated) (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
- Urine or serum THC panel (at Months 3, 6 and 9)
- Whole blood CBD (at Months 3, 6, and 9)
- Collect plasma sample for AED PK and document time of last dose (at Months 3, 6, and 9 unless otherwise clinically indicated)
- Tanner Staging for subjects > 7 to 18 years of age (Month 6 only) (Appendix 5)
- Collect, review, and dispense diary. Ensure diary is being completed daily; if diary compliance is low (i.e. <90%), re-train parent/caregiver.
- C-SSRS Since Last Visit Assessment (Appendix 2)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- BRIEF (Month 6 only) (Appendix 3)
- QOLCE (Month 6 only) (Appendix 6)
- HADS (Month 6 only) (Appendix 7)
- Record AEs
  - Perform an abbreviated physical and/or neurological examination as appropriate based on last exam and reported AEs


- Collect plasma sample for AED pharmacokinetic evaluation if clinically indicated
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

The next study visit should be Visit 30 (EOS), unless a 1-year extension is granted. If extending study participation, the decision should be made during Visit 21 (or at least prior to conducting Visit 22 procedures) by the Investigator and the consent from the subject or parent/caregiver obtained. After approval from Investigator and Sponsor for extension, Subject will return every 3 months for the 1 year extension (i.e. Month 12, 15, 18, 21). The End of Study will be Visit 30, on the 24<sup>th</sup> month of OLE, unless another 1 year extension is granted, in which case the subject will continue to return for clinic visits every 3 months (i.e. Month 24, 27, 30, 33) until the EOS Visit 30 on the 36<sup>th</sup> month of OLE.

# 6.2.4 Clinic Visit 22 (OLE Month 12)

Subjects will report to the clinic and the following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications
- Obtain weight (Note: if the subject's weight is ±25% of the weight at Part 2 Day 15, the IMP dose will be recalculated)
- Complete physical examination, including height and weight, and calculation of BMI
- Complete neurological examination
- Obtain vital signs
- 12-lead ECG
- Doppler ECHO (must be performed any time between Study Day 344 and Study Day 365).
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry and hematology, and urinalysis)
- Urine or serum THC panel
- Whole blood CBD
- Collect plasma sample for AED PK evaluation (must document time of last dose)
- Tanner Staging for subjects > 7 to 18 years of age (Appendix 5)
- Collect and review diary
- C-SSRS Since Last Visit Assessment (Appendix 2)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- BRIEF (Appendix 3)
- QOLCE (Appendix 6)
- HADS (<u>Appendix 7</u>)
- Zarit Caregiver Burden Inventory (Appendix 8)


- Record AEs
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

# Clinic Visits 23-41 (OLE Months 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69) approval is not vot a 6.2.5

If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk.

From Visit 26/Month 24 (or a later visit if Visit 26/Month 24 has already occurred at the time of Protocol Amendment 4.0 approval), if approved for the extensions, subjects will report to the clinic every 6 months and will have a phone visit 3 months after each in-clinic visit for Part 2 Clinic Visits 26 through 41.

The following procedures will be performed during in-clinic vi

- Record concomitant medications
- Obtain weight (Note: if the subject's weight is ±25% of the weight at Part 2 Day 15, the IMP dose will be recalculated)
- Obtain vital signs
- Abbreviated physical examination, as appropriate based on last exam and reported AEs
- Abbreviated neurological examination, as appropriate based on last exam and reported
- 12-lead ECG, if clinically indicated
- Doppler ECHO
- Urine or serum pregnancy test for females of child-bearing potential
- Only if clinically indicated:
  - Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
  - Collect plasma sample for AED PK and document time of last dose
- Seizure Assessment by Investigator
- C-SSRS Since Last Visit Assessment (Appendix 2)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- Record AEs
- Record AESI


- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

The following procedures will be performed <u>during phone visits</u>:

- Record concomitant medications
- Record AEs
- Record AESI

alithoritation vi The next study visit after Visit 25/Month 21, Visit 29/Month 33, Visit 33/Month 45, Visit 37/Month 57 or Visit 41/Month 69 should be Visit 42 (EOS), unless another 1-year extension is granted. If extending study participation, the decision should be made during the in-clinic visit preceeding the annual reconduction by the Investigator and the consent from the subject or parent/caregiver obtained. After approval from Investigator and Sponsor for extension and starting after Visit26/Month 24 (or a later visit if Visit 26/Month 24 has already occurred at the time of Protocol Amendment 4.0 approval), subject will return to the clinic every 6 months and will have a phone visit 3 months after each in-clinic visit for the 1 year extension. The End of Study will be Visit 42, the 72<sup>nd</sup> month of the OLE, or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever occurs first.

## Clinic Visit 42: End of Study/Early Termination 6.2.6

The End-of-Study participation in Part 2 for an individual subject occurs after he/she has received IMP for up to 5 years in the Part 2 OLE Treatment Period, or until ZX008 is approved in a subject's country of residence and listed on a patient's health plan formulary, whichever occurs first. The End-of-Study visit may also occur if the subject withdraws participation from in Part 2 or the Sponsor terminates the study.

Subjects will visit the clinic for the End-of-Study visit if one the following events occur:

- 1. The subject withdraws or is withdrawn from participation in the study.
- 2. The Sponsor terminates the study.
- The subject completes all study related visits and procedures (at least up to Month 12, but extensions may be granted for up to 72 months).
- 4. ZX008 is approved in a subject's country of residence and is listed on a patient's health plan formulary

The following procedures will be performed for subjects who did not extend Part 2 participation past 12 months:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record concomitant medications


- Complete physical examination, including height and weight, and calculation of BMI
- Complete neurological examination
- Obtain vital signs
- 12-lead ECG
- Doppler ECHO (must be performed within 3 weeks of the visit; if subject terminates early from the study, the ECHO should be scheduled as soon as practical). If the previous ECHO was completed ≤ 30 days prior to early termination, the Visit 30 ECHO will not be performed provided the parent/guardian agrees to bring the subject to the clinic for the cardiac follow-up visit (see Table 12).
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
- Urine or serum THC panel
- Whole blood CBD
- Collect plasma sample for AED PK evaluation (must document time of last dose)
- Tanner Staging for subjects > 7 to 18 years of age (Appendix 5)
- Collect and review diary C-SSRS Since Last Visit Assessment (Appendix 2)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- BRIEF (Appendix 3)
- QOLCE (Appendix 6)
- HADS (<u>Appendix 7</u>)
- Zarit Caregiver Burden Inventory (Appendix 8)
- Record AEs
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication (not applicable for subjects transitioning to commercial drug)

The following procedures will be performed for subjects who are extended Part 2 participation past 12 months:

- Record concomitant medications
- Complete physical examination, including height and weight, and calculation of BMI
- Complete neurological examination
- Obtain vital signs
- Doppler ECHO (must be performed within 3 weeks of the visit; if subject terminates early from the study, the ECHO should be scheduled as soon as practical). If the previous ECHO was completed ≤ 30 days prior to early termination, the Visit 30 ECHO will not be performed provided the parent/guardian agrees to bring the subject to the clinic for the cardiac follow-up visit (see Table 12).
- Urine or serum pregnancy test for females of child-bearing potential
- Only if clinically indicated:


- Collect plasma sample for AED PK evaluation (must document time of last dose)
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
- o 12-lead ECG
- Collect and review diary C-SSRS Since Last Visit Assessment (<u>Appendix 2</u>)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- Seizure assessment by investigator
- Record AEs
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication (not applicable for subjects transitioning to commercial drug)

# 6.2.7 POST-DOSE VISIT (CLINIC Visit 43; 14 DAYS AFTER LAST DOSE OF IMP)

If the subject completes the study (or discontinues from the study early), and is not switching to commercially available drug, the subject will visit the clinic for Visit 43 (14 days after the EOS or day of discontinuation). Visit 43 may be conducted as a phone call if physical and neurological examinations are not clinically indicated, provided diaries (if applicable) and study medication are returned by this time. The following procedures will be performed:

- Review current seizure activity (number/type/duration) from diary since previous visit
- Record AEs
- Perform an abbreviated physical and/or neurological examination as appropriate based on last exam and reported AEs
- Obtain weight
- Record AESI
- Record concomitant medications
- Collect and review diary with parent/caregiver
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver

# 6.2.8 CARDIAC FOLLOW-UP VISIT (CLINIC VISIT 44, 45; 3 AND 6 MONTHS AFTER LAST DOSE OF IMP)

If the subject completes Part 2 or discontinues from the Part 2 early, and is not switching to commercially available drug, the subject will return to the clinic for follow-up cardiac testing. The timing and frequency of exams are in Table 12. As the ECHO and ECG will be administered


in a separate clinic than the pediatric neurology clinic, an asymptomatic subject receiving a second follow-up ECHO and ECG does not require a physical examination.

Subjects with positive findings on safety follow-up examinations should continue to be followed until the finding is resolved or stable and unlikely to change.

If the subject completes the study (or discontinues from the study early) and is switching to commercially available drug, the subject will complete the EOS visit and follow the drug administration process outlined for commercial product as advised by the subject's physician. The EOS/ET and cardiac follow-up visits are not required.

Table 12. Schedule of Post-Treatment Cardiac Follow-up for Part 2

| | Duration of Fenfluramine Treatment | | | |
|---|---|---|---|---|
| | | | | Have had any cardiac sign or symptom |
| | Less than | | | regardless of the time on study drug <sup>a</sup> |
| Parameter | 2 weeks<br>Cumulative | 2 and<br>≤ 13 weeks | > 13 weeks | disi b |
| ЕСНО | No | Yes, | Yes, | Yes, |
| | | 3 months post- | 3 and 6 months | 3 and 6 months post-treatment, and until |
| | | treatment | post-treatment | resolved, or stable and unlikely to change |
| ECG | No | Yes, | Yes, | Yes, |
| | | 3 months post- | 3 and 6 months | 3 and 6 months post-treatment and until |
| | | treatment | post-treatment | resolved, or stable and unlikely to change |
| Physical | No | Yes, | Yes, | Yes, |
| examination | | 3 months post- | 3 months post- | 3 and 6 months post-treatment, and until |
| | | treatment | treatment only | resolved, or stable and unlikely to change |

<sup>&</sup>lt;sup>a</sup> Positive sign or symptom includes any development of valve thickening or regurgitation ("trace" or greater in mitral, aortic; mild or greater in pulmonary, tricuspid), or sign or symptom indicative of potential pulmonary hypertension as adjudicated by the ICAB.

# 6.3 STUDY CONDUCT DURING COVID-19

In March 2020, the World Health Organization declared a global pandemic related to an illness caused by a novel coronavirus known as COVID-19. Alternative procedures and allowances are permitted due to restrictions related to COVID-19, including delays to in-person visits and specific assessments, performing remote phone or video visits if in-person visits cannot be conducted, and arranging shipments of investigational product directly to subjects. These allowances are detailed in Appendix 10. Though every attempt should be made to conduct study visits as described in this protocol, any implementation of alternative processes should be properly documented, including what was done differently, and which assessments or visits were missed or performed via phone or video.

## 6.4 ESTIMATED BLOOD VOLUME COLLECTION

The maximum total blood volume collected during Part 1 of the study for clinical laboratory testing, genotyping, and PK will be approximately 84.0 mL, as outlined in Table 13 The


maximum total blood volume collected during Part 2 of the study for clinical laboratory testing and PK will be variable as the clinical laboratory testing will be performed as clinically indicated for the majority of in clinic visits after Visit26/Month 24, and will be approximately 104.0 mL at the minimum and will equal up to 351.5 mL , as outlined in Table 14.

**Table 13:** Maximum Estimated Blood Volume Collection for Part 1\*

| PART 1 | Visit 1 (Day -28) | Visit 3<br>(Day -1) | Visit 8<br>(Day 43) | Visit 12<br>(Day 99) | TOTAL |
|---|---|---|---|---|---|
| Coagulation | | 3.0 mL | | | 3.0 mL |
| Chemistry | 5.0 mL | 5.0 mL | 5.0 mL | 5.0 mL | 20.0 mL |
| Pregnancy test (serum) | included in<br>Chemistry | included in<br>Chemistry | included in<br>Chemistry | included in<br>Chemistry | 0.0 mL |
| Hormones | | 5.0 mL | 5.0 mL | 5.0 mL | 15.0 mL |
| Immunoglobulin | 2.5 mL | 2.5 mL | 2.5 mL | 2.5 mL | 10.0 mL |
| Hematology | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | 8.0 mL |
| Genotype Panel | | 4.0 mL | | ' .;(0) | 4.0 mL |
| AED PK plasma sample* | | 2.0 mL | 2.0 mL | 2.0 mL | 6.0 mL |
| ZX008 PK plasma sample | | | 8.0 mL | | 8.0 mL |
| Volume for flushing indwelling catheter | | | 2.0 | | 2.0 mL |
| Cannabidiol/THC | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | 8.0 mL |
| TOTAL | 11.5 mL | 25.5 mL | 28.5 mL | 18.5 mL | 84.0 mL |

AED=Anti-epileptic drugs; PK=pharmacokinetics

Table 14. Maximum Estimated Blood Volume Collection for Part 2\*

| PART 2 | Visit 19<br>(Day 90) | Visit 20 (Day<br>180) | Visit 21 (Day 270) | Visit 22 (Day 360) | Visits 23-<br>42 (in<br>clinic<br>only) | TOTAL |
|---|---|---|---|---|---|---|
| Chemistry | 5.0 mL | 5.0 mL | 5.0 mL | 5.0 mL | | 20.0 mL |
| Pregnancy test (serum) | included in<br>Chemistry | included in<br>Chemistry | included in<br>Chemistry | included in<br>Chemistry | 2.5 mL | 2.5 mL |
| Hormones | 5.0 mL | 5.0 mL | 5.0 mL | 5.0 mL | | 20.0 mL |
| Immunoglobulin | 2.5 mL | 2.5 mL | 2.5 mL | 2.5 mL | | 10.0 mL |
| Hematology | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | | 8.0 mL |
| AED PK plasma sample | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | | 8.0 mL |
| Cannabidiol/THC | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | | 8.0 mL |
| TOTAL | 18.5 mL | 18.5 mL | 18.5 mL | 18.5 mL | 30 mL | 104.0 mL |

AED=Anti-epileptic drugs; PK=pharmacokinetics


<sup>\*</sup>Blood collection for AED pharmacokinetic evaluation may be collected on Visits 6 and 10 if clinically indicated. If collected during these visits, the total blood volume per subject would equal up to 88.0 mL.

<sup>\*</sup>Laboratory testing may be conducted on Visits 16-18 and 23-42 if clinically indicated. After Visit 26, in-clinic visits will occur every 6 months. If collected during these visits, the total blood volume per subject would equal up to 351.5mL.

<sup>\*</sup>In concordance with The Seattle Children's Research Foundation Guidance (Appendix 9),

blood collection volumes for children weighing up to 15 kg will be:

- The maximum allowable volume of blood in one draw is 22-30 mL (2.5% of total blood volume)
- The maximum in a 30-day period is 44-60 mL.

On Part 1 Day 43/Visit 8 the pharmacokinetic blood draw will be completed as the priority and the blood draw for chemistry and hematology will be skipped for those subjects who weigh less than 13.5 kg, unless medical concerns (for example, from previous tests or reported side effects) prioritize chemistry and/or hematology.

If blood collection is restricted due to volume or due to inability to draw adequate volume, collection should be prioritized as shown in Table 15

**Table 15: Priorities for Blood Sample Collections** 

| Table 13. | THOTHES IOI DIOUG Sain | |
|---|---|---|
| | Assessment | Priority |
| ZX008 PK sa | | Priority 1 |
| Clinical chem | nistry | Priority 2 |
| Cannabidiol | | Priority 2 |
| AED plasma | sample | Priority 2 |
| LH, FSH, est | radiol, testosterone, GH, | Priority 3 |
| prolactin | | |
| Hematology | | Priority 3 |
| IGF-1 | | Priority 4 |
| Genotyping | | One time optional collection any time during or after Visit 3 |
| 71 0 | | (Randomization) in Part 1 |
| Coagulation | 05 | One time collection any time before Part 1 PK day |
| (his docum | ant cannot be used and an | Nextens, |


## 7. EFFICACY, SAFETY, AND PHARMACOKINETIC **ASSESSMENTS**

Variables used to measure treatment compliance with respect to administration of the IMP are described in Section 5.7.

7.1 EFFICACY/EFFECTIVENESS ASSESSMENTS

Baseline is defined.

Baseline is defined as the frequency of motor seizures resulting in drops during the 4 Baseline Period prior to administration of IMP.

Retrospective diary data (up to 6 months) will be collected, if available, for an exploratory evaluation of the duration of baseline data capture on interpretation of po treatment effect.

For all questionnaires and rating scales, the same evaluator (at the clinical site and parent/caregiver) should complete the assessments for the duration of the study. Substitutions at the clinic with another rater that has established inter-rater reliability is acceptable on an infrequent basis. For the in-clinic questionnaires and rating scales completed by the parent/caregiver, if the same parent/caregiver cannot complete the questionnaire/rating scale at a visit, the questionnaire/rating scale will not be completed. For the diary, the same parent/caregiver will complete all entries throughout the study.

## 7.1.1 **Seizure Assessments**

Seizure frequency by type and duration will be recorded daily by the parent/caregiver in a diary during Part 1 and up to 12 months in Part 2 (i.e., up to Visit 22). Seizure types include:

- Hemiclonic (note lateralization right body, left body, or independent right A: and left)
- Focal With or Without Retained Awareness B:
- C: Secondarily Generalized Tonic Clonic (evolving to bilateral convulsive seizure from focal seizure)
- Generalized Tonic Clonic

Convulsion E: Absence or Atypical

Absence

- Myoclonic
- G: Tonic
- Atonic
- Clonic
- J: Tonic/Atonic (cannot differentiate)
- K: Infantile Spasms (if under 3 years of age)
- L: Epileptic Spasms (if 3 years of age and older)
- 0:


<sup>\* &</sup>quot;Other" indicates a seizure type that cannot be classified in any of the above seizure

types A-L. All other seizures must be classified appropriately based on the Investigator's medical opinion and Epilepsy Study Consortium approval.

Parents/caregivers will also indicate in the diary entry whether the seizure resulted in a drop, or would have resulted in a drop were it not for the position (ie, in a chair). This includes seizures involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the subject's head hitting a surface or that could have led to a fall or injury, depending on the patient's position at the time of the seizure.

Efficacy/effectiveness endpoints that will be derived from the diary data include frequency of seizures that result in drops and seizures that do not result in drops, motor seizures, and all seizures, and the number/duration of seizure-free intervals.

Seizures that evolve into status epilepticus (SE) will be captured by type and duration (>10 minutes) as are all seizures. SE should be entered as an SAE if a prolonged seizure or series of seizures persists for 30 minutes or longer, regardless of administration of rescue medication, and is either diagnosed by a medical professional or occurs more than once in a day. SE lasting for less than 30 minutes should be entered as an AE, unless one of the other SAE criteria (eg, hospitalization) are met. If this incident involves multiple seizures close in time, the SE definition applies if the seizures are close together such that consciousness is not regained between ictal events.

After 12 months in Part 2, seizure diaries are not required. Rather, based on discussions with the parent/caregiver, clinical evaluation, and review of any documentation provided by the caregivers, investigators will assess the percent improvement in seizure burden on a 5-point scale:  $\langle 25\%, \geq 25\%, \geq 50\%, \geq 75\%, 100\%$  [ie, seizure-fee] improvement.

## 7.1.2 Clinical Global Impression - Improvement

Both the parent/caregiver and the investigator will rate their global impression of the subject's condition throughout the study according to the schedule in Table 1 and Table 2.

The CGI scale measures the change in the subject's clinical status from a specific point in time, ie, the Baseline Period. The CGI rating scale permits a global evaluation of the subject's improvement over time. The severity of a patient's condition is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows:

1=very much improved

2=much improved

3=minimally improved

4= no change

5=minimally worse

6=much worse

7=very much worse

The parent/caregiver will be asked to indicate the appropriate response that adequately describes how their child's symptoms have improved or worsened relative to baseline before the beginning of the study (before any study drug was taken).

The investigator (or appropriately trained designee) will be asked to indicate the appropriate response that adequately describes how the subject's symptoms have improved or worsened


relative to baseline before the beginning of the study (before any study drug was taken). A paragraph describing symptoms and function at baseline will be document in the source file prior to rating.

## 7.1.3 Vineland Adaptive Behavior Scale (VABS)

The VABS (Appendix 4) is a parent/caregiver completed assessment that looks at the personal and social skills of individuals from birth through adulthood. Because adaptive behavior refers to an individual's typical performance of the day-to-day activities required for personal and social sufficiency, these scales assess what a person actually does, rather than what he or she is able to do. The VABS assesses adaptive behavior in 4 domains: communication, daily living skills, socialization, motor skills, and will be conducted according to the schedule in Table 1.

## **7.1.4 QOLCE**

The QOLCE (Appendix 6) is a parent/caregiver completed assessment that looks at how epilepsy affects day-to-day functioning of their child in various life areas, including physical activities, well-being, cognition, social activities, behavior and general health, will be conducted according to the schedule in Table 1 and Table 2. The QOLCE has been validated in children aged 4 and older, and there are published data on the use of the QOLCE in children with epilepsy as young as 2 years of age (Sabaz et al., 2000; Talarska 2007).

# 7.1.5 Parent/Caregiver Affective Symptoms

7.1.5.1 The impact on anxiety and depressive symptoms of the parent/caregiver responsible for a patient with LGS will be assessed according to the schedule in Table 1 and Table 2 using 2 scales: the HADS and the Zarit Caregiver Burden Inventory. Parents/caregivers who do not give consent to collect this rating scale will not complete them. The same parent/caregiver should complete this rating throughout the study. If that person is not available at the visit, the scale should not be completed. Hospital Anxiety and Depression Scale (HADS)

The HADS (<u>Appendix 7</u>) is a tool commonly used to determine the levels of anxiety and depression that a person is experiencing. It is a 14-item scale that generates ordinal data. Seven of the items relate to anxiety and 7 relate to depression.

The HADS (Appendix 7) is a tool commonly used to determine the levels of anxiety and depression that a person is experiencing. It is a 14-item scale that generates ordinal data. Seven of the items relate to anxiety and 7 relate to depression.

## 7.1.5.2 Zarit Caregiver Burden Inventory

The impact on caregiver burden will be assessed according to the schedule in Table 1 and Table 2 using the Zarit Caregiver Burden Inventory. Parents/caregivers who do not give consent to collect this rating scale will not complete them. The same parent/caregiver should complete this rating throughout the study. If that person is not available at the visit, the scale should not be completed.

The Zarit Caregiver Burden Inventory (Appendix 8) is a 22-item inventory derived from the original 29-item Zarit inventory. It is the most widely used standardized, validated scale to


assess caregiver burden, administered previously in various neurological disorders, including epilepsy (Kim, 2010; Westphal-Guitti, 2007). The 22 items evaluate the effect of disease on the caregiver's QOL, psychological suffering, financial difficulty, shame, guilt, and difficulty in Demographics, Medical/Neurological/Epilepsy History, and Pre-Study Medication

Ographics (sex, age, height, weight, and BMI), all one ry from the past 5 years (including bject's current and blooming bject's current and social and family relationships. Scores range from 0 to 88 with higher scores indicating higher burden (<20: little or no burden, 21–40: mild-to-moderate burden, 41–60: moderate-to severe burden, 61–88: severe burden).

## 7.2

# 7.2.1

Subject demographics (sex, age, height, weight, and BMI), all ongoing conditions and relevant medical history from the past 5 years (including all major hospitalizations and surgeries) as well as the subject's current medical status will be recorded at the Screening visit. Significant medications taken during the 30 days prior to the Screening visit will be documented.

Medication history will be updated as outlined in Table 1 and Table 2

#### 7.2.2 **Adverse Events**

Adverse events (AEs) will be collected from the time of signing the informed consent form/assent form until the end of the study, including the follow-up clinic visit. Details of the definitions and categorization of AEs, and procedures for the reporting of AEs, are available in Section 9.

Severity and causality of AEs will be evaluated according to the criteria specified in Section 8.2 and Section 8.3, respectively. The observation period for AE reporting is specified in Section 8.4. At the beginning of each visit at the study site, the study personnel will specifically inquire about any AEs that might have occurred since the last study site visit. As described below, an abbreviated physical and/or neurological examination for each subject will be conducted based on reported AEs.All AEs will be recorded on the appropriate eCRF page.

## **Physical Examinations** 7.2.3

Complete and abbreviated physical examinations, including height and weight, will be conducted by the investigator or designee during the study as outlined in Table 1 and Table 2. A complete standard of care physical examination for each subject will be performed and will cover the following body systems: general appearance, skin, eyes, ears, nose, throat, heart, lungs, abdomen, neurological system, lymph nodes, spine, and extremities. An abbreviated physical examination for each subject will cover the following body systems: heart, lungs, and follow up of other systems as appropriate based on last exam and reported AEs.

Any unfavorable findings not present at screening, or worsened from the baseline assessment and considered by the investigator as clinically significant, occurring at any point in the study will be documented in the eCRF as an AE.

### 7.2.4 **Neurological Examinations**

Complete and abbreviated neurological examination will be conducted by the investigator or designee during the study as outlined in Table 1 and Table 2. A complete standard of care


neurological examination for each subject will be performed and will cover the following: cranial nerves, muscle strength and tone, reflexes, coordination, sensory function, and gait. An abbreviated neurological follow-up examination for each subject will evaluate any

7.2.5 Vital Signs (Including Height and Weight)

Height, weight, and vital signs (blood pressure, heart rate, temperature, and respiratory rate) will be documented for subjects during study as outlined in Table 1 and Table 2.

7.2.6 Laboratory Measurements

Laboratory safety parameters will be analyzed using standard validated methors. Table 2 and Table 10:

• Hematology.

- leukocytes, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets
- Blood Biochemistry: albumin (ALB), alkaline phosphatase (ALP), alanine aminotransferase (ALT; SGPT), aspartate aminotransferase (AST; SGOT), bicarbonate, blood urea nitrogen (BUN), calcium (Ca), carbon dioxide (CO2), chloride (Cl), creatinine, creatine kinase, gamma-glutamyl transferase (GGT), glucose, lactate dehydrogenase (LDH), phosphorus, potassium (K), sodium (Na), total bilirubin, direct bilirubin, total cholesterol, total protein, triglycerides, uric acid, eGFR.
- Tests of growth and precocious puberty: Growth hormone (GH), insulin-like growth factor-1 (IGF-1), prolactin, Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH), testosterone, estradiol, thyroid function (T3, T4, and thyroid stimulating hormone [TSH]),
- Immunoglobulin (IgG, IgA, IgM)
- Epilepsy genotype panel
- Coagulation: Prothrombin time (PT)/International normalized ratio (INR), activated partial thromboplastin time (PTT)
- Whole blood cannabidiol
- Urinalysis: analysis for pH, glucose, ketones, nitrite, protein, bilirubin, urobilinogen, leukocyte esterase, and occult blood. Microscopic analysis will be performed for blood, all cell types, and casts.
- Urine or serum pregnancy test: Urine or serum pregnancy testing will be performed in


female subjects of childbearing potential.

- Urine or serum THC panel
- The investigator will receive the laboratory report from the central laboratory. After reviewing the report and evaluating any results that are outside the normal range for clinical significance, the investigator must sign and date the laboratory report in a timely fashion.

Tests resulting in abnormal laboratory values that have been classified by the investigator as abnormal, clinically significant should be repeated as soon as possible after receiving the laboratory report to rule out laboratory errors.

At Screening, any laboratory values that deviate from the reference ranges that are not exclusionary and are considered by the investigator as clinically relevant must be documented on the medical history form of the eCRF. Any deviation outside of the reference range considered by the investigator as clinically significant (ie, classified as an abnormal, clinically significant value) at any visit after screening will be documented in the eCRF as an AE (see Section 9).

## 7.2.7 Plasma Sample for Concomitant Antiepileptic Drug(s)

Plasma samples to ensure that concomitant AEDs dosing is within an acceptable range will be conducted during the study as outlined in Table 1 and Table 2. All samples will be analyzed at study end and do not constitute safety assessments. (Importantly, plasma samples for concomitant AEDs can be performed at any time if considered clinically indicated. In these instances results will be provided to the unblinded Medical Monitor and discussed with the Principal Investigator.)

## 7.2.8 Electrocardiograms

Twelve-lead ECGs will be conducted during study as outlined in Table 1 and Table 2 after the subject has been in the supine position resting for ≥5 minutes. Heart rate, PR duration, QRS duration, QT duration, QTcF (Fridericia's correction formula), and the investigator's overall interpretation will be recorded.

# 7.2.9 Doppler Echocardiography

Doppler echocardiography will be conducted at a facility with experience for the subject's age during study as outlined in Table 1 and Table 2. Doppler echocardiography uses ultrasound technology to examine the heart or blood vessels. An ECHO uses high frequency sound waves to create an image of the heart while the use of Doppler technology allows determination of the speed and direction of blood flow by utilizing the Doppler effect. Predetermined standard guidelines on the proper evaluation of certain measurements, as well as abnormality thresholds, were constructed by the sponsor's ICAB prior to study initiation. These thresholds are provided in Table 9 and Table 11. A manual of proper ECHO technique for sites is provided in a separate document.

## 7.2.10 Behavior Rating Inventory of Executive Function (BRIEF)

The Behavior Rating Inventory of Executive Function (BRIEF) is a parent or teacher report


measure designed to address the multidimensional nature of the executive function construct and will be used to assess the effects of ZX008 on cognition. The BRIEF assesses eight theoretically and statistically derived subdomains of executive function. It was designed to be used for a wide range of childhood disorders in order to augment traditional clinic-based assessments, and to provide an increased level of ecological validity for clinical assessments (Rabbit, 1997). Age-appropriate versions of the BRIEF (BRIEF-P: 2 to 5 year olds; BRIEF: 6 to 18 year olds; BRIEF-A: 19 to 35 year olds), will be conducted according to the schedule in Table 1.

## 7.2.11 Tanner Staging

Tanner Staging (Appendix 5) will be assessed for subjects >7 to 18 years old during the study as outlined in Table 1 and Table 2. Conceptually, pubertal maturation can be described in terms of sequence, timing, and tempo. Puberty consists of a series of predictable events, and the sequence of changes in secondary sexual characteristics has been categorized by several groups. The staging system used most frequently was published by Marshall and Tanner (1969, 1970) and the sequence of changes are commonly referred to as 'Tanner stages'.

## 7.2.12 Columbia-Suicide Severity Rating Scale

C-SSRS (Appendix 2) will be assessed during study as outlined in Table 1 and Table 2. The C-SSRS is a validated rating scale that assesses suicidal behavior and ideation. The scale is used to assess and track suicide events and provides a summary measure of suicidal tendency. Age and intellectual development appropriate versions of the C-SSRS (Baseline/Screening and Since Last Visit) will be used in this study.

Subjects who are younger than 7 years chronologically, or who are judged by the investigator not to have the mental capacity to understand the questions as specified on the C-SSRS, will not complete the rating. The investigator should use his/her judgment to substitute intellectually-appropriate questions to probe the tendency for self-harm.

# 7.3 PHARMACOKINETIC ASSESSMENTS

Blood samples for PK assessments of fenfluramine and its metabolite (norfenfluramine) will be obtained from all subjects via an indwelling cannula or by venipuncture.

Blood samples for PK assessment (2 mL) will be obtained at the following time points:

• Part 1 Study Day 43: within 1 hour prior to the morning dose, and 1 ( $\pm$  15 min), 2 ( $\pm$  15 min), and 4-6 hours after the morning dose.

A total of 4 PK samples will be drawn for each subject for a total of approximately 8 mL of blood.

When blood draws for PK coincide with other assessments, the PK draws take precedence.

The procedure for the collection and handling of PK samples is outlined in a separate study manual.

## 7.4 EPILEPSY GENOTYPE PANEL

Optional blood samples for genetic analysis are being collected for a comprehensive analysis for a broad epilepsy gene panel that will be analyzed at the end of the study to investigate


genetic characteristics of study responders and non-responders. Whole genome sequencing is not being performed. Testing is restricted to a 377 childhood epilepsy gene panel; thus, the risk of revealing clinically relevant or medically actionable incidental findings is low. Samples may be retained for up to 24 months after the end of the study.

The field of genetics related to epileptic encephalopathies are developing rapidly, thus, in the event that new theories emerge on the genetics associated with LGS, the retained samples might be used to investigate this genotype in the study population. Results of genetic testing will only be provided upon written request; therefore, unless required by law individual results of genotyping will not be disseminated outside of the Sponsor, including to the study site. Genotyping samples will be double-coded (pseudonymized) so that it is impossible to trace back the personal identifying information from the sample number.

### 7.5 APPROPRIATENESS OF MEASUREMENTS

All of the variables assessed are standard tests or procedures that are commonly used in studies of this type.


## 8. ADVERSE EVENTS

## 8.1 **DEFINITIONS**

## **8.1.1** Adverse Events

According to ICH guidelines, an AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. The period of observation for adverse events extends from the time the subject gives informed consent until the end of study.

## Adverse events may include:

- Exacerbation (ie, an increase in the frequency or severity) of a pre-existing condition. Illness present before study entry should be recorded in the medical history section of the eCRF and only be reported as an AE if there is an increase in the frequency or severity of the condition during the study. Exacerbation of seizures is considered an AE if there was an increase in frequency beyond the subject's typical pre-study fluctuations, or in the event that seizures lengthen in duration in a clinically meaningful way compared with baseline, or if a new seizure type emerges.
- A clinical event occurring after consent but before IMP administration.
- Intercurrent illnesses with an onset after administration of IMP.

## Adverse events do not include:

- Medical or surgical procedures (the condition that leads to the procedure is the AE, eg, tonsillitis is the AE if a tonsillectomy is performed)
- Situations where an untoward medical occurrence has not taken place. For example:
  - Planned hospitalizations due to pre-existing conditions, which have not worsened.
  - Hospitalizations that occur for procedures not due to an AE (eg, cosmetic surgery).
  - Hospitalizations for a diagnostic procedure where the hospital stay is less than 24 hours in duration or for normal management procedures (eg, chemotherapy).

For laboratory safety parameters, any instances of absolute values being outside the reference range or changes at any visit after study start that are considered by the investigator as clinically significant must be recorded in the eCRF as AEs. In addition, at the investigator's discretion, any changes or trends over time in laboratory parameters can be recorded in the eCRF as AEs if such changes or trends are considered to be clinically relevant, even if the absolute values are within the reference range.

Laboratory findings do not need to be reported as AEs in the following cases:


- 1. Laboratory parameters are already beyond the reference range, unless a further increase/decrease can be considered an exacerbation of a pre-existing condition.
- 2. Abnormal laboratory parameters caused by mechanical or physical influences on the blood sample (eg, hemolysis) and flagged as such by the laboratory in the laboratory report.
- 3. Abnormal parameters that are obviously biologically implausible (eg, values that are incompatible with life).
- 4. An abnormal laboratory value that cannot be confirmed after a repeated analysis, preferably in the same laboratory (eg, the previous result could be marked as not valid and should not necessarily be reported as an AE).

## 8.1.2 Serious Adverse Events

A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose:

- 1. **Results in death** The event must be the cause of death for the SAE to meet this serious criterion.
- 2. **Is life-threatening** The term "life-threatening" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it had been more severe.
- 3. Requires in-patient hospitalization or prolongation of existing hospitalization The sponsor considers "hospitalization or prolongation of existing hospitalization" for at least 24 hours as the defining criterion for an SAE. Hospital admissions for planned surgery or for normal disease management procedures (eg, chemotherapy) are not considered as defining criteria for SAEs.
- 4. Results in persistent or significant disability or incapacity.
- 5. Is a congenital anomaly or birth defect.
- 6. **Is medically significant** A medically significant event is defined as an event that does not meet any of the other 5 SAE criteria, but which is judged by a physician to potentially jeopardize the subject or require medical or surgical intervention to prevent one of the above outcomes listed as an SAE criterion. Anaphylaxis that is successfully treated by administration of epinephrine prior to other sequelae is an example of a potentially medically important event.

The most important term should be selected as the criteria for the SAE. Medically significant should be used when none of the other terms apply.

Suspected Unexpected Serious Adverse Reactions (SUSARs) are defined as SAEs that do not meet determination of expectedness as determined in accordance with applicable product information (Investigator's Brochure or other reference documentation). Upon receipt of a SAE report from an Investigator site, all suspected adverse reactions related to the IMP which occur within the clinical trial will be assessed for expectedness. Any SAE not listed in the reference documentation is considered a Suspected Unexpected Serious Adverse Reaction (SUSAR). SUSARs will be reported by the Sponsor, or its designee, in compliance with local legal requirements. During the course of the study, the Sponsor will report within required timelines all SAEs that are both unexpected and at least reasonably related to the IMP (SUSARs) to the Health Authorities, IECs / IRBs as appropriate and to


the Investigators. This study will comply with all applicable regulatory requirements and adhere to the full requirements of ICH Topic E2A (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting [1994]).

For the purpose of data collection in this study, a prolonged seizure or series of seizures from which the subject does not regain consciousness between ictal events, that is at least

30 minutes in duration, is termed status epilepticus (SE). SE should be entered as an SAE if a prolonged seizure or series of seizures persists for 30 minutes or longer, regardless of administration of rescue medication, *and* is either diagnosed by a medical professional or occurs more than once in a day. SE lasting for less than 30 minutes should be entered as an AE, unless one of the other SAE criteria (eg, hospitalization) are met. If this incident involves multiple seizures close in time, the SE definition applies if the seizures are close together such that consciousness is not regained between ictal events.

Adverse events that do not fall into the above categories are defined as nonserious AEs.

## 8.1.3 Adverse Events of Special Interest

As per ICH guidance (E2F Development Safety Update Report [2011]), the sponsor has identified the following AESIs for the ZX008 program (Table 16).

## **Table 16:** Adverse Events of Special Interest

## Metabolic/Endocrine

- 1. Elevated prolactin level  $\ge 2x$  above the upper limit of normal (ULN)
- 2. Hypoglycemia <3.0 mmol/l or 54 mg/dl, whether that level is associated with symptoms or not

## **Neuropsychiatric**

1. Suicidal thoughts, ideation or gestures

## 8.2 SEVERITY OF ADVERSE EVENTS

The severity of AEs (whether nonserious or serious AEs) is to be assessed by the investigator as follows (Table 17).


**Table 17: Severity Definition of Adverse Events** 

| Severity | Definition |
|---|---|
| Mild: | A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. |
| Moderate: | A type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. |
| Severe: | A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. |

#### 8.3 CAUSALITY OF ADVERSE EVENTS

The causal relationship of an AE to IMP must always be assessed by the investigator. All AEs will be classified as either related or not related to IMP. If a causality assessment is not provided for an AE (including an SAE), that AE will be considered as related to IMP.

The degree of certainty with which an AE is attributed to IMP or an alternative cause (eg, natural history of the underlying disease, concomitant medication) will be determined by how well the event can be understood in terms of:

- Known pharmacology of ZX008
- Clinically and/or pathophysiologically plausible context
- Reaction of a similar nature previously observed with similar products, or reported in the literature for similar products as being product related (eg, headache, facial flushing, pallor)
- Plausibility supported by the temporal relationship (eg, the event being related by time to administration or termination of treatment with IMP drug withdrawal or reproduced on rechallenge)

The following classifications should be used in categorization of relatedness:

Not Related: Concomitant illness, accident or event with no reasonable association with study drug.

Related: The event follows a reasonable temporal sequence from administration of study drug and is definitive pharmacologically; cannot to be attributed to concurrent disease or other factors or medications. A clinically reasonable response should be observed if the study drug is withdrawn or dose reduced.

#### 8.4 OBSERVATION PERIOD FOR ADVERSE EVENT REPORTING

The observation period for AE and SAE reporting in an individual subject will start at the time


of giving written informed consent for participation in the current study and finish 15 days after the last dose of study drug or the last visit, whichever is later. For subjects who enroll in the open-label extension (Part 2), ongoing AEs will be followed in that study.

If the investigator becomes aware of an SAE that has started after the observation period has finished, and the event could in some way be associated with IMP (irrespective of whether or not it is considered by the investigator to be causally related to IMP), then this must also be reported to the sponsor (see Section 8.6).

## 8.5 ADVERSE EVENT REPORTING

## **8.5.1** Adverse Events

At each clinical evaluation, the investigator (or delegate) will determine whether any AEs have occurred. Adverse events will be recorded in the AE page of the eCRF. If known, the medical diagnosis of an AE should be recorded in preference to the listing of individual signs and symptoms. The investigator must follow up on the course of an AE until resolution or stabilization. If an AE is ongoing after the end of study visit, the AE will continue to be followed up until resolution or stabilization.

If, during the study period, a subject presents with a pre-existing condition that was not noted at the time of study entry, the condition should be retrospectively recorded in the Medical History section of the eCRF.

# 8.6 SERIOUS ADVERSE EVENTS REPORTING

This study will comply with all applicable regulatory requirements and adhere to the full requirements of ICH Topic E2A (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting [1994]).

In the event of a SAE the investigator or delegate must:

- 1. Enter all relevant information in the AE page of the eCRF
- 2. Inform the safety group and/or the Medical Monitor of the SAE via email or **fax** within 24 hours of becoming aware of the SAE.
- 3. Follow the initial notification with a completed SAE report form. The SAE form must be emailed or faxed to iHC within 24 hours of becoming aware of the SAE.

All SAEs that occur during the course of the study, beginning the day Informed Consent is signed, whether or not causally related to IMP must be reported immediately via fax or email (within 24 hours of the investigator becoming aware of the event) to the sponsor/designee or the Medical Monitor.

Adverse events occurring in the period between the time the subject gave written informed consent and the first exposure to IMP that meet one or more of the seriousness criteria for AEs must be reported to the sponsor/designee and the Medical Monitor in the same manner as other SAEs and will be included in the clinical study database.

Any SAE that occurs 15 days after the last dose of study drug or the last visit, whichever is later that is considered to be causally related to IMP must be reported immediately (ie, within 24 hours of the investigator becoming aware of the event) to the sponsor/designee and the


## Medical Monitor.

e specified by Contact details and guidance for reporting SAEs will be provided to study site before the study starts.

### 8.6.1 Requirements for Immediate Reporting of Serious Adverse Events

The minimum reporting requirements for immediate reporting of SAEs include:

- 1. Identifiable subject
- 2. Suspected drug product
- 3. Event description
- 4. Identifiable reporting

source In addition, the investigator

must:

- 1. Report all SAEs to the relevant IRB/IEC within the timeframe specified by the IRB/IEC.
- 2. Submit follow-up reports to the sponsor Global Clinical Safety and Pharmacovigilance/designee and the Medical Monitor until the SAE has resolved, or, in the case of permanent impairment, until stabilized.
- 3. Ensure that the AE term(s) and causality assessment for all SAEs is entered in the eCRF.

If the minimum requirements for reporting are fulfilled, the investigator should not wait to receive additional information to fully document the event before notifying the sponsor/designee.

When submitting SAE reports to the sponsor/designee, subjects should be identified only by their subject number and study number. The investigator should not include the subject's name and address.

SAE update reports can be submitted to the sponsor/designee any time that additional relevant information becomes available. In cases of death, the investigator should supply the sponsor/designee and the IEC/IRB (as applicable, see Section 8.7) with any additional requested information as it becomes available (eg, autopsy reports and detailed medical reports). Once an SAE is reported to the sponsor/designee's Safety Group, a Safety Specialist may contact the investigator with follow-up questions.

The procedure to be followed if an ongoing AE becomes an SAE after the end of the observation period for AEs is described in Section 8.9.

## REPORTING OF SERIOUS ADVERSE EVENTS BY INVESTIGATOR TO IEC/IRB

The timeframe within an IEC/IRB must be notified of a death or an unexpected SAE considered at least possibly related to the IMP is stipulated by each individual IEC/IRB. The investigator is responsible for complying with the requirements for IEC/IRB notification. The investigator will notify the relevant IEC/IRB within the applicable timeframe by forwarding the


safety report (eg, MedWatch/CIOMS form) completed by the sponsor/designee for the notifiable event.

## 8.8 REPORTING OF EVENTS OTHER THAN SERIOUS ADVERSE EVENTS BY INVESTIGATOR TO SPONSOR

Even if none of the criteria for an SAE are fulfilled, any of the following events must be reported by the investigator to the Medical Monitor within 72 hours from the time the investigator is notified.

- 1. Hypersensitivity reactions
- 2. Pulmonary hypertension
- 3. Cardiac symptoms requiring intervention, or valvulopathy, if identified outside of study-related monitoring

#### 8.9 FOLLOW-UP OF ADVERSE EVENTS

ean AE or lation ( Every effort should be made to follow-up subjects who continue to experience an AE or an SAE on completion of the study or until the AE resolves. All follow-up information (and attempted follow-up contacts) should be documented in the subject's medical records. Details of the subject's progress should also be submitted to the sponsor/designee's Global Clinical Safety and Pharmacovigilance and the Medical Monitor.

Subjects who are discontinued from the study or complete the study and have been found to have any signs of valvulopathy or pulmonary hypertension on ECHO will be followed until the condition has resolved or stabilized where no further changes are likely, for a minimum of

6 months from the last dose of study medication, unless it is determined after unblinding that the subject did not receive ZX008.

## 8.9.1 Follow-up of Echocardiogram Findings

All ECHOs will be evaluated by a central reader, in consultation with the ICAB, if warranted. Findings related to pulmonary hypertension or valvulopathy on any of the four valves (aortic, mitral, pulmonary, tricuspid) will be reported to the investigator with grades of normal, trace, mild, moderate or severe. If the ECHO result has progressed in severity since the last reading then new oversight measures will be enacted as described below in Table 18 which describes the severity of ECHO findings with the level of increasing oversight if the subject is to remain in the study.

Table 18: Clinical Measures Enacted Upon Increasing Severity of ECHO Findings

| | Valve | | | |
|-------------------|---------|---------|-----------|-----------|
| Severity | Aortic | Mitral | Pulmonary | Tricuspid |
| Trace (≤18 years) | Level 2 | Level 2 | Level 1 | Level 1 |
| Trace (>18 years) | Level 1 | Level 1 | Level 1 | Level 1 |
| Mild (≤18 years) | Level 2 | Level 2 | Level 1 | Level 1 |
| Mild (>18 years) | Level 2 | Level 1 | Level 1 | Level 1 |
| Moderate | Level 3 | Level 3 | Level 3 | Level 3 |
| Severe | Level 3 | Level 3 | Level 3 | Level 3 |

Level 1: Continue per protocol


#### Level 2:

- 1. If there is a desire to continue study medication:
  - a. The investigator will evaluate the efficacy to date based on study diaries and consult with the parent/guardian, and determine whether study treatment was associated with significant, meaningful benefit in number, severity and/or duration of seizures and/or on the impact on daily functioning.
  - b. The investigator will consider whether the subject has had reasonable trials (dose and duration) of other available anticonvulsants (eg, valproic acid, clobazam, or topiramate), alone or in combination, and not maintained the level of seizure control achieved with study medication.
- 2. If the investigator feels consideration of continued treatment is warranted considering benefit and potential risk, and the parent/guardian feels strongly that the subject be maintained on the study medication when understanding the risks, the parent/guardian must sign a new consent which describes the additional risks and the subject should provide assent if appropriate.
  - a. If both of these conditions are not met, the subject is discontinued from treatment.
- 3. The investigator prepares a case history and rationale for continuation to be submitted to the IDSMC for review, including consideration of effects on seizures and comorbidities.
- 4. The cardiac reviewers (from the central reader, and potentially ICAB) prepare an evaluation of the cardiopulmonary risks and proposed monitoring plan if applicable, for submission to the IDSMC.
- 5. IDMSC will review the submissions from the Investigator and cardiac central reader and unblind the subject treatment if warranted.
- 6. IDSMC makes a determination of appropriate path, including the possible outcomes:
  - a. Discontinue study medication
  - b. Increase frequency of ECHO and ECG monitoring
  - c. Add additional ECG and/or ECHO measures to be monitored
  - d. Reduce the dose of study medication

#### Level 3:

- 1. The investigator will evaluate efficacy to date based on study diaries and consult with the parent/guardian, and determine whether the achieved benefit justifies the consideration of continuing study treatment by the IDSMC. MINIMAL efficacy criteria for IDSMC consideration:
  - a. Seizures must be more than 75% improved (number of motor seizures per 28 days) on treatment over baseline, and improvement must be consistent.
  - b. The number, type, duration, and distribution of seizures at baseline should be of a severity, which justifies the risks of cardiopulmonary complications, considering the subject's age and overall health.
  - c. Subject has had reasonable trials (dose and duration) of other available anticonvulsants (eg, valproic acid, clobazam, topiramate), alone or in


combination, and not maintained the level of seizure control achieved with study medication.

- 2. If the investigator feels consideration of continued treatment is warranted considering benefit and potential risks, and the parent/guardian feels strongly that the child be maintained on the study medication when understanding the risks, the parent/guardian must sign a new consent, which describes the additional risks and the child should provide assent if possible.
  - a. If both of these conditions are not met, the subject is discontinued from treatment.
- The investigator prepares a case history and rationale for continuation to be submitted
  to the IDSMC for review, which includes effects of study medication on seizures and
  comorbidities related to LGS.
- 4. The cardiac reviewers (from the central reader, and potentially ICAB) prepare an evaluation of the cardiopulmonary risks and proposed monitoring plan if applicable, for submission to the IDSMC.
- 5. IDMSC will review the submissions from the Investigator and cardiac central reader and unblind the subject treatment if warranted.
- 6. IDSMC makes a determination of appropriate path, including these possible outcomes:
  - a. Discontinue study medication
  - b. Increase frequency of ECHO and ECG monitoring
  - c. Add additional ECG and/or ECHO measures to be monitored

#### 8.10 PREGNANCY

This study is open to female and male subjects. Whenever possible, a pregnancy in a female subjects or the female partner of a male subject exposed to IMP should be followed to term so as to assess any potential occurrence of congenital anomalies or birth defects. Any follow-up information, including premature termination and the status of the mother and child after delivery, should be reported by the investigator to the sponsor/designee using a pregnancy reporting/outcome form.

## 9. DATA HANDLING PROCEDURES

## 9.1 RECORDING OF DATA

The investigator (or delegate) will maintain individual records for each subject. These records should include dates when a subject visited the study site, study-required information and data, and other notes as appropriate. These records constitute source data.

An eCRF and a subject diary will be provided by the sponsor (or delegate) for each subject enrolled into the study. Study site staff will enter data directly into the validated electronic data capture (EDC) system by completing the eCRF via a secure internet connection. The investigator is responsible for ensuring accurate and proper completion of the eCRF and subject diary for recording data according to the instructions given in the eCRF and subject diary.

All entries in the eCRF must be backed up by the relevant source data at the study site. All source data will be kept according to all applicable regulatory requirements (see Section 12.8). Source data must follow good documentation practices, be completed legibly for each subject


enrolled into the study and signed by the investigator (or delegate).

Data entry in the eCRF and subject diary must be completed in a timely manner so that they always reflect the latest observations on the subjects enrolled in the study.

The subject's diary will be completed by the parent/caregiver at home. Data entries will be reviewed by the investigator for completion and consistency.

#### 9.2 DATA QUALITY ASSURANCE

An initiation meeting will be held before starting the study, during which the study design, procedures to be followed, and measures for ensuring standardized performance will be explained by a delegate from the sponsor, and a common understanding of the requirements of the study will be reached with the investigator and other relevant personnel at the study site.

Data generated throughout the study will be monitored and the data entered in the eCRFs will be checked against the subject records for completeness and accuracy. The sponsor's study monitor will perform this function.

The computer system used for study data handling will be fully FDA 21 CFR Part 11 compliant. All creation, modification or deletion of electronic study records will be documented through an automated Audit Trail. Following completion of eCRF pages and entry of the data into a database, the data will be checked electronically for consistency and plausibility. Data queries will be generated for questionable data and response clarification will be sought from the investigator. These data queries must be resolved in a timely manner by the investigator (or delegate).

#### 9.3 RECORD RETENTION

A study document binder will be provided by the sponsor for the investigator at each site for all requisite study documents (constituting the "Investigator Study File").

Following completion of the study, the investigator will retain copies of the approved study protocol, ICF, relevant source documents, and all other supporting documentation related to the study according to applicable regulatory requirements.

The investigator is responsible for archiving the Investigator Study File, the subject's records, and the source data according to applicable regulatory requirements. These documents have to be archived for at least 15 years or at least 2 years after the last approval of a marketing application in an ICH region, but should be retained for longer if required by regulatory requirements or by agreement with the sponsor.

If the investigator can no longer maintain the archive of study records (eg, due to retirement or relocation), the sponsor must be informed in writing about any change in responsibility for record retention, including the name of the new responsible party, contact information, and location of the study records. Records may not be destroyed without prior written consent from the sponsor.


#### 10. STATISTICS

#### 10.1 STATISTICAL ANALYSIS: PART 1

The primary analyses of the study will be performed on data from Part 1 Cohort A after the last subject enrolled in Cohort A has completed the last study visit of Part 1. Data from Part 1, Cohort B will be analyzed independently after the last subject in Cohort B completes Part 1. An interim analysis of Part 2 will be performed after all Cohort B subjects complete 12 months in Part 2. A secondary analysis will be conducted after the last Cohort B subject has enrolled and completed the last study visit of Part 2. Analysis results for Part 1 from Cohort A and Cohort B will be compared through descriptive statistics, and if reasonable, some analysis may be performed using data from Cohort A and Cohort B combined. Subjects randomized to 0.5 mg/kg/day (ie, those taking concomitant STP) will be grouped with subjects randomized to 0.8 mg/kg/day for all efficacy analyses.

#### 10.1.1 DETERMINATION OF SAMPLE SIZE

The sample size for Part 1 Cohort A was estimated under the assumption that adding ZX008 at 0.8 mg/kg/day to current therapy will lead to a mean decrease in drop seizures that is 30 percentage points greater than adding placebo to current therapy. For example, if adding placebo leads to a 10% decrease in seizures, then adding the high dose of ZX008 would be expected to decrease seizures by at least 40%.

The variability expected in the trial was estimated from a Phase 3 trial of clobazam for patients with Lennox-Gastaut syndrome (Ng 2011) leading to an assumption that the SD is 50%. Other assumptions include an allowance for 20% dropouts between randomization and the start of the maintenance period.

Under these assumptions, and using a Wilcoxon rank-sum test to approximate the primary comparison between the ZX008 0.8 mg/kg/day and placebo groups, a sample size of 63 subjects per treatment group affords 90% power to detect a difference between groups that is significant at the  $\alpha$ =0.05 level. Assuming a 20% drop-out rate prior to the start of the maintenance period yields a requirement for an additional 16 subjects per group for a total of 79 subjects per treatment group. Similar calculations for the 0.2 mg/kg/day ZX008 group lead to a total required sample size of 237. The number of subjects randomized into Part 1 Cohort A is estimated to be approximately 250 due to the long baseline period.

The sample size of 10 to 15 subjects per treatment group in Cohort B is expected to provide a descriptive assessment of whether the treatment effect in Japanese subjects is similar that observed in Cohort A subjects from the rest of the world.

## 10.1.2 ANALYSIS POPULATIONS

#### 10.1.2.1 Safety (SAF) Population

All Part 1 safety analyses will be performed on the SAF Population defined as all randomized subjects who receive at least one dose of ZX008 or placebo.


#### 10.1.2.2 Modified Intent-to-Treat (mITT) Population

The mITT Population is defined as all randomized subjects who receive at least one dose of ZX008 or placebo and for whom at least one week of diary data are available. Subjects will be analyzed according to the treatment group to which they were randomized. The primary comparison of ZDX008 0.8 mg/kg/day to placebo, who complete at least 4 weeks of diary data in the maintenance period, as well as key secondary analyses, will be performed on the mITT Population.

#### 10.1.2.3 Per Protocol (PP) Population

The PP Population is defined as all randomized subjects who receive at least one dose of ZX008 or placebo, and have no major protocol deviations that would have a significant impact on clinical outcome.

#### 10.1.3 SUBJECT COHORTS

#### 10.1.3.1 Cohort A

Cohort A comprises all randomized subjects from North America, Europe, and Australia

#### 10.1.3.2 Cohort B

Cohort B comprises all randomized subjects from Japan only.

#### 10.1.4 TREATMENT GROUPS

Subjects will be randomly assigned to one of three treatment groups: ZX008 0.8 mg/kg/day, ZX008 0.2 mg/kg/day, or placebo.

#### 10.1.5 TREATMENT PERIODS

#### **Baseline Period**

The Baseline Period covers the 28 days immediately prior to randomization. The baseline frequency of seizures that lead to drops will be calculated from data collected during this period.

#### **Titration Period**

The Titration Period covers the first 14 days of treatment while subjects are titrated to their randomized dose. It begins on the first full day of treatment (Study Day 1) and extends through Study Day 15 regardless of the exact day on which a subject reaches his or her assigned dose. The Titration Period applies to all subjects including placebo recipients.

## Maintenance Period

The Maintenance Period covers the 12 weeks following the end of the titration period. It begins on Study Day 16 and extends through Study Day 99.

#### Titration + Maintenance (T+M) Period

The T+M period combines the Titration and Maintenance periods, beginning on Study Day 1 and extending through Study Day 99. The T+M period is considered the treatment period.

#### Taper/Transition Period

The Taper/Transition Period begins immediately at the end of T+M period and extends to Visit


13, 2 weeks later; ie, from Study Day 99 through Study Day 113.

#### STATISTICAL ANALYSES AND METHODS 10.1.6

A complete description of the statistical analyses and methods will be available in a SAP which will be finalized before the database is locked.

10.1.6.1 Efficacy Analyses

Primary Efficacy Analysis

The primary efficacy endpoint for Part 1 is the percent change in frequency per 28 day daintenance (T+M) and Baseline as vailable data soll

available data collected during the Baseline and T+M Periods without imputation. The percent change from baseline DSF will be calculated as the the change in DSF between T+M and Baseline / DSF during Baseline × 100. Both the mean and median percent change in DSF Both the mean and median percent change in DSF will be presented.

The primary endpoint will be assessed using a nonparametric, rank analysis of covariance (ANCOVA) with treatment group (ZX008 0.8 mg/kg/day, ZX008 0.2 mg/kg/day or placebo) and weight group (<37.5 kg,  $\ge 37.5 \text{ kg}$ ) as factors; rank baseline DSF as a covariate; and rank percent change in DSF from baseline as the response variable. The primary analysis will compare the ZX008 0.8 mg/kg/day group to the placebo group at the  $\alpha$ =0.05 level of significance. The difference between the ZX008 0.8 mg/kg/day group and the placebo group in percent change in DSF, and its 95% confidence interval, will be estimated using the Hodges-Lehmann method.

As a sensitivity analysis, the primary endpoint will also be analyzed using a parametric ANCOVA that incorporates treatment group and weight group as factors; log baseline DSF as a covariate; and log DSF during T+M as the response variable. Significance will be assessed by a model contrast that compares the ZX008 0.8 mg/kg/day group to the placebo group. The size of the treatment effect will be estimated by exponentiating the difference between the ZX008 0.8 mg/kg/day group and the placebo group derived from the model. Another sensitivity analysis will compare the ZX008 0.8 mg/kg/day group to the placebo group using a Wilcoxon rank-sum

#### Key Secondary Analyses

The first key secondary endpoint for the ZX008 0.8 mg/kg/day group – the proportion of subjects who achieve a ≥50% reduction from baseline in the frequency of seizures that result in drops – is derived directly from the primary endpoint, but is widely considered a benchmark for clinical meaningfulness of a medical intervention for seizures. The comparison will be made using a logistic regression model that incorporates the same factors and covariate as the ANCOVA used in the primary analysis. The second key secondary endpoint – the proportion of


subjects assessed by the Investigator as minimally, much, or very much improved on the CGI-I will be analyzed using a Cochran-Mantel-Haenszel test (CMH) stratified by weight strata.

The percent change from baseline DSF in the ZX008 0.2 mg/kg/day group will be compared to the placebo group using the same methods employed for the primary analysis. In particular, the same ANCOVA model will be used. Nonparametric methods will be used if normality assumptions do not hold. Analyses of other key secondary endpoints involving the ZX008 0.2 mg/kg/day group will employ similar methods as those used to compare ZX008 0.8 mg/kg/day to placebo.

#### Multiplicity Strategy and Testing Hierarchy

The efficacy analyses will employ a serial gatekeeper strategy to maintain the Type 1 error rate at  $\alpha$ =0.05 across the family of analyses that support the primary and key secondary objectives. The strategy specifies a hierarchy of significance tests where each test acts as a gatekeeper to the tests below it.

The hierarchy starts with the primary analysis comparing ZX008 0.8 mg/kg/day to placebo on the percent change from baseline in DSF. The next two steps in the hierarchy also entail comparisons of ZX008 0.8 mg/kg/day to placebo on two key secondary endpoints. The last three steps in the hierarchy all involve comparisons of ZX008 0.2 mg/kg/day to placebo.

Below is a complete list of steps in the testing hierarchy in order:

- 1. Compare ZX008 0.8 mg/kg/day to placebo on the percent change in DSF from baseline in DSF.
- 2. Compare ZX008 0.8 mg/kg/day to placebo on the proportion of subjects who achieve a  $\geq$ 50% reduction from baseline in DSF.
- 3. Compare ZX008 0.8 mg/kg/day to placebo on the change from baseline in the number of all countable motor seizures.
- 4. Compare ZX008 0.2 mg/kg/day to placebo on the percent change from baseline in DSF.
- 5. Compare ZX008 0.2 mg/kg/day to placebo on the proportion of subjects who achieve a ≥50% reduction from baseline in the DSF.
- 6. Compare ZX008 0.2 mg/kg/day to placebo on the CGI-I at Visit 12.

#### Part 1 Cohort B

Efficacy analyses for Part 1 Cohort B will use the same methods as described for Part 1 Cohort A. Some subsets analyses may not be feasible in Cohort B due to its smaller sample size.

#### 10.1.6.2 Safety Analyses

Summaries of safety data will be presented by treatment – ZX008 0.8 mg/kg/day, ZX008 0.2 mg/kg/day or placebo – for the T+M period. The number and percentage of subjects in each treatment group with AEs will be displayed by body system and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). Summaries of AEs by severity and relationship to study drug will also be presented. A separate summary will be provided for all


serious AEs (SAEs). If warranted, selected summaries will be repeated broken out by weight group, ie, for subjects who weigh <37.5 kg and those who weigh ≥37.5 kg.

Laboratory tests, vital signs, physical examinations, neurological examinations, ECG, Doppler echocardiogram, C-SSRS, Tanner Staging results, etc, will be summarized appropriately, by treatment. All safety summaries will be based on the SAF Population.

#### 10.1.6.3 Pharmacokinetic Analyses

Model-derived plasma PK parameters of fenfluramine and norfenfluramine ( $C_{max\_ss}$ ,  $C_{min\_ss}$ ,  $AUC_{0-t}$ ,  $AUC_{0-t}$ ) will be summarized descriptively by treatment group when sufficient data are available. A population PK model, previously developed using data from healthy adults and pediatric patients with Dravet syndrome, will updated to include the fenfluramine and norfenflurmaine concentration-time data collected during the Maintenance Period. This model will be informed by all relevant data available at the time of data collection (both adults and pediatrics). The results from the PopPK modeling will be reported separately and conducted according to a separate SAP.

#### 10.2 STATISTICAL ANALYSIS: PART 2

Safety and effectiveness will be assessed in the subjects who continue into Part 2 of the study in which all subjects receive open-label ZX008.

#### 10.2.1 ANALYSIS POPULATIONS

#### **10.2.1.1 OLE Population**

Safety analyses for Part 2 will be performed on the OLE Safety Population defined as all subjects who receive at least one dose of ZX008 during the open label extension.

### 10.2.1.2 OLE mITT Population

The OLE mITT Population is defined as all randomized subjects who receive at least one dose of ZX008 and have valid seizure data during the open label extension.

#### 10.2.2 TREATMENT GROUPS

All subjects in Part 2 will receive ZX008 and will be considered a single treatment group. Selected data summaries may be broken out by the treatment received during Part 1 and/or average dose received during Part 2.

#### 10.2.3 TREATMENT PERIODS

Open-Label Extension (OLE) Treatment Period

The OLE Treatment Period covers the duration during which subjects receive open label treatment with ZX008.

#### **OLE Taper Period**

The OLE Taper Period begins immediately after the OLE Treatment period and extends for 2 weeks.


#### 10.2.4 STATISTICAL ANALYSES AND METHODS

#### 10.2.4.1 Safety Analyses

The number and percentage of subjects who experience treatment emergent AEs will be displayed by body system and preferred term using MedDRA. Summaries in terms of severity and relationship to study drug will also be provided. SAEs will be summarized separately in a similar manner. Laboratory tests, vital signs, physical examinations, neurological examinations, ECG, ECHO, cognition and body weight will be summarized using appropriate methods.

#### 10.2.4.2 Effectiveness Analyses

Effectiveness will be assessed by the change from baseline (prior to randomization into Part 1) in DSF. The DSF per 28 days will be calculated as the number of seizures recorded divided by the number of days in the period and multiplied by 28. The change in DSF during the OLE Treatment Period will be calculated as the difference between DSF during the OLE and the baseline DSF measuredprior to randomization in Part 1. The percent change in DSF is the change in DSF between OLE and Baseline / DSF during Baseline x 100. Both the mean and median percent change in DSF will be presented and the statistical significance of the percent change will be assessed using a Wilcoxon signed-rank test. Other secondary assessments will be compared to baseline from prior to Part 1, or by visit throughout Part 1 and Part 2, as appropriate.

For subjects continuing in Part 2 past Visit 22, effectiveness will be assessed by investigator rating of overall change in seizure frequency (<25%,  $\ge25\%$ ,  $\ge50\%$ , or  $\ge75\%$ , 100% (seizure-free) improvement compared to last visit).

# 10.2.5 ANALYSES PROVIDED TO AN INDEPENDENT DATA AND SAFETY MONITORING COMMITTEE

A safety oversight monitoring plan will be in place with an IDSMC evaluating data from the subjects. Details will be provided in the IDSMC charter. The IDSMC's primary responsibility is to ensure that study subjects are not exposed to unanticipated harm that could have been prevented by timely review and intervention. The IDSMC is established to review safety data at predefined time points, and to recommend to the sponsor whether to continue, modify, or terminate the study as necessary. The IDSMC is composed of expert permanent members who cover relevant specialties. The IDSMC members may request assistance from a number of additional and ad hoc members if needed.

#### 11. ETHICAL & REGULATORY CONSIDERATIONS

#### 11.1 CETHICAL CONSIDERATIONS

The procedures set out in this study protocol are designed to ensure that the sponsor and the investigator abide by the principles of the current ICH GCP guideline on the conduct, evaluation and documentation of this study, as described in ICH Topic E6 Guideline. ICH GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are


protected and consistent with the principles of the Declaration of Helsinki, and that the clinical study data are credible.

The study will also be carried out according to all applicable international and national regulatory requirements.

The sponsor and the investigator must inform each other (eg, during a study initiation visit, via e-mail, etc) that all ethical and legal requirements have been met before the first subject is enrolled into the study.

#### 11.2 INFORMED CONSENT

The investigator is responsible for obtaining a subject's written informed consent to participate in the study.

A Subject Information Sheet and a master ICF will be prepared by the sponsor according to the provisions of ICH GCP and local legal requirements.

All subjects will be informed that the study will be registered in the public database at ClinicalTrials.gov in accordance with the FDA Amendments Act of 2007 (Section 12.3).

Before undergoing screening procedures for possible enrollment into the study, subjects must be informed, in an understandable form, about the nature, scope, and possible consequences of the study. This information must be given orally to subjects by a physician or medically qualified person (according to applicable regulatory requirements) who is well informed about the nature, scope, and possible consequences of the study. Written information about the study will also be provided in a Subject Information Sheet. The date on which this oral and written information on the study was provided to the subject, and by whom it was provided, must be documented in the ICF.

As specified in ICH GCP Section 4.8 and the US 21CFR Section 50.25, the informed consent discussion must emphasize that participation in the study is voluntary and that subjects have the right to withdraw their consent at any time without giving a reason and without any disadvantage for their subsequent care.

Subjects must be given ample time and opportunity to inquire about details of the study and to consider their participation in the study. If, after reading the Subject Information Sheet and the ICF, consent is given to participate in the study, then the ICF must be signed and personally dated by the subject and the person conducting the informed consent discussion (and an impartial witness, if required). The subject will be provided with a copy of the signed ICF.

Verification of the signed ICF will be recorded in the subject's eCRF. The original signed ICF will be filed with the subject's records and/or in the Investigator Study File.

The Subject Information Sheet and ICF have to be approved by the IEC/IRB before they can be used in the study.

The Subject Information Sheet and ICF must be revised whenever important new information becomes available that may be relevant to the subject's consent. Any revision of these documents must be approved by the IEC/IRB before they can be used in the study. Subjects must be informed in a timely manner if new information becomes available that may be relevant to their willingness to continue participation in the study. The communication of this


information should be documented by having all parties concerned sign and personally date the revised ICF.

#### Subject or Subject's Legally Acceptable Representative Unable to Read

If a subject is unable to read, or if a legally acceptable representative is unable to read, an impartial witness should be present during the entire informed consent discussion. After the ICF and any other written information provided to the subject, parent or guardian has been read and explained to the subject or the subject's legally acceptable representative, and after the subject or the subject's legally acceptable representative has orally consented to the subject's participation in the study and, if capable of doing so, has signed and personally dated the ICF, the witness should also sign and personally date the ICF. By signing the ICF, the witness attests that the information in the ICF and any other written information was accurately explained to, and apparently understood by, the subject or the subject's legally acceptable representative, and that informed consent was freely given by the subject or the subject's legally acceptable representative.

### Assent for Subjects Under the Age of Consent (Pediatric Subjects)

All subjects are under the age of consent (ie, pediatric subjects under 18 years of age); the written informed consent of a legally acceptable representative is required. Pediatric subjects who can understand the nature, scope, and possible consequences of the study must also give their assent, orally and/or in writing via the assent document, as appropriate. After the ICF and any other written information to be provided to subjects has been read and explained to the subject and the subject's legally acceptable representative, and after the subject and the legally acceptable representative have orally consented to the subject's participation in the study and, if capable of doing so, the subject has signed and personally dated the assent document, the legally acceptable representative should sign and personally date the ICF. By signing the ICF, the legally acceptable representative attests that the information in the ICF and any other written information was accurately explained to, and apparently understood by, the subject, and that assent was freely given by the subject.

# 11.3 REGULATORY CONSIDERATIONS AND INDEPENDENT ETHICS COMMITTEE/INSTITUTIONAL REVIEW BOARD

The sponsor (or delegate) will submit the appropriate documents to all applicable competent regulatory authorities and IEC/IRBs, and will await all relevant approval before enrolling any subjects into the study. Written approval should mention the study protocol by study title, study number, and version date.

This study will be conducted under Investigational New Drug (IND) Application and documented in accordance with the applicable regulatory guidelines and requirements.

The sponsor (delegate) will ensure that the investigators conduct the study as stipulated in this study protocol and in accordance with all applicable regulatory requirements. The sponsor (delegate) is obliged to obtain evidence of the investigator's qualification to perform the clinical study. Therefore, the investigator has to provide a signed and dated copy of his or her professional curriculum vitae (prepared no more than 2 years beforehand and preferably written in English) before the start of the study, including information on his or her experience in conducting


clinical studies according to ICH GCP and other applicable regulatory requirements.

Written notification of the identity and occupation of the members of the IEC/IRB is also required by the sponsor (delegate). Should the IEC/IRB be unwilling to provide this information, a letter stating that the committee was constituted in accordance with applicable regulatory requirements should be provided.

#### 11.4 PROTOCOL COMPLIANCE

The investigator must conduct the study in compliance with this study protocol as agreed to by the sponsor and, if required, by any competent regulatory authority, and which has been approved by, or given a favorable opinion by, the IEC/IRB.

The investigator should not implement any deviation from, or changes to, the study protocol without agreement by the sponsor (delegate) and prior review and documented approval or favorable opinion from the IEC/IRB of an amendment to the study protocol. Exceptions include only cases of medical emergency to address immediate hazards to study subjects, or when the changes involve only logistic or administrative aspects of the study.

In the event of a medical emergency, the investigator at each site may institute any medical procedures deemed appropriate to address an immediate hazard to a subject without prior IEC/IRB approval or favorable opinion. As soon as possible, the implemented deviation or change, the reason(s) for it, and, if appropriate, the proposed study protocol amendment(s) should be submitted to:

- The sponsor (delegate) for agreement.
- The IEC/IRB for review and approval or favorable opinion (if required).
- The applicable competent regulatory authority (if required).

Details of the procedure for implementing study protocol amendments are available in Section 12.10.

At the earliest opportunity, the investigator (or delegate) must inform the sponsor (delegate) about any notable protocol deviations and explain any deviation from the approved study protocol in the eCRF and/or in the Protocol Deviation Log, if applicable.

#### 12. ADMINISTRATIVE ASPECTS

#### 12.1 CLINICAL TRIAL AGREEMENT

This study will be conducted under a Clinical Trial Agreement between the sponsor (or delegate) and the respective institutions representing the study sites. Any financial support given to the study sites will be detailed in the Clinical Trial Agreement. The Clinical Trial Agreement, which must be signed before the start of any study related procedures, will clearly delineate the responsibilities and obligations of the investigator and the sponsor (delegate), and will form the contractual basis upon which the study will be conducted.

#### 12.2 FINANCIAL DISCLOSURE BY INVESTIGATOR

Prior to study initiation, the investigator and any subinvestigator(s) to be directly involved in


the treatment or evaluation of study subjects at each study site will disclose to the sponsor (delegate) any relevant financial or proprietary interests in either the study product or the sponsor company. The appropriate disclosure form(s) will be provided by the sponsor provided by the investigator and subinvestigator (s) to the sponsor (delegate). All financial disclosure information provided by the investigator and subinvestigator(s) will be submitted to appropriate competent authorities according to the applicable regulatory requirements

12.3

CLINICAL COMMON AND ADDRESS AND ADD (delegate) for this purpose. Any relevant updates to the financial disclosure information that

#### CLINICAL STUDY REGISTRATION AND RESULTS DISCLOSURE 12.3

The sponsor will provide the relevant study protocol information in a public database (ClinicalTrials.gov) before or at commencement of the study, as required by the 2007 FDA Amendments Act. The sponsor (delegate) may also provide study information for inclusion in national registries according to local regulatory requirements.

If a potential subject contacts the sponsor regarding participation in the study, the investigator agrees that the sponsor (delegate) may forward the relevant study site and contact details to the subject. Based on the inclusion and exclusion criteria for the study, the investigator will assess the suitability of the subject for enrollment into the study. Results of this study will be disclosed according to the relevant regulatory requirements. All publications in peer-reviewed medical journals resulting from this study will be listed in the original study protocol registration record on ClinicalTrials.gov.

#### STUDY FILES AND MATERIALS 12.4

Before the start of any study related procedures, all essential documents specified by ICH GCP and other applicable regulations must be available in the relevant files maintained by the sponsor (or delegate) and the investigator. An Investigator Study File prepared by the sponsor (or delegate), containing all applicable documents for use at the study site, will be made available to the investigator before the start of the study. A list of personnel and organizations responsible for conduct of the study as well as the list of investigators will be included in the Investigator Study File. The respective files will be kept and updated by the sponsor (or delegate) and the investigator, as applicable.

All study documentation and materials maintained in the Investigator Study File at the study site must be available for inspection by the sponsor's study monitor (or delegate) to determine that all required documentation is present and correct (see Section 12.9).

The study may be audited or inspected by qualified delegates from the sponsor or a competent regulatory authority (see Section 12.11).

#### INITIATION OF THE STUDY

Before the start of the study at each study site, the sponsor's study monitor (or delegate) will ensure adequacy of the facilities and discuss responsibilities regarding study protocol adherence with the investigator and other personnel involved in the study.

The investigator may not enroll any subjects into the study before the sponsor has received written approval or a favorable opinion from the IEC/IRB for conducting the study and a


formal meeting has been conducted by the sponsor's study monitor (or delegate) to initiate the study (study initiation visit).

#### 12.6 SUBJECT REIMBURSEMENT

Where relevant, subjects will be reimbursed for reasonable travel costs associated with participation in this study, after presentation of receipts for the travel in question, at a rate to be approved by the IEC/IRB. Subjects will not be paid for participating in the study.

#### 12.7 LIABILITY AND INSURANCE

The civil liability of the involved parties with respect to financial loss due to personal injury and other damage that may arise as a result of this study being conducted are governed by the applicable legal requirement(s).

The sponsor will provide insurance to the investigator if required by the applicable regulatory and legal requirement(s).

If required by local law, subjects taking part in this study will be insured against any injury caused by the study in accordance with the applicable regulatory and legal requirement(s).

#### 12.8 SUBJECT IDENTIFICATION AND CONFIDENTIALITY

All study documents, including the study protocol and eCRFs, are the confidential property of the sponsor and should be treated as such.

All subjects screened for the study will be documented in a screening log in compliance with the requirements of individual study sites. Subjects not enrolled into the study will be documented as such in the screening log together with the reason for not having been enrolled.

The investigator will maintain a personal list of subject names and subject numbers (Subject Identification List) for participants in the study to enable records to be identified at a later date. These records should be retained in a confidential manner for the duration stipulated by applicable regulatory requirements. All subject names will be kept in confidence and will not be revealed to the sponsor. Subject names must be made unreadable on any documents made available to the sponsor.

Subjects participating in the study will be identified in the eCRF by the subject number allotted to them during the study.

The ICF will include a statement that all study findings, irrespective of the medium on which they are stored, will be handled in strictest confidence in accordance with applicable data protection laws (eg, the European Data Protection Directive [95/46/EC] and the USA Health Insurance Portability and Accountability Act [HIPAA]), and will be evaluated by the sponsor and/or a competent regulatory authority in an anonymized form. The subjects are also to be informed that their medical records may be audited or inspected by qualified delegates from the sponsor or a competent regulatory authority. The subject's written consent authorizing direct access to his medical records, and computer processing and publishing of his anonymous personal data, must be obtained prior to participation in the study.

A subject's identity will be disclosed by the investigator only in case of emergency (ie, to address any immediate health hazard).


#### 12.9 MONITORING OF THE STUDY

The investigator at each site will allow the sponsor's study monitor (or delegate) reasonable access to the eCRFs and direct access to related source documents for monitoring purposes as frequently as the sponsor deems necessary. These documents include records of tests performed as a requirement for participating in the study as well as other medical records required to confirm information contained in the eCRF, such as past history and secondary diagnoses.

Before each monitoring visit, the investigator (or delegate) should record all data generated since the last monitoring visit in the eCRF. The investigator and other relevant personnel at each study site will be expected to cooperate with the sponsor's study monitor to assist in providing any missing information.

The study monitor will require access to the Investigator Study File to ensure completeness of all documentation required for the study. The study monitor will ensure that the investigator at each site has been provided with adequate means for organization and filing of study documentation (see Section 12.4).

The date on which the study monitor (or delegate) visits the study site will be recorded in the Site Visit Log. During monitoring visits, the study site's coordinator (if applicable) and the investigator should be available, the source documentation should be accessible, and a suitable environment should be provided for the study monitor to review study related documentation.

The main objectives of monitoring visits conducted by the study monitor include:

- Resolution of any problems.
- Examination of all study documentation for completion, adherence to the study protocol, and possible AEs.
- Clarification of inconsistencies or missing data.
- Verification of study data against source documents.
- Checks that investigator obligations have been fulfilled.
- Review of ICFs and dates of consent.
- Inspection of IMP with respect to storage, labeling, and documentation.
- Drug accountability

After each subject's visit to the study site, the investigator (or delegate) will ensure that all data have been entered into the eCRF correctly and in a timely manner, after which the investigator will sign the eCRF.

#### 12.10 PROTOCOL AMENDMENTS

A "substantial" amendment of a study protocol is any written description of change(s) to, or formal clarification of, a study protocol that may have a significant impact on the safety or physical or mental integrity of subjects, the scientific value of the study, the conduct or management of the study, or the quality or safety of any IMP used in the study. The IEC/IRB must approve all substantial protocol amendments prior to their implementation. If required by


applicable local regulatory requirements, the local regulatory authority must also approve all substantial protocol amendments prior to their implementation.

A "non-substantial" amendment of a study protocol includes minor corrections or clarifications that have no significant impact on the way the study is to be conducted and has no effect on the safety of participating subjects (eg, change in study monitor, contact details, etc). If required by applicable local regulatory requirements, the IEC/IRB, and/or the local regulatory authority should be notified of all non-substantial protocol amendments. The substantial and non-substantial protocol amendments will be integrated into an updated study protocol at the discretion of the sponsor if the changes to the original study protocol are numerous, or if required by applicable regulatory requirements.

#### 12.11 AUDITS AND INSPECTIONS

The study may be audited or inspected by qualified delegates from the sponsor or a competent regulatory authority.

In the event of an audit by the sponsor, the investigator must make all study related documentation available to the auditor(s). Regulatory authorities may request access to all study related documentation, including source documents, for inspection and copying in keeping with applicable regulations. The sponsor will immediately notify the investigator (or vice versa) of an upcoming audit or inspection.

If an audit or inspection occurs, the investigator and relevant personnel at the study site must allocate sufficient time to discuss the findings and any relevant issues.

### 12.12 CLINICAL STUDY REPORT

After completion of the study, a clinical study report covering clinical and statistical aspects of the study will be prepared by the sponsor (or delegate) in consultation with the coordinating investigator. As required by the applicable regulatory requirements, the clinical study report will be signed by the sponsor's responsible medical officer as well as the coordinating investigator (if applicable).

Progress reports and/or a summary of the clinical study report will be provided to the IEC/IRB and competent regulatory authorities in accordance with applicable requirements.

#### 12.13 USE OF DATA AND PUBLICATIONS

The rights and obligations of investigators and the sponsor concerning any formal presentation or publication of data collected as a direct or indirect result of this study will be addressed specifically in the Clinical Trial Agreement for the study (see Section 12.1).

For multicenter studies, the first publication must be based upon all data obtained from all analyses, as stipulated in the study protocol by the biostatistician and not by the investigators. Investigators participating in multicenter studies must agree not to present data gathered individually or by a subgroup of study sites before the full, initial publication is available or

5 years after the last clinical study visit, whichever is later, unless this has been agreed to by all other investigators and by the sponsor.

The sponsor must receive a copy of any intended communications in advance of the proposed


Jude el from the e


#### 13. REFERENCE LIST

Aicardi J and Gastaut H. Treatment of self-induced photosensitive epilepsy with fenfluramine (3 cases). NEJM 1985; Nov 28;313(22):1419.

Aicardi J, Gastaut H, and Misès J. Syncopal attacks compulsively self-induced by Valsalva's maneuver associated with typical absence seizures. A case report. Arch Neurol 1988 Aug;45(8):923-5.

Arzimanoglou A, French J, Blume WT, Cross JH, et al. Lennox-Gastaut syndrome: a consensus approach on diagnosis, assessment, management, and trial methodology. Lancet Neurol 2009;8(1):82-93.

Boel M and Casaer P. Add-On therapy of fenfluramine in intractable self-induced epilepsy. Neuropediatrics. 1996; 27: 171-173.

Casaer P and Boel M. Fenfluramine as a potential antiepileptic drug. Epilepsia. 2002; 43(2): 205-206.

Center for Disease Control. Cardiac valvulopathy associated with exposure to fenfluramine or dexfenfluramine: U.S. Department of Health and Human Services Interim Public Health Recommendations, November 1997. Morbidity and Mortality Weekly Report. 1997; 46(45):1061-1084.

Ceulemans B, Boel M, Leyssens K, Van Rossem C, Neels P, Jorens PG, Lagae L. Successful use of fenfluramine as an add-on treatment for Dravet syndrome. Epilepsia 2012; 53: 1131-1139.

Ceulemans B, Schoonjans A, Marchau F, Paelinck B, Lagae, L. Five-year extended follow-up status of 10 patients with Dravet syndrome treated with fenfluramine. Epilepsia 2016; 1-6.

Connolly HM, Crary JL, McGoon MD, Hensrud DD et al. Valvular heart disease associated with fenfluramine-phentermine, New Engl J Med 1997;337(9):581-8. Erratum in: N Engl J Med 1997 Dec 11;337(24):1783.

Cross JH. Auvin S, Falip M, Striano P, Arzimanoglou A. Expert opinion on the management of Lennox-Gastaut syndrome: treatment algorithms and practical considerations. Front Neurol. 2007;8:505.

Hancock EC, Cross JH. Treatment of Lennox-Gastaut syndrome. Cochrane Database of Systematic Reviews 2013, Issue 2. Art. No.: CD003277. DOI: 10.1002/14651858.CD003277.pub3.

ICH Topic E2F: Development Safety Update Report, 2011.

ICH Topic E2A: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting, 1994.

Kim KR, Lee E, Namkoong K, Lee YM, Lee JS, and Kim HD, "Caregiver's burden and quality of life in mitochondrial disease," Pediatric Neurology, vol. 42, no. 4, pp. 271–276, 2010.

Lagae L, Schoonjans A, Gammaitoni AR, Galer BS, Ceulemans B. A pilot, open-label study of


the effectiveness and tolerability of low-dose ZX008 (fenfluramine HCl) in Lennox-Gastaut syndrome. Epilepsia, 2018; doi: 10.1111/epi.14540

Lagae B, Schoonjans A, Gammaitoni A, Galer B, and Ceulemans B. A pilot, open-label study of the effectiveness and tolerability of low dose fenfluramine (ZX008) in Lennox-Gastaut syndrome: Findings from a long-term extension. American Epilepsy Society Annual Meeting 2017: Abstract 2.284.

Lancellotti P, Tribouilloy C, Hagendorff A, Moura L, Popescu BA, Agricola E, et al. European Association of Echocardiography recommendations for the assessment of valvular regurgitation. Part 1: aortic and pulmonary regurgitation (native valve disease). Eur J Echocardiogr. 2010;11(3):223-244.

Lancellotti P, Moura L, Pierard LA, Agricola E, Popescu BA, Tribouilloy C, et al. European Association of Echocardiography recommendations for the assessment of valvular regurgitation. Part 2: mitral and tricuspid regurgitation (native valve disease). Eur J Echocardiogr. 2010;11(4):307-332.

Marshall WA, Tanner JM. Variations in the pattern of pubetal changes in boys. Arch Dis Child 1970; 45:13.

Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969;44(235):291-303.

Morford, L. L., Inman-Wood, S. L., Gudelsky, G. A., Williams, M. T. and Vorhees, C. V. (2002), Impaired spatial and sequential learning in rats treated neonatally with d-fenfluramine. European Journal of Neuroscience, 16: 491–500. doi:10.1046/j.1460-9568.2002.02100.x

Ng Y, Conry J, Drummond R, Stolle J, Weinberg M for the OV-1012 Study Investigators. Randomized, phase III study results of clobazam in Lennox–Gastaut syndrome. Neurology 2011; 77:1473–1481.

Panayiotopoulos C. Epileptic encephalopathies in infancy and early childhood in which the epileptiform abnormalities may contribute to progressive dysfunction. In Panayiotopoulos C (Ed) The epilepsies: seizures, syndromes and management. Oxfordshire, UK: Bladon Medical Publishing, 2005:137–206.

Rabbit, P. (Ed.). (1997). /react-text Methodology of frontal and executive function react-text: 2931. East Sussex, UK: Psychology Press.

Sabaz, M., Cairns, D. R., Lawson, J. A., Nheu, N., Bleasel, A. F., & Bye, A. M. (2000). Validation of a new quality of life measure for children with epilepsy. Epilepsia, 41(6), 765–774.

Schoonjans A, Marchau F, Paelinck B, Gunning B, Verhoeven JS, Gammaitoni AR, Galer BS, Lagae L, Ceulemans B. Low-Dose Fenfluramine Provides Significant and Long-Term Seizure Reduction in Dravet Syndrome: Update and Follow-Up of the Prospective Study. American Epilepsy Society Annual Meeting 2017: Abstract 3.264.

Schoonjans A-S, Lagae L, Ceulemans B. Low-dose fenfluramine in the treatment of neurologic disorders: experience in Dravet syndrome. *Therapeutic Advances in Neurological Disorders*. 2015;8(6):328-338. doi:10.1177/1756285615607726.

Talarska, D. (2007). The usefulness of Quality of Life Childhood Epilepsy (QOLCE)


questionnaire in evaluating the quality of life of children with epilepsy. Advances in Medical Sciences, 52 Suppl 1, 191–193.

Webb RH, Gentles TL, Stirling JW, et al. Valvular regurgitation using portable echocardiography in a healthy student population: implications for rheumatic heart disease screening. J Am Soc Echocardiogr. 2015;28:981 988.

Westphal-Guitti C, Alonso NB, Migliorini RCVP et al., "Quality of life and burden in caregivers" of patients with epilepsy," The Journal of Neuroscience Nursing, vol. 39, no. 6, pp. 354–360, 2007.

Wheless JW, Clarke DF, Arzimanoglou A, et al. Treatment of pediatric epilepsy: European expert opinion, 2007. Epileptic Disord 2007;9:353–412.

de V deficit. rtical outpu

.d valvular heart dise.
.d of Medicine 1998, 65:
, 2020. Williams, M. T., Morford, L. L., McCrea, A. E., Wood, S. L., & Vorhees, C. V. (2002) Administration of d,l-fenfluramine to rats produces learning deficits in the Cincinnati water maze but not the Morris water maze: relationship to adrenal cortical output. Neurotoxicology and

Wong J, Reddy SS, Klein AL. Anorectic drugs and valvular heart disease: a biological and clinical perspective. Cleveland Clinical Journal of Medicine 1998; 65:35-41.


#### 14. APPENDICES

# APPENDIX 1 – LIST OF PROHIBITED CONCOMITANT MEDICATIONS

The below table lists examples of medications in the classes prohibited under the exclusion criteria defined in the protocol, but it is not an exhaustive list. Please consult the medical monitor in your region if a participant is on a medication that falls into any prohibited classifications but is not listed in the below table.

| ADHD Medications | | | (8) |
|---|---|---|---|
| Atomoxetine | A 1 / 1 11 1 | Methamphetamine 🔪 | Guanfacine |
| Methylphenidate | Amphetamine and derivates | Lisdexamfetamine ( | Bupropion |
| Dexmethylphenidate | Dextroamphetamine | Clonidine | |
| Anti-arrhythmics | Antibiotics | Anti-nausea | Anti-pyretic |
| Mexiletine | Linezolid | Metoclopramide | Phenacetin |
| Propafenone | 1 | Ondansetron | |
| Anticonvulsants | 7 | W: 10 | |
| Felbamate** | Retigabine/ezogabine | THC and derivatives | |
| Epidiolex | Cannabidiol products | ( 1,0 | |
| Antidepressants (SSRIs, SI | | | |
| Amitriptyline | Clomipramine | Fluvoxamine | Paroxetine |
| Bupropion | Desipramine | Imipramine | Sertraline |
| Buspirone | Duloxetine | Nefazodone | Trazodone |
| Citalopram | Fluoxetine | Nortriptyline | Vortioxetine |
| Antihistamines | 70 70 75 | | |
| Astemizole | Hydroxyzine | Chlorphenamine | |
| Cyproheptadine | | Diphenhydramine | |
| Anti-migraine | 5 01 | | |
| Almotriptan | Eletriptan | Naratriptan | Sumatriptan |
| Cafergot | Ergotamine tartrate | Rizatriptan | Zolmitriptan |
| Antipsychotics/Neuroleptic | es (serotonin agonists/ antagonists, nor | adrenergic agonists/an | tagonists) |
| Amisulpride | Guanfacine | Paliperidone | Risperidone |
| Amphetamine | Haloperidol | Perospirone | Sulpiride |
| Aripiprazole | Levomepromazine | Perphenazine | Ziprasidone |
| Asenapine | Lurasidone | Promethazine | Zuclopenthixol |
| Clozapine | Methylphenidate | Propanolol | |
| Clonidine | Olanzapine | Quetiapine | |
| ~ | | | Cough |
| Anti-viral | Beta Blocker | Chemotherapy | Suppressant |
| Interferon | Alprenolol | Dasatinib | Dextromethorphan |
| Ritonavir | Bufuralol | | |
| Telaprevir | | | |
| Centrally-acting anorectic | agents | | |
| 1 | | Naltrexone- | Phentermine- |
| Lorcaserin | Phentermine | bupropion | topiramate |
| Diethylpropion | Benzphetamine | Phendimetrazine | |
| Decongestants (allowed for | short-term use only) | Statins | |
| Phenylpropanolamine | | Cerivastatin | |
| Ergot Alkaloids, their deri | vatives, and Antiparkinson agents | | |


| Pergolide | Cabergoline | Ergotamine Tartrate | |
|---|---|---|---|
| Monoamine-oxidase inhib | itors | | |
| Isocarboxazid | Selegiline | Tranylcypromine | Phenelzine |
| Opioids | | | |
| Alfentanil | Levacetylmethadol (LAAM) | Meperidine | Oxycodone |
| Codeine | Fentanyl | Methadone | Tramadol |

an felbamate for a valory tests, the dose ain constant throughout the dose ain constant throughout the deliberation and arrived the deliberation and the deliberation arrived th






APPENDIX 5 – TANNER STAGING


Sparra, plgmonthal, long, straight, marrly along labra and at

Darker, coatest, quities

Because the onset and progression of puberty are so variable, Tanner has proposed a scale, Because the onset and progression of pubertal changes (Fig. 9and girls are rated for breast development and pubic hair growth The Tanner Stages publichadi growth,

Pubic hair growth in feprales is staged as follows (Fig 9-24, B):

- Stage I (Preadolespeat) Velfach air develops over the pubes in a manner not greater than that over eris no sekus the anterior wall. They
- hair, which is straight or only slightly ourled, appears. These o quantitate on black and white photographs, particularly when pictures are of hairs are seen mainly along tige Jabia. Stage II - Sparse, long, prigmented, do
- sars. The hair has now spread Stage III - Considerably darker, coerser, and curies sexual hair sparsely over the junction of the puber
- Stage IV The hair distribution is adult in 1998 but decreased in total quantity. There is no spread to Stage V - Hair is adult in quantity and type and appears to have an inverse triginale of the dassically feminine type. There is spread to the medial surface of the thigh but not above the base of the the medial surface of the thighs.

The stages in male pubic hair development are as follows Fig. 9-24, B):

inverse triangle

 Stage I (Preadolescent) - Vellos hair appears over the pubes with a eggree of devalopment similar to that over the abdorninal wall. There is no androgen-sensitive pubic hair.

Adultin quantity and type with spread to medial thight

- Stage II There is sparse development of long pigmented downy hair, which, only slightlycurled or straight. The hair is seen chiefly at the base of penis. This stage may be difficult be evaluated. photograph, especially if the subject has fair hair.
- Stage III The public hair is considerably darker, coarser, and curlier. The distributions your spread over the junction of the pubes, and at this point that hair may be recognized easily on black and white photographs
- Stage IV The hair distribution is now adult in type but still is considerably less that seen in adults. Thereas go spread to the medial surface of the thighs

· Stage V - Hair distribution is adult in quantity and type and is described in the inverse triangle. Then can be present to the medial surface of the thighs


Amed on a black and vinne.

Stage III - Enther growth of the penis has occur.

Stage III - Enther growth of the penis has occur.

In length, although with some increase in dicumference. Inne.

Stage IV - The penis is significantly enlarged in length and dicumference, lawns in significantly enlarged and there is distinct dankening of the scrotal skin. This is digitally to every continue to enlarge, and there is distinct dankening of the scrotal skin. This is digitally to every continue to enlarge, and there is distinct dankening of the scrotal skin. This is digitally to every continue to enlarge, and there is distinct dankening of the scrotal skin. This is digitally to every continue to enlarge, and there is distinct dankening of the scrotal skin. The scrotal skin. This is digitally and discussed in the scrotal skin. The scrotal skin. The scrotal skin. The scrotal skin. The scrotal skin. This is digitally and discussed in the scrotal skin. The scrotal skin. The scrotal skin. The scrotal skin. This is digitally scrotal skin. The scrotal skin. N Further development Conthued Briengement epided pue ece ent budding 0 0 State I (Preadolescent) - Only the papilla is elevated above the feed of the chest wall. Stage IV - The areolae and papiliae elevate above the level Stage II - There is enlargement of the scrotum and tests and a change in the texture of the scrotal skin. The scrotal the level of the chest wall.

the level of the chest wall.

Stage Ir. (Beest Budding) - Elevation of the breasts and

Stage Ir. (Beest as small mounds along with some have a size and proportion similar to those seen in early of the breasts and form secondary mounds with further · Stage (I) The breaks and areolae continue to enlarge, The stages for male genitalia development although they show he separation of contour. Stage I (Preadolescent)- The testes, scrotal sac development of the operall breath issue. breasts as the result of the regession of the papillae may extend slightly above the Stage V - Mature female breasts have follows: (Fig. 9-24, A): childhood.


### APPENDIX 6 – QOLCE QUALITY OF LIFE

- . day to day functioning in various life areas. If
  ...ing your child's day to day functioning. Your answers
  ... not to participate it will not affect the care you or your child receive.

  5. Please answer the questions by marking the appropriate box, like this...

  6. Certain questions may look alike, but each one is different. Some questions and allout problems your child may not have, but it's important for us to know this infurnation too. Please answer each question to the best of your knowledge. Remember to answer and unless instructed otherwise.

  5. There are no right or wrong answers. If you are unguire how to affine a question, please give the best answer you can and make a commembration.

  All comments will be read, so please feel free tojmake as night, as you wist.

  You may not be abile to answeregoing questions afroit difficult to tell how your child fashing about they feelings. In


2

| | The following question | | | | | d.Elde | | |
|---|---|---|---|---|---|---|---|---|
| | 3.1. In his/her daily act | tivities during | the past 4 | weeks, how ofto | en has your o | :hild: | | |
| | | Very Often | Fairly<br>Often | Sometimes | Almost<br>Never | Never | Not<br>Applicable | × |
| | a, needed more<br>supervision than<br>other children his/her<br>age? | | | | | | Not Applicable | 90 |
| | b. needed special<br>precautions (ie<br>wearing a helmet)? | | | | | | | I S |
| | c. played freely in the<br>house like other<br>children his/her age? | | | | | | SIX | 5 |
| | d. played freely<br>outside the house like<br>other children his/her<br>age? | | | | 1 0 | 13 | (S)(O) | |
| | e. gone swimming?<br>(ie. swam<br>independently) | | | OX. | N. | | 9. 0 | |
| | f. participated in<br>sports activities<br>(other than<br>swimming)? | | 0 | CUPI | 100 | 0 | | |
| | g. stayed out<br>overnight (with<br>friends or family)? | 296 | *C | | Oi | | | |
| | h. played with friends<br>away from you or<br>your home | 50 | 00 | tien. | | | | |
| | i. gone to parties<br>without you or<br>without supervision | 2 | 90 | | | | | |
| | | 90 | | | | | | |
| | Callina | | | | | | | |
| en | esilo. | | | | | | | |
| is document | SII. | | | | | | | |
| 90, 01 | | | | | | | | |
| 113 | | | | | | | | |


3

| 3.2. During the past 4 weeks how much of the time do you think your child: All of the some of A listle of the time the time the time the time the time the time the time. Applicable a felt timed be felt energetic | 3.2. During the past 4 wee | ks how much of th | e time do you | think your c | hild: | | |
|---|---|---|---|---|---|---|---|
| a. felt tired b. felt energetic 3.3 is there anything else you would like to tell us about your child's activities? COPY ANY TRAINER TO BE AND | | All of the | Most of the time | Some of<br>the time | A little of<br>the time | None of<br>the time | Not<br>Applicable |
| 3.3 Is there anything else you would like to tell us about your child's activities? OPA the anything else you would like to tell us about your child's activities? | a, felt tired | | | | | | |
| 3.3 Is there anything else you would like to tell us about your child's activities? ORAL ANY MAINTAIN CALLINGS OF VARIABLE CORRECTIONS OF VARIABLE CALLINGS | b. felt energetic | | | | | | |
| 3.3 Is there anything else you would like to tell us about your child's activities? OR A Land White Hill College of the Colle | | | | | | | 0 |
| document cannot be used any extensions of variations to | 3.3 Is there anything else y | you would like to t | ell us about yo | ur child's ac | tivities? | | 0 |
| Accument cannot be used any extensions of variations to | | | | | | | |
| document cannot be used any extensions of variations and any extensions of variation and any extensions. | | | | | | 7/2 | 3, 11 |
| document cannot be used any extensions of variation. | | | | | | 0, | 5 |
| document cannot be used any extensions of variation and any extension and extension | | | | 4 | . < | | <i>3</i> / · |
| document cannot be used any extensions of value and any extension of value and any extensions of value and any extension of value and any extensions of value and any exte | | | ~ | 1 | 1 | : 0) | • |
| document cannot be used and any extensions of the document cannot be used to supplication and any extension of the document cannot be used to supplication and the document cannot be used | | | $\sim$ | | 9 | | |
| document cannot be used any extensions of | | | 9 | | " 1, | | |
| document cannot be used any extensions and any extension and extension and exten | | <i>C</i> | \ | 20 | 0 | | |
| document cannot be used any and any application and application and applic | | , 10 | 9,, ' | ~ C | | | |
| document camot be used and and and and alocument camot be used to the list of | | SV. | 5. | ,0' | | | |
| document cannot be used any extent | | ) | $\sim$ | | | | |
| 90chuseur caulou and aux exc | X | 9 | ×O, | | | | |
| Aocument cannot be land any | | S | + | | | | |
| document cation and and and and all and | | 7, 1 6 | ) | | | | |
| Aociment cannot and a | 100 | 303 | | | | | |
| Gocument canno aino | o' ' A | .0. | | | | | |
| 40clinent califor a | | <i>y</i> | | | | | |
| 40CIMent Certion | 2 | | | | | | |
| 90crius blication | * 00 .: 01, | | | | | | |
| 40c11Me dibblice | | | | | | | |
| 90crill sibbi. | 100 | | | | | | |
| 900, 36, | chi, coi, | | | | | | |
| | 100, 36, | | | | | | |
| | 0, | | | | | | |
| | ) | | | | | | |


| SECTION 4: WELL-BEING Below is a list that describes how your child might feel in general. 4.1. During the next 4 weeks, how much of the time do you think your child All of the Most of the Some of A little of time the time the time the time. a. felt down or depressed? b. felt calm? c. felt helpless in situations? d. felt happy? e. wished she was dead? f. felt in centrol? g. felt tense and anxious? h. felt frustrated? i. felt overwhelmed by events? j. worried a lot? k. felt confident? l. felt excited or interested in something? m. felt pleased about collecting a something? m. felt pleased about collecting a something? n. got easily embarrassed? o. felt different or singless out? q. felt who was fiely pool at the singless out? q. felt who was fiely pool at the singless out. | | s a list that describes he<br>ring the past 4 weeks, b | | | | child | | |
|---|---|---|---|---|---|---|---|---|
| I. felt excited or interested in something? m. felt pleased about activing something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | | | All of the | Most of the | Some of | A little of<br>the time | None of<br>the time | Not<br>applicable |
| I. felt excited or interested in something? m. felt pleased about activing something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | a. felt d | own or depressed? | | | | | | |
| I. felt excited or interested in something? m. felt pleased about activing something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | b. felt c | alm? | | | | | | |
| I. felt excited or interested in something? m. felt pleased about active ving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | c. felt h | elpless in situations? | | | | | | Silver de |
| I. felt excited or interested in something? m. felt pleased about selfieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | d. felt h | арру? | | | | | | Spirito |
| I. felt excited or interested in something? m. felt pleased about selfieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody indepstood him/her? | ę, wish | ed s/he was dead? | | | | | | S |
| I. felt excited or interested in something? m. felt pleased about selfieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody inderstood him/her? | f. felt is | n control? | | | | | Ca | 000 |
| I. felt excited or interested in something? m. felt pleased about achieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | g. felt t | ense and anxious? | | | P | | | |
| I. felt excited or interested in something? m. felt pleased about selfieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody inderstood him/her? | h. felt t | frustrated? | | | | Na. | Ø, | |
| I. felt excited or interested in something? m. felt pleased about softieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | i, felt o | verwhelmed by events? | | CO. | | | 0 | |
| I. felt excited or interested in something? m. felt pleased about softieving something? n. got easily embarrassed? o. felt different or singled out? p. felt nobody understood him/her? | j. wom | ied a lot? | | 9 | O. | 0 | | |
| o. felt different or singled out? p. felt nobody understood him/her? | k, felt | confident? | | 0/6 | DC | 0 [ | | |
| o. felt different or singled out? p. felt nobody understood him/her? | | | SY | 5 | 0 | | | |
| o. felt different or singled out? p. felt nobody bidentood him/her? | | | 0 | | | | | |
| p. felt nobody understood | n. got | easily embarrassed? | | +N | | | | |
| him/her? | | different or singled | | ) [ | | | | |
| q. fels college? | him/h | er? | J. D. | | | | | |
| inglining? s. felt no operated? | q, felt | scalucit? | | | | | | |
| s. felt 10 Opercared? | r felt | s/he was not good at | | | | | | |
| | s. felt | no ope-cared? | | | | | | |


This document cannot be used any extensions or validations the real to support any national delivers the real to support and the real to support any national delivers the real to support any national delivers the real to support any national delivers the real to support any national delivers the real to support and the real to support any national delivers the real to support and the real to support any national delivers the real to support any national delivers the real to support any national delivers the real to support any national delivers the real to support and the real to support any national delivers the real to support any national delivers the real to support any national delivers the real to support any national delivers the real to support and the real to s


6

| | 5.1. Compared to other | | her own ag | g, how often du | ring the past | 4 weeks has | your | |
|---|---|---|---|---|---|---|---|---|
| | child | | | | | | Non | |
| | | Very Often | Fairly<br>Often | Sometimes | Almost | Never | Applicable | |
| | a. had difficulty<br>attending to an activity? | | | | | | | (D) |
| | <ul> <li>b. had difficulty<br/>reasoning or solving<br/>problems?</li> </ul> | | | | | | Not Applicable | , e |
| | c. had difficulty making<br>plans or decisions? | | | | | | 21/1 | |
| | d. had difficulty keeping<br>track of conversations? | | | | | 75 | O | |
| | e. had trouble<br>concentrating on a task? | | | 8 | | 70 | Sp. | |
| | f. had difficulty<br>concentrating on<br>reading? | | | 08 | V DO. | TO. | | |
| | g. had difficulty doing<br>one thing at a time? | | F | .00 | 00 | | | |
| | h. reacted slowly to<br>things being said &<br>done? | B | · 0 | 301 | | | | |
| | i. completed activities<br>that needed organising<br>& planning? | | X | SUP | | | | |
| | j. found it hard<br>remembering things? | 15 | ET. | | | | | |
| | k. had trouble<br>remembering names of<br>people? | | 1 0 | | | | | |
| | 1. had probble<br>remembering where the<br>put thirtys? | 0 0 | | | | | | |
| * | remembering things | | | | | | | |
| | 5.1. continued: Compa | red to other ch | ildren his/l | er own age, ho | v often duri | ng the past 4 | weeks | |
| Illia | | | | | | | | |
| is document | | | | | | | | |
| . 6 | | | | | | | | |


| | | | 7: | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Very Often | Fairly<br>Often | Sometimes | Almost | Never | Not<br>Applicable | |
| | n. had trouble<br>remembering things s/he<br>read hours or days<br>before? | | | | | | | 317 |
| | o. planned to do<br>something then forgot? | | | | | | | _ |
| | p. had trouble finding<br>the correct words? | | | | | | | 2, |
| | q. had trouble<br>understanding or<br>following what others<br>were saying? | | | | | | Not Applicable | |
| | r. had trouble<br>understanding<br>directions? | | | | | 700 | illo 19 | |
| | s. had difficulty<br>following simple<br>instructions? | | | 2 | | 10 | Silv | |
| | t. had difficulty<br>following complex<br>instructions? | | | O <sub>E</sub> | X P | 10, | | |
| | u. had trouble<br>understanding what s/he<br>read? | | 0 | 100 | 50 | | | |
| | v. had trouble writing? | 18 | | 10 | | | | |
| | w. had trouble talking | Cec | | SUS | | | | |
| This document | 5.2. Is there anything elspeech? | g all | | anout you ve | | | | |
| izis 90chlusibli | Co | | | | | | | |


| | 6.1. During the past 4 we | eks, how often | has your cl | aild's epilepsy | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Very Often | Fairly<br>Often | Sometimes | Almost<br>Never | Never | Not<br>Applicable | **/0 |
| | a. limited his/her social<br>activities (visiting<br>friends, close relatives,<br>or neighbours? | | | | | | | autho a |
| | b. helped him/her<br>to make friends? | | | | | | | ) . © |
| | c. affected his/her social<br>interactions at school or<br>work? | | | | | | VSEII! | Nel |
| | d. improved his/her<br>friendships &<br>relationships with<br>others? | | | | | 40 | HORS | |
| | <ul> <li>e. limited his/her leisure<br/>activities (hobbies or<br/>interests)?</li> </ul> | | | PEN | To. | | 9,0 | |
| | f, isolated him/her from others? | | 6 | | | 78 | | |
| | g. improved his/her<br>relations with family<br>members? | | | | 50. | | | |
| | h. made it difficult for<br>him/her to keep friends? | 160 | (O | 50 | | | | |
| | i, frightened other people | 600 | 4 | 30.71 | | | | |
| | 6.2. During the past 4 v | vecks, how limi | ted are you<br>y or epileps | r child's social<br>y-related probl | activities con<br>ems? | npared with | others | |
| | | | ned . | Yes,<br>but<br>rarely | No,<br>not<br>limited | | | |
| his document | Cation | | | | | | | |
| 90cn1,366 | * | | | | | | | |
| :19 | | | | | | | | |


| | | | | 9 | | | |
|---|---|---|---|---|---|---|---|
| | 6.3. <u>During the friends?</u> | e past 4 weeks, h | ow often has you | r child freely disc | ussed his/her epilepsy with | | ,;\C |
| | ☐<br>Very often | Fairly often | Sometimes | Almost never | Not applicable | | :121 |
| | 6.4. During th | ne past 4 weeks, 1 | ow often has you | ır child freely disc | ussed his/her epilepsy with | iff | ), |
| | ☐<br>Very often | Fairly often | Sometimes | Almost never | Not applicable | 30 | <b>X</b> • |
| | 6.5. Is there a | anything else you | would like to tell | us about your chi | id's social activities? | ons there | |
| | | R | BLICA | Suppositions | ons | | |
| This document | califo | or and | | | | | |
| Khis | | | | | | | |


10

| Very Often Fairly Often Never Not Applicable | 7.1. Compared to other child<br>the following statements des | fren his/her ow<br>cribe your chil | n age, how<br>d? | often during th | he past 4 wee | ks do each o | | |
|---|---|---|---|---|---|---|---|---|
| h. swore in public i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for seelf a. did not warry about what others throught People along with other safeldren | | Very Often | | Sometimes | Almost<br>Never | Never | Not<br>Applicable | |
| h. swore in public i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self n. did provery about what | do things for him/her that<br>s/he was able to do | | | | | | | 0 |
| h. swore in public i. joined in activities with other children j. feared unfamiliar places, situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self | b. asked for reassurance | | | | | | 4 | ~ C |
| h. swore in public i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self n. did preswurry about what | (said or did something out | | | | | | Silter Co | 7/1. |
| h. swore in public i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others i. was obedient m. set high standards for self n. did preswury about what | | | | | | Q | ifo, | |
| h. swore in public i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self | e, did not give up easily | | | 0 | 4 | | On | |
| h. swore in public i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self n. did personary about yaba | f. angered easily | | | <b>О</b> р. | XI | SE | | |
| i. joined in activities with other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self n. did personary about when | g, hit or attacked people | | | ) LC | | П | | |
| other children j. feared unfamiliar places situations or people k. preferred his/her own company instead of seeking out others l. was obedient m. set high standards for self n. did personery about when | h. swore in public | | Uh | YO, | d | | | |
| situations or people k. preferred his/her own company instead of seeking out others 1. was obedient m. set high standards for self n. did perswarty about yaba | | 3 | □C | | | | | |
| company instead of seeking out others I. was obedient m. set high standards for self n. did provery about when | | J <sub>0</sub> | ×Q | (6) | | | | |
| m. set high standards for self a. did presswery about salar a. | company instead of seeking | 500 | 4 | 0.0 | | | | |
| a. did perwary about what | I. was obedient | | | | | | | |
| | m. set high standards for self | Sign | | | | | | |
| p. wishershipe was someone | n. did not wary about what<br>others thought | 0 | | | | | | |
| p. wished the was someone | orget along with other | | | | | | | |
| | p. wished the was someone or somewhere else | | | | | | | |


| | | | - 11 | | | | | | ( |
|---|---|---|---|---|---|---|---|---|---|
| | 7.1 continued: Compared to<br>do each of the following state | other childres<br>ements describ | n his/her ov<br>e your child | n age, how ofte | en during the | past 4 week | 15 | | dio |
| | | Very Often | Fairly<br>Often | Sometimes | Almost<br>Never | Never | Not<br>Applicable | | il.o. |
| | q. acted without thinking | | | | | | | ~ | O. |
| | r, demanded a lot of attention | | | | | | | Silli | ٨. |
| | s, was decisive | | | | | | | 0,0 | Э, |
| | t, was independent | | | | | | | | |
| | u. preferred routines or<br>disliked changes | | | | | | The. | HILL | |
| | v, did things just to prove<br>s/he could | | | | | | | 12 | |
| | w. preferred the company of adults | | | | | | : Oll | | |
| | 7.2. Is there anything else y | ou would like | to tell us ab | out your child' | behaviour? | 12 | | | |
| This document | cation and | JBI | | ensile | 3NS | | | | |


Jour child's quality of life been?

Very Good Good Fair Poor

| Door | Door Child's quality of life been? | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | Door | e a copy of any detachable sheet for all he detachable she


This appendix


| D | Α | | D | Α | | |
|---|---|---|---|---|---|---|
| | | I feel tense or 'wound up': | | | I feel as if I am slowed down: | |
| | 3 | Most of the time | 3 | | Nearly all the time | |
| | 2 | A lot of the time | 2 | | Very often | .4 |
| | 1 | From time to time, occasionally | 1 | | Sometimes | . 0 |
| | 0 | Not at all | 0 | | Not at all | |
| | | | | | | .10 |
| | | I still enjoy the things I used to enjoy: | | | I get a sort of frightened feeling like 'butterflies' in the stomach: | Nithori Zatio |
| 0 | | Definitely as much | | 0 | Not at all | 1100 |
| 1 | | Not quite so much | | 1 | Occasionally | |
| 2 | | Only a little | | 2 | Quite Often | × × · |
| 3 | | Hardly at all | | 3 | Very Often | CO. |
| | | | | | | ~(0 |
| | | I get a sort of frightened feeling as if something awful is about to | | | I have lost interest in my appearance: | O' |
| - | 3 | happen: Very definitely and quite badly | 3 | | Definitely | |
| | 2 | Yes, but not too badly | 2 | | I don't take as much care as I should | |
| | 1 | A little, but it doesn't worry me | 1 | -1 | I may not take quite as much care | |
| | 0 | Not at all | 0 | 2 | I take just as much care as ever | |
| | 0 | Not at all | O | × · | Trake just as much care as ever | |
| | | I can laugh and see the funny side of things: | | | I feel restless as I have to be on the move: | |
| 0 | - | As much as I always could | | 3 | Very much indeed | |
| 1 | - | Not quite so much now | | 2 | Quite a lot | |
| 2 | | Definitely not so much now | 5 | 1. | Not very much | |
| 3 | | Not at all | | 6 | Not at all | |
| | 4 | Worrying thoughts go through my | ~ | 13 | I look forward with enjoyment to | |
| | | mind: | 9 | | things: | |
| | 3 | A great deal of the time | 0 | | As much as I ever did | |
| | 2 | A lot of the time | 1 | | Rather less than I used to | |
| | 1 | From time to time, but not too often | 2 | | Definitely less than I used to | |
| | 0 | Only occasionally | 3 | | Hardly at all | |
| | | -0, 9 | | | | |
| | | I feel cheerful: | | | I get sudden feelings of panic: | |
| 3 | 0 | Not at all | | 3 | Very often indeed | |
| 2 | G | Not often | | 2 | Quite often | |
| Ple | | Sometimes | | 1 | Not very often | |
| 0 | | Most of the time | | 0 | Not at all | |
| 1 | ic | | | | | |
| - | 3/1, | I can sit at ease and feel relaxed: | | | I can enjoy a good book or radio or TV | |
| Q. | | | | | program: | |
| '0' | 0 | Definitely | 0 | | Often | |
| | 1 | Usually | 1 | | Sometimes | |
| | 2 | Not Often | 2 | | Not often | |
| | | T. Control of the Con | | | | |

| 0 | |
|--------|-----------------------|
| Scorin | |
| Totals | score: Depression (D) |
| 0-7 | = Normal |


This document cannot be used any extensions or validations the read.


### APPENDIX 8 – ZARIT CAREGIVER BURDEN INVENTORY

## The Zarit Burden Interview

| The Zarit Burden In | terview | | | |
|---|---|---|---|---|
| 0: NEVER | | | | no althoriz |
| 1: RARELY | | | | NY K. |
| 2: SOMETIMES | | | | 0, |
| 3: QUITE FREQUENTLY | | | 11 | |
| 4: NEARLY ALWAYS | | 7 | Sy, | KVE |
| Please circle the response the best descr | ibes how you feel. | OI, | -0 | 5 |
| 0 | 1 | · i | <u>(0,</u> | |
| Question | 27 200 | Scor | е | |
| 1 Do you feel that your relative asks for more relative | in he/she needs? | 0 1 2 | 3 4 | |
| Do you feel that because of the time you spend with you don't have enough time for yourself? | your relative that | 0 1 2 | 3 4 | 8 |
| 3 Do you feel stressed between caring for your relative meet other responsibilities for your family or work? | e and trying to | 0 1 2 | 3 4 | A. |
| 4 Do you feel embarrassed over your relative's behave | (iour? | 0 1 2 | 3 4 | ā |
| 5 Do you feel angry when you are around your relative | e? ( | 0 1 2 | 3 4 | B. |
| 6 Do you feel that your relative currently affects our re<br>other family members of mends in a negative way? | elationships with | 0 1 2 | 3 4 | 8 |
| 7 Are you afraid what the future holds for your relative | 9? ( | 0 1 2 | 3 4 | 6 |
| 8 Do you feel your relative is dependent on you? | C | 0 1 2 | 3 4 | a l |
| 9 Do you fee strained when you are around your rela | tive? | 0 1 2 | 3 4 | |
| 10 Do you feel your health has suffered because of you with your relative? | ur involvement ( | 0 1 2 | 3 4 | ă |
| Do you feel that you don't have as much privacy as because of your relative? | you would like | 0 1 2 | 3 4 | A. |
| Do you feel that you don't have as much privacy as because of your relative? 12 On you feel that your social life has suffered because for your relative? | se you are caring | 0 1 2 | 3 4 | 8 |


| Do you feel uncomfortable about having friends over because of your relative? Do you feel that your relative seems to expect you to take care of him/her as if you were the only one he/she could depend on? Do you feel that you don't have enough money to take care of your relative in addition to the rest of your expenses? Do you feel that you will be unable to take care of your relative much longer? Do you feel you have lost control of your life since your relative's illness? | 0 | 1 1 | 2 2 | 3 | 4 |
|---|---|---|---|---|---|
| him/her as if you were the only one he/she could depend on? Do you feel that you don't have enough money to take care of your relative in addition to the rest of your expenses? Do you feel that you will be unable to take care of your relative much longer? Do you feel you have lost control of your life since your relative's | 0 | 1 | 2 | 3 | 4 |
| relative in addition to the rest of your expenses? Do you feel that you will be unable to take care of your relative much longer? Do you feel you have lost control of your life since your relative's | | 1 | 2 | -3 | |
| longer? Do you feel you have lost control of your life since your relative's | 0 | 9 | | S. | 4 |
| | | 14 | 2 | 3 | \$4 |
| | 0 | t | 2 | 3 | 4 |
| Do you wish you could leave the care of your relative to someone else? | 2/8 | 1 | 2 | 3 | 4 |
| Do you feel uncertain about what to do about your relative? | 0 | 1 | 2 | 3 | 4 |
| Do you feel you should be doing more for your relative? | 0 | 1 | 2 | 3 | 4 |
| Do you feel you could do a better lob in caring for your relative? | 0 | 1 | 2 | 3 | 4 |
| Overall, how burdened do you feel in caring for your relative? | 0 | 1 | 2 | 3 | 4 |
| rpretation of Score: 21 little or no burden 40 mild to moderate burden 60 moderate to severe burden | 0 | 1 | 2 | 3 | |

∠1 little or no burd. ∠1 - 40 mild to moderate. 41 - 60 moderate to seve. 61 - 88 severe burden


## APPENDIX 9 – MAXIMUM ALLOWABLE BLOOD DRAW VOLUMES




### APPENDIX 10 – STUDY CONDUCT DURING COVID-19

In March 2020, the World Health Organization declared a global pandemic related to an illness caused by a novel coronavirus known as COVID-19. As a result, public health initiatives, such as laws, regulations and policies were enacted at country and institutional levels to protect the health of the general public. These initiatives and policies have affected the ability of study sites to conduct the trial per protocol and the ability of the sponsor and/or delegate to conduct trial oversight and monitoring visits. In an effort to support the rights, safety and welfare of subjects and ensure as little impact on the integrity of the research as possible the following alternative processes have been implemented due to restrictions related to COVID-19. Though every attempt should be made to conduct study visits per protocol, any implementation of alternative processes should be properly documented. If there are no impacts or accommodations for COVID-19 at a study site, these allowances must not be followed.

### 1. Allowance of Delays to In-person Study Visits

If sites are unable to conduct study visits, or subjects are unable to travel to the study site due to COVID-19 circumstances, an in-person visit may be delayed up to 6 weeks from the protocol-defined visit due date. Data will need to be entered per normal procedures in the EDC, with a description indicating COVID-19 as the cause for delay in response to queries. If a subject is unable to travel to the study site within this expanded 6-week window, a telephone or video telemedicine visit should be attempted, as described below. If a telephone or video telemedicine visit cannot be conducted in the 6-week window, the visit should be considered missed and the next scheduled visit conducted.

### 2. Allowance of Remote Telemedicine/Telephone/Video Visits:

Visits 1-5 should be conducted in person. For Visits 6, 8, 10, 15-21, remote visits via telephone or video are acceptable when subjects are unable to travel to the site for in-person visits due to COVID-19 circumstances. The following information should be collected and recorded in the source documentation and in the EDC where applicable. Log pages (e.g. AEs, concomitant medication changes) will be entered normally as they are not associated with specific visits; assessment forms located within a particular visit page will also be entered normally, however, queries will be fired to capture specific information explaining the basis for missing or alternatively collected (ie. remote) data. Detailed instruction for EDC entry may be found in the CRF Completion Guidelines (CCGs).

- Date and time of the telephone/video visit
- Any changes in health status
- AEs/SAE assessment
- Concomitant medication query
- Review seizure and medication diary with parent/caregiver for compliance and any abnormalities in seizure activity
- Scales and Questionnaires, when applicable and if feasible
  - C-SSRS
  - CGI-I (by Investigator and Parent/Caregiver)
  - BRIEF
  - Tanner Staging
  - o QOLCE
  - o Zarit Caregiver Burden
  - HADS


### 3. End-of-Study/Early Termination (EOS/ET) and Follow-up Visits:

Cardiac follow-up visits (Visits 14, 24, or 25) must be conducted in-person.

### EOS/ET for subjects tapering off ZX008:

For the EOS/ET visit (Visit 12 or 22) and Post-Dosing Follow-up visit (Visit 13 or 23), every attempt should be made to conduct these visits in-person. For subjects tapering off study-drug that are unable to come to the study site, the EOS/ET and Post-Dosing Follow-up visits may be conducted via telephone or video. However, subjects should return to the study site in person, as soon as feasible to conduct any safety assessments that were unable to be evaluated remotely. If an in-person visit cannot be scheduled within 6 months of the EOS/ET and/or Post-Dosing Follow-up visit windows to conduct the required safety assessments, these assessments will be considered as missed.

### EOS/ET for subjects transitioning to another Extension Study:

For subjects transitioning into another ZX008 extension study that are unable to attend the EOS/ET visit due to restrictions to traveling to the study site, delays in the start-up of the extension study, or other COVID-related delays, the EOS/ET visit may be delayed until an in-person visit is conducted. Therefore, subjects may remain on study for longer than the planned duration of participation. If the delay is over 6 weeks, medical monitor review and approval is required. If approval to extend beyond 6 weeks is granted, telephone or video visits should be conducted at least every 12 weeks until the inperson EOS/ET transitional visit to the other extension study is performed. The telephone or video visits will collect the following data, at minimum:

- Date and time of the telephone/video visit
- Any changes in health status
- AEs/SAE assessment
- Concomitant medication query
- Review seizure and medication diary with parent/caregiver for compliance and any abnormalities in seizure activity

# 4. Allowance of delays to ECHO, ECG, Chest X-Ray, EEG and clinical lab assessments when inperson study visits are missed or delayed

If it is not possible to obtain the above assessments as described below, a documented risk/benefit discussion with the medical monitor is required to determine a course of action, which may include approval to delay further for a pre-specified duration, subject withdrawal, or other actions. The risk/benefit analysis will take into account AEs, previous assessment findings, duration of delay, clinical improvement while on study drug (seizure and non-seizure outcomes), and region-specific risk of attending in-person visits to complete the assessments.

### Doppler ECHO:

If subjects are unable to travel to the study site due to COVID-19 circumstances, ECHOs may be delayed up to an additional 3 months from the protocol-designated ECHO due date (for a total of 6 months from the time of the last ECHO) for subjects that exhibited the following on their previous, most recent ECHO: absent aortic regurgitation, absent or trace mitral regurgitation, and PASP <30 mmHg.

All subjects with regurgitation  $\geq$  trace aortic regurgitation,  $\geq$ mild mitral regurgitation, or PASP  $\geq$ 30 mmHg may have ECHO delayed from the protocol-designated ECHO due date by up to 6 weeks only.


In those cases where an ECHO cannot be performed in the specified time period at the study-authorized facility by a certified sonographer, the Sponsor may approve administration of the ECHO at an alternative facility to minimize need for travel. If the ECHO cannot be performed, a benefit risk/benefit analysis must be conducted as described above.

If a delayed ECHO was conducted within 30 days of a scheduled Cardiac Follow-up Visit and there were no findings meeting Level 2 criteria (see Protocol Table 17), the Cardiac Follow-up Visit may be cancelled. If Level 2 or greater findings were observed, then the Cardiac Follow-up Visit should be rescheduled 3 months from the date of the delayed ECHO.

### ECG, Chest X-ray and EEG:

If clinically indicated and where applicable, delays in these assessments may be implemented based on the investigators' clinical discretion, weighing the risk/benefit of the clinical necessity of the assessment versus the risk of an in-person visit. All decisions should be documented appropriately in the source documentation. If not conducted at the study site, ECG, chest X-ray and EEG can be performed at any qualified local facility with results sent to the Principal Investigator for safety overread and documentation.

If the ECG (or in the case of certain country-specific regulations: Chest X-ray or EEG) was conducted within 30 days of a scheduled Cardiac Follow-up Visit, these assessments do not need to be repeated at the Cardiac Follow-up Visit provided there were no significant findings that require additional follow-up.

### Clinical Laboratory Assessments:

If clinically indicated and where applicable, delays in these assessments may be implemented based on the investigators' clinical discretion, weighing the risk/benefit of the clinical necessity of the assessment versus the risk of an in-person visit. All decisions should be documented appropriately in the source documentation. If not conducted at the study site, clinical laboratory assessments can be performed at any qualified local facility with results sent to the Principal Investigator for safety overread and documentation.

### 5. Alternative Dispensation for Study Drug

Shipments of investigational product may be sent by courier from site pharmacy to the subject's home via Sponsor-approved processes if the subject cannot or will not attend the dispensation visit(s). This shipment of drug should be arranged for patients who are due in the clinic for a drug dispensation visit. Other alternative dispensation, such as curbside pickup, may be implemented provided they are approved by the Sponsor and appropriate safeguards are taken to ensure compliance with existing regulatory requirements for maintaining investigational product accountability. Detailed instructions for drug handling, storage, accountability, etc. are described in the Pharmacy Manual.


### APPENDIX 11 - SUMMARY OF PROTOCOL AMENDMENT 4.0

### **Rationale for Protocol Amendment 4.0**

The protocol is being amended to simplify the visit schedule and reduce burden on the remaining participating subjects and their caregivers in Japan. The reduced <u>in-clinic</u> visit schedule (in-clinic visits every six months) will provide longitudinal safety data in an open-label setting which will inform the ongoing monitoring of Safety and Efficacy for Lennox-Gastaut syndrome subjects receiving fenfluramine as an Investigational Product. The reduction in in-clinic visit frequency is also considered to reduce risk for subjects in terms of exposure to COVID19 during a period when the global pandemic still poses considerable uncertainty. The assessment of cardiac function by ECHO performed every six months is aligned with the Sponsor's Global Safety Surveillance for fenfluramine which has now achieved approval in the US and Europe for the indication of Dravet's Syndrome. Information on seizure data and study drug administration will continue to be reported by the parents/caregivers which will enable the Investigator to monitor the subject appropriately and assess benefit-risk despite the decrease in visit schedule. A phone visit will be performed in between in-clinic visits to collect adverse events, concomitant medications and any change in the health status of the subject. Further detail is presented in the Summary of Change section.

This amendment also extends the subject's study participation for up to 5 years in Part 2, to allow subjects to remain on treatment until ZX008 becomes commercially available in the subject's country of residence.

### **List of Specific Changes**

Additions are marked in <u>red</u> and deletions are marked in <u>strikethrough</u>. Minor editorial and nonsubstantive changes, such as the correction of typing or formatting errors, updated use of abbreviations, updating headers and footers, tables of contents, list of abbreviations, signature pages, etc., are not listed. The list of specific changes below is grouped by rationale and not necessarily presented in the order in which they appear in the protocol.

1. Update of Sponsor Information (address, sponsor's representative and medical contact) to reflect the acquisition of Zogenix International Limited by UCB Biosciences Inc.


### CLINICAL STUDY PROTOCOL

Study Title: A Two-Part Study of ZX008 in Children and Adults with

Lennox-Gastaut Syndrome (LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures in Children and Adults with LGS, Followed by Part 2: An Open-label Extension to Assess Long-Term Safety of ZX008 in Children and Adults

with LGS

Study Number: ZX008-1601

Study Product: Fenfluramine Hydrochloride Oral Solution: ZX008

IND Number: 132604

2017-002628-26 EudraCT Number:

Sponsor: Zogenix International Limited

A wholly owned subsidiary of Zogenix UCB Biosciences,

4000 Paramount Pkwy,

Carolina 27560, United States 5959 Horton Street, FL 5 Emeryville, CA 94608 USA

Sponsor's Medical Contact:

Program Physician UCB Biosciences Inc

Date and Version of Study Protocol:

Draft 27-25 June-July

29 July 2020 (PA 3 2

PANIJapan JPO OF Jarrations thereof.

The part of the pacipation in Part 2 to up to 5 years (5 annual 2. Update to extend the subject extensions, 72 months)

Updates were made to the language in study synopsis, sections 3.1, 3.3, 3.5, 6.2. Table 2: Schedule of Assessme **©** ohort B only- and Table 11 have also been updated to add proced extension to up to 5 years, Month 72 (see. next section for study visits to accome detailed modific

### Estimated Duration of Individual Subject Participation:

The duration of participation in the study for an individual subject in the decoration of participation in the open-label extension (Part 2) is up expected to be up to 20 weeks. The duration of participation in the open-label extension (Part 2) is up in the study for an individual subject in the double-blind study (Part 1) is ZX008 is approved in a subject's country of residence and listed on a patient's plan form (w), whichever occurs first. The total participation time is up to approximately 417 ins. Regardiess of whether subjects end participation early, do not continue with the open-label xy, whichever occurs first. The total participation time is up to approximately 4177 tension, or roll over to the open-label extension, all subjects who do not transition to commercial drug will have a follow-up visit 3 to 6 months after the last dose of study medication for final safety monitoring

Objectives:


### **Duration of Treatment:**

In Part 1 all subjects will receive ZX008 or matching placebo for up to approximately 16 weeks (Titration Period=2 weeks; Maintenance Period=12 weeks; Taper/Transition Period=2 weeks). At the end of the 12-week Maintenance Period, eligible subjects may enroll into Part 2, the open-label extension, after completing a 2-week transition period with blinded study medication. Subjects who enroll in Part 2 will have the option to receive ZX008 for up to 3672 months (plus a 2-week taper at the end of the open-label extension), or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever comes first. Subjects who do not enroll in the open-label extension will undergo a taper off of study medication (doses will be administered in a blinded fashion similar to the titration, ie, doses will be decreased in 4-day increments). Follow-up

### Study synopsis/Methodology

- Neiling authoritation Part 2 is an open-label, long-term safety study of ZX008 for subjects who have successfully completed 14 weeks of treatment (titration + maintenance) in Part 1 and are candidates for continuous treatment for an extended period of time; subjects who have not completed the entire 14 weeks of treatment in Part 1 may be eligible to participate in Part 2 on a case-by-case basis and only following sponsor approval. Part 2 will consist of a 12-month Open-Label Extension (OLE) Treatment Period and a 2week Post-Dosing Period. Thus, subjects who complete 12 months of OLE in Part 2 will have been treated with ZX008 for at least 70 weeks (including their participation in both Part 1 and Part 2). If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary. Up to 2-5 annual extensions can be applied, for a total treatment time of up to 36 72 months in the OLE. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk.

### Section 3.1:

treated with ZX008 for at least 70 weeks (including their participation in both Part 1 and Part 2). If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary. Up to 25 annual extensions can be applied, for a total treatment time of 3672 months in the OLE. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk.

### Section 3.3:

Subjects who enroll in Part 2 will have the option to receive ZX008 for up to 3672months (plus a 2-week taper at the end of the open-label extension), or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever occurs first-

Subjects will receive investigational medicinal product (IMP; ZX008 or placebo) in addition to their existing antiepileptic medications at their stable doses throughout the entire Part 1. Thus, subjects receiving placebo will not be denied active therapy; they will continue to receive their existing medications at the exact same dosages. As the principal study measurement (seizures that result in drops) might be considered subjective, a double-blind study design will prevent subjective bias. Upon completion of Part 1, eligible subjects will be able to receive ZX008 in Part 2, the open-label extension, for up to 45 additional years of treatment.

### Section 6.2.5:


The next study visit after Visit 25/Month 21, Visit 29/Month 33, Visit 33/Month 45, Visit 37/Month 57 or Visit 41/Month 69 should be Visit 3042 (EOS), unless another 1-year extension proved er an in is granted. If extending study participation, the decision should be made during Visit 25/Month-21 (or at least prior to conducting Visit 26/Month 24 procedures) the in-clinic visit preceeding the annual reconduction by the Investigator and the consent from the subject or parent/caregiver obtained. After approval from Investigator and Sponsor for extension and starting after Visit26/Month 24 (or a later visit if Visit 26/Month 24 has already occurred at the time of Protocol Amendment 4.0 approval), sSubject will return to the clinic every 36 months and will have a phone visit 3 months after each in-clinic visit for the 1 year extension. The End of Study will be Visit 42, the 3672nd month of the OLE, or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever occurs first.

### Section 6.2.6:

### 6.2.6 Clinic Visit 42: End of Study/Early Termination

The End-of-Study participation in Part 2 for an individual subject occurs after he/she has received IMP for up to 53 years in the Part 2 OLE Treatment Period, or until ZX008 is approved in a subject's country of residence and listed on a patient's health plan formulary, whichever occurs first. The End-of-Study visit may also occur if the subject withdraws participation from in Part 2 or the Sponsor terminates the study.

Subjects will visit the clinic for the End-of-Study visit if one the following events occur

- 1. The subject withdraws or is withdrawn from participation in the study.
- 2. The Sponsor terminates the study.
- The subject completes all study related visits and procedures (at least up to Month 12, but extensions may be granted for up to 3672 months).
- 4. ZX008 is approved in a subject's country of residence and is listed on a patient's health plan formulary

## 3. Update to reduce the in-clinic study visit schedule to every 6 months.

From Visit 26/Month 24 (or a later visit if Visit 26/Month 24 has already occurred at the time of Protocol Amendment 4.0 approval), subjects will perform in-clinic visits every 6 months. Study visits have been added to accommodate the addition of the annual extensions for up to 5 years. Phone visits will be performed between in-clinic visits (3 months after the last in-clinic visit).

Updates were made to Table 2 and Table 11, as well as Sections 6.2 in order to increase the number of visits (phone or in-clinic visits) up to 72 months. Visit numbers have been updated accordingly.

### Study Synopsis/ Methodology

the 12 month QLE subjects will have ECG and ECHO assessments at months 1, 3, 6, and 9, and at the end of study visit. In the event the OLE is extended, subjects will continue to have ECG (if clinically indicated) and ECHO assessments every 63 months until the end of their participation in the study.

Table 2: Schedule of Assessments: Part 2 Cohort B only


ZX008 (Fenfluramine Hydrochloride) ZX008-1601 Clinical Study PA 4.0 (Japan) 25 July 2022

### Table 2. Schedule of Assessments: Part 2 Cohort B only-

| Last Visit Number/Study Month pre approval of Amendment 4.0 | <u>N</u> o | ext In Clinic Visits to be S | cheduled (until ZX008 ap<br>-Every 6 months- | proval by health authori | ty) |
|---|---|---|---|---|---|
| Visit 26 / Month 24 | Visit 28/M30 | Visit 30/M36 | Visit 32/M42 | Visit 34/M48 | Visit 36/M54 |
| Visit 27 / Month 27 | Visit 29/M33 | Visit 31/M39 | Visit 33/M45 | Visit 35/M51 | |
| Visit 28 / Month 30 | Visit 30/M36 | Visit 32/M42 | Visit 34/M48 | Visit 36/M54 | |
| Visit 29 / Month 33 | Visit 31/M39 | Visit 33/M45 | Visit 35/M51 | | |
| Visit 30 / Month 36 | Visit 32/M42 | Visit 34/M48 | Visit 36/M54 | | |

| After Visit 26 Month 24 (or a later visit if V26 Month 24 visit has already been performed at the time of Protocol Amendment 4.0 approval), in clinic study visits will occur every 6 months until XX008 is approved by the subject country of residence and listed on the patient health plan formulary. A phone visit will be performed between in clinic visits (with a 3-month interval). During the phone visits, only a review of concomitant medications, adverse events and adverse events of special interest will be performed. Last Visit Number/Study Month pre approval of Amendment 4.0 | the matient benith along forms | | | | | | ed by the subject cou | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit 27 / Month 27 | me panem neam pian form | ulary. A ph | one visi | t will be | performed be | tween in clir | nic visits (with a 3-m | onth interva | al)Durin | g the phone | |
| Visit 27 / Month 27 | visits, only a review of con- | comitant me | edication | is, adve | rse events and | adverse eve | nts of special interes | t will be per | formed. | | |
| Visit 27 / Month 27 | | | | | | | | | | | . (2) |
| Visit 27 / Month 27 | | | | | | | | | | | . 19 |
| Visit 27 Month 27 | | | | | | | | | | | |
| Visit 27 Month 27 | | pre approval | | | Next In Clini | c Visits to be Sc | | roval by healtl | h authority) | | |
| Visit 27 / Month 27 | of Amendment 4.0 | | | | | | -Every 6 months- | | | | _ ( ) ` |
| Number Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 15* | Visit 26 / Month 24 | | Vi | isit 28/M30 | Visit | 30/M36 | Visit 32/M42 | Visit 34/M | [48 | Visit 36/M54 | |
| Number Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 15* | | | | | | | | | | | XI |
| Number Visit 15* Visit 16* Visit 17-21 (Months 1, 2, 3, 6 and 9**) Visit 22* (Month 12) Visit 23-241 (Months 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 56) (EOS/ET) Visit 43* (EOS/ET) Visit 44* and 45* (EOS/ET) Visit 43* (EOS/ET) Visit 44* (EOS/ET) Visi | | | | | | | | Visit 36/M | <u>154</u> | | |
| Number Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 15* | | | | | | | | | | | J. C. |
| Number Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 16* Visit 15* Visit 15* | Visit 30 / Month 36 | | Vi | isit 32/M42 | Visit | 34/M48 | Visit 36/M54 | | | | |
| Number Visit 15* | v Assessments – PART 2 | | | | OLE Tre | atment Period* | * | | Post- | Cardiac Follow-up | .(0) |
| Clinic Phone | • | | | | | | | | | | |
| Study Day 1 | Number | Visit 15* | Visi | t 16 <sup>b</sup> | | | | | Visit 43 | Visit <u>44</u> and <u>45</u> | <b>')</b> |
| Study Day 1 | | | | | | (Month 12) | | (EOS/ET) | | | |
| Study Day 1 | | | | | 3, 0 and 9^^) | | | | | Lo XX. | |
| 180, and 270 | | | | | | | | | ( ) | | |
| 1170, 1260, 1350, 1350, 1440, 1530, 1620, 1710, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1890, 1980, 2070 1710, 1890, 1890, 1890, 1890, 1890, 1890, 1980, 2070 1710, 1890, | Study Day | la la | 1 | 5 | | 360 | 450, 540, 630, 720, | 2160 | 2174k.q | (3 and 6 months post | |
| 1440, 1530, 1620, 1710, 1890, 1890, 1970 1980, 2070 | | | | | 180, and 270 | | | | ~'0" | last dose) <sup>d,k</sup> | |
| Clinic Phone | | | | | | | 1170, 1260, 1350, | | | | |
| Clinic Phone Cffrite Phone | | | | | | | | | | | |
| Clinic Phone Cfinie Cfinie Cfinie Phone Cfinie | | | | | | | | | | | |
| Criteria | | | Clinic | Phone | | | | 7 | ·. 0 | | |
| | | | | | | X** | X** | | 1 | | |
| cal Neurological History X° psv History X° X X X X X | | | | | | | | * | 1 . | | |
| psy History X <sup>a</sup> cal Examination, complete X <sup>a</sup> X X | agraphice | | | | | | 77 | | <b>^</b> | | |
| cal Examination, complete X <sup>a</sup> X X | | | | | | | | - | | | |
| | cal/Neurological History | | I | | | (11 | | . V | | v | |
| ical Examination, abbreviated X <sup>m</sup> X <sup>m</sup> X | cal/Neurological History<br>psy History | | | | | | | | | | |

| Study Assessments – PART 2 | | | | | atment Period** | | ) | | Post-<br>Dosing | Cardiac Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | Visit 15ª | Visi | 16 <sup>b</sup> | Visits 17-21<br>(Months 1, 2,<br>3, 6 and 9**) | Visit 22<br>(Month 12) | Visits 23-4<br>15, 18, 21,<br>33, 36, 39,<br>51, 54, 57, | 24, 27, 30, | Visit 42°<br>(EOS/ET) | Visit 43 | Visit <u>44</u> and <u>45</u> |
| | | | | 0.0 | XC | 51, 54, 57,<br>69 | <u>00, 03, 00,</u><br>9) | | | |
| Neurological Examination, complete | X <sup>e</sup> | | | ~ | X | | | X | | |
| Neurological Examination, abbreviated | | X <sup>m</sup> | | X <sup>m</sup> | | X <sup>m</sup> | | | $X^{m}$ | |
| Vital signs | X | X | | X | X | X | | X | | |
| Weight | X <sup>a</sup> | X | | ✓ X ( | X | X | | X | X | |
| Height | X <sup>a</sup> | | 0 | - 1 | X | | | X | | |
| 12-lead ECG | X <sup>a</sup> | | | X | X | <u>X</u> q | | $X^q$ | | X |
| Doppler ECHO | X <sup>a</sup> | V | | Xts | X | Xg | | X | | X |
| Urine or Serum Pregnancy Testh | X <sup>a</sup> | 4. | 7 | X <sup>n</sup> | X | X | | X | | |
| Clinical laboratory evaluation<br>(hematology/chemistry/urinalysis <sup>p</sup> , etc) | X <sup>i</sup> | X <sup>i</sup> | 2 | CX <sup>n</sup> | X | $\underline{X}^q$ | | Xq | | |
| Urine or serum THC Panel | X <sup>a</sup> | | | X <sup>n</sup> | X | | | X <sup>s</sup> | | |
| Whole blood CBD | X- | | | X <sup>n</sup> | X | | | X <sup>s</sup> | | |
| Plasma sample for background AEDs | | X <sup>m</sup> | | X <sup>n</sup> | X | <u>X</u> q | | X <sup>q</sup> | | |
| Tanner Staging (for subjects >7 to 18 years old) | X | - 6 | | X <sup>j</sup> | X | | | X <sup>s</sup> | | |
| C-SSRS | $X^{a}$ | | | X | X | <u>X</u> | | X | | |
| CGI-I (assessed by parent/caregiver) | X <sup>a</sup> | | | X | X | X | | X | | |
| CGI-I (assessed by investigator) | X <sup>a</sup> | | | X | X | <u>X</u> | | X | | |
| Overall change in seizure frequency<br>(assessed by investigator) | 111 | ) | | | | <u>X</u> <sup>r</sup> | | Xr | | |
| HADS (Effect of parent/caregiver) | X | | | X° | X | | | X <sup>s</sup> | | |
| BRIEF | X- | | | X <sup>o</sup> | X | | | X <sup>s</sup> | | |
| QOLCE | $X_{a}$ | | | X° | X | | | X <sup>s</sup> | | |
| Zarit Burden | X <sup>a</sup> | | | | X | | | X <sup>s</sup> | | |
| Subject Diary | C/R/D | C/R/D | R | C/R/D | Xr | <u>X</u> <sup>r</sup> | | C/R <sup>r</sup> | C/R | |
| Study Medication | C/R/D | C/R | R | C/R/D | C/R/D | C/R/D | | C/R/D | C/R | |
| Daily Diary Completion | | X | | | | | | | | |
| Concomitant Medication | Xa | | | | X | | | | | |
| Adverse Events | Xa | | | | X | | | | | |
| Adverse events of special interest | Xa | | | | X | | | | | X <sup>i</sup> |

nabidiol; D=Dispense; ECG=electrocardiogram; EOS=end of study; ET=early termination; HADS=Hospital Anxiety and Depression Scale; BRIEF=Behavior Rating Inventory of Executive Function


nation. — up visits will be conducted for subjects who terminate early from Part 2 and for those who complete Part 2. Standard follow-up visits should occur 3 and 6 months after the last dose. If there are any findings at a post-dose in 12 minutes of stabilized.

It? I afformation unless complete earnoulogical examination is warranted based on significant changes in subject status.

| Study Assessments – PART 2 | | | Post-<br>Dosing | Cardiac Follow-up | | | | |
|---|---|---|---|---|---|---|---|---|
| Visit Number | Visit 15 <sup>a</sup> | Visit 16 <sup>b</sup> | Visits 17-21<br>(Months 1, 2,<br>3, 6 and 9**) | Visit 22<br>(Month 12) | Visits 23-41 (Months<br>15, 18, 21, 24, 27, 30,<br>33, 36, 39, 42, 45, 48,<br>51, 54, 57, 60, 63, 66,<br>69) | Visit 42°<br>(EOS/ET) | Visit <u>43</u> | Visit <u>44</u> and <u>45</u> |

- ECHOs will be performed at Months 1, 3, 6, and 9.

  The Months 3, 6, 9, 12, 18, 12, 124, 27, 30, 33, 36, 59, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69 & 72, ECHO may be performed any time within 3 weeks prior to the study visit. If a subject discontinues early from the study, the ECHO should be Females of Called New Parts Part of Called New Part 1 Visit 12 unless clinical laboratory evaluation is optional based on subject status. Visit 20 only.

- Visit 20 only

  For subjects who are transitioning to commercial drug, do not initiate drug taper or conduct post-dosing and cardiac follow-up visits.

  Only adverse events related to cardiac safety will be collected at this visit.

  An abbreviated physical and on encodogical examination to be conducted as appropriate based on last exam and reported AEs.

  Visit 19, 20, and 21 (Months 3, 6, and 9) only.

  Visit 20 (Month 9) only

  Visit 20 (Month 9

### Table 11: Time Windows for Assessments in Part 2:

### Table 11. Time Windows for Assessments in Part 2

| Visit Number | Visit 15 <sup>a</sup> | Visit 16b | Visits 17-21 | Visit 22 | Visits 23-41 (Months | Visit 42° | Visit 43 | Visit <u>44</u> and <u>45</u> |
|---|---|---|---|---|---|---|---|---|
| Visit Number | VISIT 13 | VISIT 10 | (Months 1, 2,<br>3, 6 and 9**) | (Month 12) | 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, | (EOS/ET) | | |
| f: ECHOs will be performed at Months 1, 3, 6, and 9 | | | | | <u>51, 54, 57, 60, 63, 66,</u><br><u>69</u> ) | | | e study, the ECHO should be subject status. of the study past 12 months). will assess the percent |
| f: ECHOs will be performed at Months 1, 3, 6, and S g: The Months 3, 6, 9, 12, 18, 21, 24, 27, 30, 33, 36, scheduled as soon as practical. h: Females of child-bearing potential | 39, 42, 45, 48, 51, 5 | 4, 57, 60, 63, 66, 69 & | 72_ECHO may be perfo | ormed any time within | :3 weeks prior to the study visit. If a | a subject discontinu | ses early from the | study, the ECHO should be |
| i: For Visit 15, use data collected at Part 1 Visit 12 u<br>j: Visit 20 only.<br>k: For subjects who are transitioning to commercial of | | | _ | | status. For Visit 16, clinical laborate | ory evaluation is op | tional based on sy | abject status. |
| <ol> <li>Only adverse events related to cardiac safety will?</li> <li>An abbreviated physical and/or neurological exam</li> </ol> | ll be collected at this vi | visit. | - | | | | | |
| n: Visits 19, 20, and 21 (Months 3, 6, and 9) only. o: Visit 20 (Month 6) only Urine for urinalysis may be collected at home, the | | | | | | | | |
| | | | | | | bjects who do not coided by the caregive | ontinue in Part 2 | of the study past 12 months).<br>will assess the percent |
| improvement in seizure burden on a 5-point scale:<br>s: Only applicable for subjects ending Part 2 particip | .: <25%, ≥25%, ≥50%<br>ipation within the firs | <ol> <li>≥75%, 100% [ie, seiz<br/>t 12 months. Not applic</li> </ol> | zure-fee] improvement.<br>cable for subjects who c | completed Visit 22 and | i extended participation in Part 2. | | | 14 |
| ** If marketing approval is not yet received after tannual extensions can be applied, for a total treats comply with investigator's instructions, and for v | the end of the OLE T<br>ment time of 3672 m<br>whom the investigato | reatment Period, treatment on the OLE. Cont or judges benefit outwer | nent may be extended or<br>tinuation will be based o<br>tighs risk. The decision to | m an annual basis in or<br>on review of safety/tole<br>to extend and informed | tder to provide continuity of treatme<br>erability and effectiveness, and be o<br>diconsent should be completed befor | ent for subjects who<br>offered for subjects<br>are the start of the fir | are enrolled in P<br>who continue to r<br>irst visit of the ear | art 2 of the study. Up to 25<br>meet eligibility requirements,<br>th annual extension (e.g. i.e. |
| Month 12, or 24, 36, 48 and 60). After approval f<br>, subject will return to the clinic every 6 months a<br>if marketing approval is not yet received | from Investigator and<br>and have a phone visi | i Sponsor for extension<br>at 3 months after the in | and starting after Visit2<br>clinic visit for each 1-y | 26/Month24 (or a later<br>year extension, until up | visit if Visit26/Month24 visit has a<br>to Month 72. The End of Study wi | ilready occurred at t<br>ill be Visit 42. Furth | the time of Protoc<br>her extensions car | ol Amendment 4.0 approval) then be applied as required |
| | | | | | | | | THE CANAL |
| | | | | | | | | O'III, NO. |
| Table 11: Time Wind | dows f | or Asse | cemente | in Part | 2. | | | to 111, |
| Table 11. Time win | <u>uows 1</u> | JI Asses | Silicitis | III I ait A | <u> </u> | | | , 25 |
| As cumucally motorated for subjects expending Part. Electronic diary is to be used the first I months of After 12 months in Part 2, settine diaries are not in improvement in settine burden on a 5-point scale. Only applicable for subjects ending Part 2 participation of the part 2 participation of the part 2 participation of the part 2 participation of the partici | indows f | for Asses | ssments ir | n Part 2 | | < | 7 | . 011 |
| Visit / Procedure | | | | | Time window | (relativ | e to sch | eduled |
| Visit 15 (Clinic; OLE Stud | | | | | visit ∤ procedu | ire) | <del>- (C</del> | - |
| Visit 15 (Clinic, OLE Stud | | | | | = 3 days | <del>)``</del> | <u>₩</u> | |
| Visits 17-41 (Clinic: OLE | | | | 270. 360. | ± 4 days | 1 | <u> </u> | |
| 450, 540 <u>*</u> , 630, 720 <u>*</u> , 810 | 0, 900 <u>*</u> , 99 | 90 <u>, 1080*,</u> | , 1170,1260 | | | | | |
| 1440*,1530, 1620*, 1710, | , 1800*, 1 | <u>1890, 1980</u> | <u>/*, 2070)</u> | <u>U</u> | 6X 6 | | | |
| Visit 42 (Clinic; OLE Stud | | | | | # 4 days | | | |
| Visit 4331 (Clinic; OLE S | | | | | ± 4 days | | | |
| Visit 4432, 4533 (ECHO of<br>AED=antiepileptic drug (s); E | ECHO=echo | nocardiogram | n | 10 | + 30 days | | | |
| <sup>a</sup> In the case of a required safe<br>extended up to 14 days to allo | ety review o | of a Visit 12 | ECHO alert, | the transiti | on period between | . Visit 12 a | and Vist 1 | 5 may be |
| *If marketing approval is not yet receive | eived after the e | end of the OLE 1 | Treatment Period | od, treatment m | ay b <u>e extended on an an</u> | mual basis in | o <u>rder to pro</u> | wide continuity |
| of treatment for subjects who are enrol<br>Continuation will be based on review of | olled in Part 2 o<br>of safety/tolera | of the study. Up<br>rability and effec | p to 5 annual extensions and be | tensions can be a<br>se offered for sub | applied, for a total treatm<br>bjects who continue to m | ment time of 7:<br>meet eligibility | 72 months in<br>ity requiremen | n the OLE.<br>ents, comply |
| with investigator's instructions, and for | or whom the in | nvestigator judge | ges benefit outwei | eighs risk. The d | decision to extend and in | informed conse | sent should b | be completed |
| Visit 26/ Month24 (or at a later visit if<br>clinic every 6 months for the 1 year ex | f Visit 26/ Mor | nth 24 visit has / | already occured | d at the time of P<br>tv will be Visit 4 | Protocol Amendment 4.0<br>42, unless another extens | .0 approval), su<br>asion is granted | subject will re<br>ed. in which o | return to the<br>case the subject |
| will continue to return for clinic visits<br>required if marketing approval is not v | every 6 month | hs and will have | a phone visit 3 | months after th | ie in-clinic visit. Further | a extensions c | can then be | applied as |
| tedimen it marketing abbroom to not 1 | et secesses. | , ~ | <i>&gt;</i> | | | | | |
| Section 6.2.5: | 0, | 0 | | | | | | |
| | D. 1 | | | | | | | |
| X | 1:40 | | | | | | | |
| | VIII | | | | | | | |
| ~\o`.'.( | .'0' | | | | | | | |
| 10. 11. | | | | | | | | |
| Ch. OK | | | | | | | | |
| 70, 8% | | | | | | | | |
| 0 | | | | | | | | |
| ı | | | | | | | | |
| Visit 26/1 Month24 (or at a later visit if clinic every 6 months for the 1 year ex will continue to return for clinic visits required if marketing approval is not y | | | | | | | | |


### 6.2.5 Clinic Visits 23-2941 (OLE Months 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69)

If marketing approval is not yet received after the end of the OLE Treatment Period, treatment may be extended on an annual basis in order to provide continuity of treatment for subjects who are enrolled in Part 2 of the study. Continuation will be based on review of safety/tolerability and effectiveness, and be offered for subjects who continue to meet eligibility requirements, comply with investigator's instructions, and for whom the investigator judges benefit outweighs risk.

From Visit 26/Month 24 (or a later visit if Visit 26/Month 24 has already occurred at the time of Protocol Amendment 4.0 approval), if approved for the extensions, Ssubjects will report to the clinic every 6 months and will have a phone visit 3 months after each in-clinic visit for Part 2 Clinic Visits 263 through 2941.

The following procedures will be performed during in-clinic visits:

- Record concomitant medications
- Obtain weight (Note: if the subject's weight is ±25% of the weight at Part 2 Day 15 the IMP dose will be recalculated)
- Obtain vital signs
- Abbreviated physical examination, as appropriate based on last exam and reported AEs
- Abbreviated neurological examination, as appropriate based on last examinated reported
- 12-lead ECG, if clinically indicated
- Doppler ECHO
- · Urine or serum pregnancy test for females of child-bearing potential
- Only if clinically indicated:
  - o Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
  - o Collect plasma sample for AED PK and document time of last dose
- Seizure Assessment by Investigator
- C-SSRS Since Last Visit Assessment (Appendix 2)
- ALST SULL STATE OF THE STATE OF CGI-I (assessed by parent/caregiver)
  - CGI-I (assessed by investigator)


- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication

### The following procedures will be performed during phone visits:

- Record concomitant medications
- Record AEs
- Record AESI

authoril ation The next study visit after Visit 25/Month 21, Visit 29/Month 33, Visit 33/Month 45, Visit 37/Month 57 or Visit 41/Month 69 should be Visit 3042 (EOS), unless another 1-year extension is granted. If extending study participation, the decision should be made during Visit 25 Month 21 (or at least prior to conducting Visit 26/Month 24 procedures) the in-clinic visit proceding the annual reconduction by the Investigator and the consent from the subject or parent/caregiver obtained. After approval from Investigator and Sponsor for extension and starting after Visit26/Month24 (or a later visit if Visit 26/Month 24 has already occurred at the time of Protocol Amendment 4.0 approval), sSubject will return to the clinic every \$6 months and will have a phone visit 3 months after each in-clinic visit for the 1 year extension. The End of Study will be Visit 42, the 3672th month of the OLE, or until ZX008 is approved in the subject's country of residence and listed on a patient's health plan formulary, whichever occurs first.

### 4. Updates to the blood volume collected during the study.

The range of blood volume collected during Part 2 has been updated to reflect the reduced visit schedule from V26/Month24 (or a later visit if V26/Month24 has already occurred at the time of PA4.0 approval).

### Section 6.4:

The maximum total blood volume collected during Part 1 of the study for clinical laboratory testing, genotyping, and PK will be approximately 84.0 mL, as outlined in Table 13 The maximum total blood volume collected during Part 2 of the study for clinical laboratory testing and PK will be variable as the clinical laboratory testing will be performed as clinically indicated for the majority of in clinic visits after Visit26/Month 24, and will be approximately 104110.0 Lhis 90011Ulable mL at the minimum and will equal up to 351.5 mL, as outlined in Table 14.


Table 14. Maximum Estimated Blood Volume Collection for Part 2\*

| PART 2 | Visit 19<br>(Day 90) | Visit 20 (Day<br>180) | Visit 21 (Day 270) | Visit 22 (Day 360) | Visits 23-<br>42 (in<br>clinic<br>only) | TOTAL | |
|---|---|---|---|---|---|---|---|
| Chemistry | 5.0 mL | 5.0 mL | 5.0 mL | 5.0 mL | | 2520.0 mL | |
| Pregnancy test<br>(serum) | included in<br>Chemistry | included in<br>Chemistry | included in<br>Chemistry | included in<br>Chemistry | 2.5 mL | 2. <del>0-5</del> mL | :1311011 |
| Hormones | 5.0 mL | 5.0 mL | 5.0 mL | 5.0 mL | | 2520.0 mL | .1.0. |
| | | | | | | <del>12.5</del> 10.0 | |
| Immunoglobulin | 2.5 mL | 2.5 mL | 2.5 mL | 2.5 mL | | mL | 0 |
| Hematology | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | | <del>10.0</del> 8.0<br>mL | |
| AED PK plasma | | | | | | <del>10.0</del> 8.0 | |
| sample | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | | mL | .0. |
| Cannabidiol/THC | 2.0 mL | 2.0 mL | 2.0 mL | 2.0 mL | | 8.010.0<br>mL | eting autilia. |
| | | | | | | | 10,100, |
| | | | | | <del>17.5</del> <u>30</u> | <del>110</del> 104.0 | Ø X() |
| TOTAL | 18.5 mL | 18.5 mL | 18.5 mL | 18.5 mL | mL | mL | |
| AED=Anti-epileptic drugs; PK=pharmacokinetics *Laboratory testing may be conducted on Visits 16-18 and 23-4239 if clinically indicated. After Visit 26, in-clinic visits will occur every 6 months. If collected during these visits, the total blood volume per subject would equal up to | | | | | | | |
| 531.3 <del>270.3</del> 1111. | 351.5276.5mL. | | | | | | |

| | | | | | <del>17.5</del> <u>30</u> | 110104.0 |
|---|---|---|---|---|---|---|
| TOTAL | 18.5 mL | 18.5 mL | 18.5 mL | 18.5 mL | mL | mL |
| APP 4 (1 11 (1 1 | Drr 1 | 4 | | | | |

AED=Anti-epileptic drugs: PK=pharmacokinetics

## 5. Update to clarify the timing of analysis of 1601 Cohort A and Cohort B

Clarification has been made to reflect the timing of data analysis performed for Cohort A and Cohort B.

Updates have been made to study synopsis and sections 10.

### Study Synopsis/ Methodology:

and Australia; Cohort B will include randomized subjects from Japan only. The primary study endpoint is assessed from Part 1 Cohort A data. The primary analysis will be conducted when the last subject in Cohort A has completed Part 1. Cohort B will be analyzed independently with the an interim analysis occurring after the last subject in Cohort B completes 12 months in Part 2 and a final analysis when the last subject in Cohort B completes Part 2. Part 2 will be an open-label, flexible-dose extension for subjects completing Part 1 of the study.

### Study Synopsis/ Statistical Methods:

The primary analyses of the study will be performed on data from Part 1 Cohort A after the last subject enrolled in Cohort A has completed the last study visit of Part 1. Data from Part 1, Cohort B will be analyzed independently after the last subject in Cohort B completes Part 1. An interim analysis of Part 2 will be performed after all Cohort B subjects complete 12 months in Part 2. A secondary analysis will be conducted after the last Cohort B subject has enrolled and completed the last study visit of Part 2. Analysis results for Part 1 from Cohort A and Cohort B will may be compared through descriptive statistics, and if reasonable, some analyses may be performed using data from Cohort A and Cohort B combined. Subjects randomized to 0.5 mg/kg/day (ie, those taking concomitant STP) will be grouped with subjects randomized to 0.8 mg/kg/day for all efficacy analyses.


<sup>\*</sup>Laboratory testing may be conducted on Visits 16-18 and 23-4239 if clinically indicated. After Visit 26, in-clinic visits of the conducted on Visits 16-18 and 23-4239 if clinically indicated. vill occur every 6 months. If collected during these visits, the total blood volume per subject would equal up to

### Part 2

The primary objective of Part 2 is to assess the long-term safety and tolerability of ZX008 in children and adults with LGS with regard to AEs, laboratory parameters, physical examination, neurological examination, vital signs, ECG, ECHO, body weight, and BMI.

The number and percentage of subjects who experience treatment emergent AEs will be displayed by body system and preferred term using MedDRA. Summaries in terms of severity and relationship to study drug will also be provided. SAEs will be summarized separately in a similar manner. Laboratory tests, vital signs, physical examinations, neurological examinations, ECG, ECHO, cognition and body weight will be summarized using appropriate methods.

Effectiveness will be assessed by the change from baseline (prior to randomization into Part 1) in DSF. The DSF per 28 days will be calculated as the number of seizures that result in drops divided by the number of days in the period and multiplied by 28. The change in DSF during the first 12 months of

Confidential Page 27 of 18

ZX008 (Fenfluramine Hydrochloride) ZX008-1601 Clinical Study PA 4.0 (Japan) 25 July 2022

Part 2 OLE Treatment Period will be calculated as the difference between DSF during the OLE and the baseline DSF measured prior to randomization in Part 1. Both the mean and median percent change in DCF will be presented and the statistical significance of the percent change will be assessed using a Wilcoxon signed-rank test. Other secondary assessments will be compared to baseline from prior to Part 1, or by visit throughout Part 1 and the first 12 months of Part 2, as appropriate.

### Section 10.1:

### 10.1 STATISTICAL ANALYSIS: PART 1

The primary analyses of the study will be performed on data from Part 1 Cohort A after the last subject enrolled in Cohort A has completed the last study visit of Part 1. Data from Part 1. Cohort B will be analyzed independently after the last subject in Cohort B completes Part 1. An interim analysis of Part 2 will be performed after all Cohort B subjects complete 12 months in Part 2. A secondary analysis will be conducted after the last Cohort B subject has enrolled and completed the last study visit of Part 2. Analysis results for Part 1 from Cohort A and Cohort B will be compared through descriptive statistics, and if reasonable, some analysis may be performed using data from Cohort A and Cohort B combined. Subjects randomized to 0.5 mg/kg/day (ie, those taking concomitant STP) will be grouped with subjects randomized to 0.8 mg/kg/day for all efficacy analyses.

# 6. Addition of language to define the study status between drug approval and launch in Japan

Language has been added in section 1.6.


The rationale for conducting the Part 2 open-label extension period is primarily to evaluate the long-term safety of ZX008 in subjects with LGS. This protocol also provides the opportunity for continued treatment for subjects responding to treatment from Part 1 and an opportunity for initial treatment with ZX008 for subjects randomized to placebo in Part 1. The study will also allow access to ZX008 for the treatment of LGS for eligible Japanese subjects until commercial product is available, as it is not approved in Japan. The period from the approval of this drug to its launch is positioned as a post-marketing study.

### 7. Clarification on the dispensation of study drug to subjects transitioning to commercial drug

Updates has been made to section 6.2.6:

- 12-lead ECG
- Doppler ECHO (must be performed within 3 weeks of the visit; if subject terminates) ECHO was completed ≤ 30 days prior to early termination, the Visit 30 ECHO will not be performed provided the parent/guardian agrees to bring the subject to the clinic for the cardiac follow-up visit (see Table 12).
- Urine or serum pregnancy test for females of child-bearing potential
- Laboratory evaluation (serum chemistry, hematology, immunoglobulin, hormones, and urinalysis) (urine for urinalysis may be collected at home, the night before the clinic visit, as long as collection procedures are followed to maintain sample stability)
- Urine or serum THC panel
- Whole blood CBD
- Collect plasma sample for AED PK evaluation (must document time of last dose)
- Tanner Staging for subjects > 7 to 18 years of age (Appendix 5)
- Collect and review diary C-SSRS Since Last Visit Assessment (Appendix 2)
- CGI-I (assessed by parent/caregiver)
- CGI-I (assessed by investigator)
- BRIEF (Appendix 3)
- QOLCE (Appendix 6)
- HADS (Appendix 7)
- Zarit Caregiver Burden Inventory (Appendix 8)
- Record AEs
- Record AESI
- Collect used, partially used and unused study medication; perform drug accountability and review with parent/caregiver
- Dispense study medication (not applicable for subjects transitioning to commercial drug)

